# **PROTOCOL**

TITLE: A Randomized, Double-Blind Phase 3 Study of Ibrutinib in

Combination With Corticosteroids versus Placebo in

Combination With Corticosteroids in Subjects with New Onset

Chronic Graft Versus Host Disease (cGVHD)

PROTOCOL NUMBER: PCYC-1140-IM

STUDY DRUG: Ibrutinib (PCI-32765)

**IND NUMBER:** 102,688

**EudraCT NUMBER: 2016-003286-26** 

SPONSOR MEDICAL

MONITOR:



SPONSOR: Pharmacyclics LLC

995 East Arques Avenue Sunnyvale, CA 94085-4521 United States of America

**DATE FINAL:** 11 August 2016

Amendment 1 Date: 25 October 2016

Amendment 2 Date: 03 October 2017

Amendment 3 Date: 06 February 2019

#### **Confidentiality Statement**

This document contains confidential information of Pharmacyclics LLC that must not be disclosed to anyone other than the recipient study staff and members of the institutional review board/ethics committee. This information cannot be used for any other purpose other than the evaluation or conduct of the clinical study without the prior written consent of Pharmacyclics LLC.

# PROTOCOL APPROVAL PAGE

Study Title: A Randomized, Double-Blind Phase 3 Study of Ibrutinib in

Combination with Corticosteroids versus Placebo in Combination with Corticosteroids in Subjects with New Onset Chronic Graft

Versus Host Disease (cGVHD)

Study Number: PCYC-1140-IM

Protocol Date: 11 August 2016

Amendment 1 Date: 25 October 2016

Amendment 2 Date: 03 October 2017

Amendment 3 Date: 6 February 2019

I have carefully read Protocol PCYC-1140-IM entitled "A Randomized, Double-Blind Phase 3 Study of Ibrutinib in Combination with Corticosteroids versus Placebo in Combination with Corticosteroids in Subjects with New Onset Chronic Graft Versus Host Disease (cGVHD)".

I agree to conduct this study as outlined herein and in compliance with Good Clinical Practices (GCP) and all applicable regulatory requirements. Furthermore, I understand that the Sponsor, Pharmacyclics, and the Institutional Review Board/Research Ethics Board/Independent Ethics Committee (IRB/REB/IEC) must approve any changes to the protocol in writing before implementation.

I agree not to divulge to anyone, either during or after the termination of the study, any confidential information acquired regarding the investigational product and processes or methods of Pharmacyclics. All data pertaining to this study will be provided to Pharmacyclics. The policy of Pharmacyclics LLC requires that any presentation or publication of study data by clinical Investigators be reviewed by Pharmacyclics, before release, as specified in the protocol.

| Principal Investigator's Signature | Date |
|---|---|
| Print Name | |
| The following Pharmacyclics LLC representative is a amendments: | uthorized to sign the protocol and any |
| | Date |

# TABLE OF CONTENTS

| PROTO | OCOL APPROVAL PAGE | 2 |
|---|---|---|
| <b>TABLE</b> | OF CONTENTS | 3 |
| LIST O | F APPENDICES | 7 |
| | F IN-TEXT TABLES | |
| | SIS | |
| | VIATIONS | |
| 1. | BACKGROUND | |
| 1.1. | Disease/Histology | |
| 1.1.1. | Disease Background. | |
| 1.1.2. | Current Treatment Options | |
| 1.2. | Ibrutinib Overview | |
| 1.2.1. | Summary of Nonclinical Data | |
| 1.2.1.1. | Pharmacology | |
| 1.2.1.2. | Safety Pharmacology and Toxicology | |
| 1.2.2. | Summary of Clinical Data | |
| 1.2.2.1. | Pharmacokinetics and Product Metabolism. | |
| 1.2.3. | Summary of Clinical Safety. | |
| 1.2.3.1. | Monotherapy Studies | |
| 1.2.3.2. | Combination Studies | |
| 1.2.3.3. | Chronic GVHD Study | 21 |
| 1.2.4. | Risks | 22 |
| 1.2.4.1. | Atrial Fibrillation | 22 |
| 1.2.4.2. | Bleeding-related Events | 22 |
| 1.2.4.3. | Cytopenias | 22 |
| 1.2.4.4. | Diarrhea | 22 |
| 1.2.4.5. | Infections | 22 |
| 1.2.4.6. | Interstitial Lung Disease (ILD) | 23 |
| 1.2.4.7. | Non-melanoma Skin Cancer | 23 |
| 1.2.4.8. | Rash | 23 |
| 1.2.4.9. | Hypertension | 23 |
| 1.2.5. | Summary of Clinical Data in Chronic GVHD | |
| 1.3. | Prednisone | 24 |
| 1.3.1. | Summary of Clinical Data | 24 |
| 1.3.2. | Summary of Clinical Safety | |
| 1.3.3. | Summary of Clinical Data in Chronic Graft versus Host Disease | 28 |
| 1.4. | Study Rationale | 28 |
| 2. | STUDY OBJECTIVES | 29 |
| 2.1. | Primary Objective | |
| 2.2. | Secondary Objective(s) | |
| 2.3. | Exploratory Objective(s) | |
| 3. | STUDY DESIGN | |
| 3.1. | Overview of Study Design | |
| 3.1.1. | Study Schema | |

| 4. | SUBJECT SELECTION | 32 |
|---|---|---|
| 4.1. | Inclusion Criteria. | |
| 4.2. | Exclusion Criteria | 33 |
| 5. | TREATMENT OF SUBJECTS | 35 |
| 5.1. | Treatment Allocation and Blinding. | 35 |
| 5.1.1. | Randomized Double-blind Phase | 35 |
| 5.1.1.1. | Blinding | 35 |
| 5.2. | Study Treatment | 36 |
| 5.3. | Study Medication | 36 |
| 5.3.1. | Ibrutinib/Placebo | 36 |
| 5.3.1.1. | Formulation/Packaging/Storage | 36 |
| 5.3.1.2. | Dose and Administration. | 37 |
| 5.3.1.3. | Overdose | |
| 5.3.1.4. | Dose Modification for Adverse Reactions | 37 |
| 5.3.1.5. | Dose Modification for Subjects with Hepatic Impairment | 39 |
| 5.3.1.6. | Ibrutinib/Placebo Hold after Withdrawal of All Immunosuppressants | 39 |
| 5.3.2. | Prednisone | 40 |
| 5.3.2.1. | Formulation/Packaging/Storage | 40 |
| 5.3.2.2. | Dose and Administration. | 40 |
| 5.3.2.3. | Overdose | |
| 5.3.2.4. | Dose Modification for Adverse Reactions | |
| 5.4. | Criteria for Permanent Discontinuation of Ibrutinib/Placebo | 42 |
| <b>6.</b> | CONCOMITANT MEDICATIONS/PROCEDURES | 42 |
| 6.1. | Permitted Concomitant Medications | 42 |
| 6.1.1. | Ancillary Therapy and Supportive Care | 42 |
| 6.1.2. | Systemic Immunosuppressant Therapy | 43 |
| 6.2. | Medications to be Used with Caution | 43 |
| 6.2.1. | CYP3A Enzyme Inhibitors/Inducers | |
| 6.2.2. | Drugs That May Have Their Plasma Concentrations Altered by Ibrutinib | 44 |
| 6.2.3. | Antiplatelet Agents and Anticoagulants | 44 |
| 6.3. | Other Systemic Immunosuppressant Therapy for cGVHD | 45 |
| 6.4. | Guidelines for Ibrutinib Management with Surgeries or Procedures | 45 |
| 6.4.1. | Minor Surgical Procedures | 45 |
| 6.4.2. | Major Surgical Procedures | 45 |
| 7. | STUDY EVALUATIONS | 46 |
| 7.1. | Description of Procedures | |
| 7.1.1. | Assessments | |
| 7.1.1.1. | Informed Consent Form (ICF) | |
| 7.1.1.2. | Confirm Eligibility | |
| 7.1.1.3. | Medical History and Demographics | |
| 7.1.1.4. | Prior and Concomitant Medications | |
| 7.1.1.5. | Adverse Events | |
| 7.1.1.6. | Physical Examination | |
| 7.1.1.7. | Karnofsky/Lansky Performance Scale | |
| 7.1.1.8. | Vital Signs | |
| 7.1.2. | Laboratory | 47 |

| 7.1.2.1. | Hematology | 47 |
|---|---|---|
| 7.1.2.2. | Chemistry (Serum) | |
| 7.1.2.3. | Infection Surveillance | |
| 7.1.2.4. | Coagulation Studies | 48 |
| 7.1.2.5. | Hepatitis Serologies | 48 |
| 7.1.2.6. | Serum Immunoglobulins | 48 |
| 7.1.2.7. | Pregnancy Test | 48 |
| 7.1.3. | Diagnostics/Procedures | 48 |
| 7.1.3.1. | Electrocardiograms (ECG) | 48 |
| 7.1.3.2. | Forced Expiratory Volume in 1 Second (FEV1) | 49 |
| 7.1.4. | Pharmacokinetics/Biomarkers | 49 |
| 7.1.4.1. | Pharmacokinetics | |
| 7.1.4.2. | Biomarkers and Pharmacodynamic Studies | |
| 7.1.4.3. | Biomarker DNA and RNA Sequencing | |
| 7.2. | Sample Collection and Handling | |
| 7.3. | Efficacy Evaluations | |
| 7.3.1. | NIH Consensus Panel Response Criteria | 50 |
| 7.3.2. | Lee cGVHD Symptom Scale and SF-36 Questionnaire | 51 |
| 7.3.3. | Late effects surveillance for adolescents (<22 years at randomization) | 51 |
| 8. | STUDY PROCEDURES | 51 |
| 8.1. | Screening Phase | 51 |
| 8.1.1. | Screening/Consenting Visit | 51 |
| 8.2. | Treatment Phase | 52 |
| 8.2.1. | Treatment Visits | 52 |
| 8.2.1.1. | Week 1 Day 1 | 52 |
| 8.2.1.2. | Week 2 | 53 |
| 8.2.1.3. | Week 5, 9, 13, 17, 21, 25 | |
| 8.2.1.4. | Week 37, 49, and every 12 weeks thereafter (± 7 days) | |
| 8.2.2. | Progressive Disease Visit | |
| 8.2.3. | End-of-Treatment Visit | |
| 8.3. | Follow-up Phase | |
| 8.3.1. | Response Follow-up | |
| 8.3.2. | Long-Term Follow-up | |
| 8.3.3. | Expected length of participation on study | 57 |
| 9. | SUBJECT COMPLETION AND WITHDRAWAL | 58 |
| 9.1. | Completion | 58 |
| 9.2. | Discontinuation from Ibrutinib/Placebo. | |
| 9.3. | Withdrawal from Study | 58 |
| 10. | STATISTICAL METHODS AND ANALYSIS | 59 |
| 10.1. | Analysis Sets | |
| 10.1.1. | Intention-to-Treat Population (ITT) | 59 |
| 10.1.2. | Safety Population (SP) | |
| 10.2. | Sample Size Determination | |
| 10.3. | Subject Information | 60 |
| 10.4. | Efficacy Analyses | 60 |
| 10.4.1. | Primary Efficacy Endpoint. | 60 |

| ) | February 2019 |
|---|---------------|
| | FINAL |

| 10.4.2. | Secondary Endpoints for Efficacy | 60 |
|---|---|---|
| 10.4.3. | Exploratory Endpoints | |
| 10.5. | Safety Analysis | |
| 10.6. | Interim Futility Review | |
| 10.7. | Data Monitoring Committee (DMC) | |
| 11. | ADVERSE EVENT REPORTING | |
| 11.1. | Definitions | 64 |
| 11.1.1. | Adverse Events. | 64 |
| 11.1.2. | Serious Adverse Events. | 65 |
| 11.1.3. | Severity Criteria (Grade 1-5) | 66 |
| 11.1.4. | Causality (Attribution) | 66 |
| 11.2. | Unexpected Adverse Events | 67 |
| 11.3. | Special Reporting Situations | 67 |
| 11.4. | Documenting and Reporting of Adverse Events and Serious Adverse Events by | <b>6</b> 7 |
| 11 / 1 | Investigators | |
| 11.4.1. | Assessment of Adverse Events | |
| 11.4.2. | Adverse Event Reporting Period | |
| 11.4.3. | Expediting Reporting Requirements for Serious Adverse Events | |
| 11.4.4. | Pregnancy | |
| 11.4.5. | Other Malignancies | |
| 11.4.6. | Eye-Related Adverse Events. | |
| 11.4.7. | Adverse Events of Special Interest (AESI) | |
| 11.4.7.1. | Major Hemorrhage | |
| 12. | STUDY ADMINISTRATION AND INVESTIGATOR OBLIGATIONS | |
| 12.1. | Regulatory and Ethical Compliance | 70 |
| 12.2. | Institutional Review Board (IRB), Research Ethics Board (REB) and Independent | 71 |
| 12.3. | Ethics Committee (IEC) Approval Informed Consent | |
| 12.3. | Quality Control and Quality Assurance | |
| 12.5. | Protected Subject Health Information Authorization. | |
| 12.5. | Study Files and Record Retention | |
| 12.7. | Case Report Forms and Record Maintenance | |
| 12.7. | Investigational Study Drug Accountability | |
| 12.9. | Study Monitoring/Audit Requirements | |
| 12.10. | Investigator Responsibilities | |
| 12.11. | Sponsor Responsibilities | |
| 12.12. | Financial Disclosure | |
| 12.13. | Liability and Clinical Trial Insurance | |
| 12.14. | Protocol Amendments | |
| 12.15. | Publication of Study Results | |
| 12.16. | Study Discontinuation | |
| 13. | REFERENCES. | |
| 14. | | 82 |

# LIST OF APPENDICES

| Appendix A. | Schedule of Assessments | 83 |
|---|---|---|
| Appendix B. | Schedule of Assessments for Pharmacokinetics, Pharmacodynamics, | |
| 11 | Biomarker and T/B/NK | 87 |
| Appendix C. | Karnofsky/Lansky Performance Status | |
| Appendix D. | Inhibitors and Inducers of CYP3A | |
| Appendix E. | Child-Pugh Score for Subjects with Chronic Liver Impairment | |
| Appendix F. | Lee cGVHD Symptom Scale | |
| Appendix G. | SF-36 Questionnaire | |
| Appendix H. | Chronic GVHD Activity Assessment – Clinician | 99 |
| Appendix I. | Response Determination for Chronic GVHD Clinical Trials based on | |
| | Clinician Assessments | 102 |
| Appendix J. | Chronic GVHD Activity Assessment – Patient Self Report | 104 |
| Appendix K. | Prednisone Equivalents Table | |
| Appendix L. | Summary of Ancillary Therapy and Supportive Care Interventions | |
| Appendix M. | Diagnosis of cGVHD – Signs and Symptoms of cGVHD | |
| Appendix N. | Staging of cGVHD | |
| Appendix O. | NIH Global Severity/Staging of cGVHD | 117 |
| Appendix P. | Late Effects Surveillance for Adolescents | |
| Appendix Q. | Corticosteroid-related toxicities and CTCAE preferred terms | |
| | LIST OF IN-TEXT TABLES | |
| Table 1. | Ibrutinib/Placebo Dose Modifications | 38 |
| Table 2. | Ibrutinib/Placebo Dose Reduction Levels | |
| Table 3. | Ibrutinib/Placebo Dose Modifications for Subjects with Hepatic Impairment. | |
| Table 4. | Prednisone Taper Schedule | |
| Table 5. | Ibrutinib/Placebo Dose Modifications for Concomitant Use of CYP3A | |
| | Inhibitors | 44 |

# **SYNOPSIS**

| A Randomized, Double-Blind Phase 3 Study of Ibrutinib in Combination With Corticosteroids versus Placebo in Combination With Placebo Will Descriptions Product and Reference Therapy: Investigational Product and Reference Therapy: Ibrutinib (IMBRUVICA*) will be supplied as 70 mg and 140 mg hard gelatin capsules for oral (PO) administration. Placebo will be supplied as hard gelatin capsules and will look identical to ibrutinib capsules. Objectives: Primary Objective: | | T |
|---|---|---|
| Study Duration: Estimated to be up to 7 years | Study Title: | Combination With Corticosteroids versus Placebo in Combination With Corticosteroids in Subjects with New Onset Chronic Graft |
| Study Duration: Estimated to be up to 7 years | <b>Protocol Number:</b> | PCYC-1140-IM |
| Investigational Product and Reference Therapy: Discription of Placebo will be supplied as 70 mg and 140 mg hard gelatin capsules for oral (PO) administration. Placebo will be supplied as hard gelatin capsules and will look identical to ibrutinib capsules. Primary Objective: To evaluate the efficacy of ibrutinib in combination with prednisone (Arm A) versus placebo in combination with prednisone (Arm B) based on the response rate at 48 weeks (the proportion of responders [CR or PR]) as determined by NiH Consensus Development Project criteria in subjects with new onset moderate to severe cGVHD. Secondary Objectives: To compare the two treatment arms in terms of the following: Efficacy Response rate at 24 weeks (the proportion of responders [CR or PR]) as defined by the NIH Consensus Development Project (2014) Duration of response (DOR) Proportion of subjects obtaining steroid dose level less than 0.15 mg/kg/d at 24 weeks Time to withdrawal of all immunosuppressants (with the exception of ibrutinib/placebo) Overall survival (OS) Lee cGVHD symptom scale improvement Safety Safety and tolerability Differences in steroid-related morbidities (eg, hyperglycemia, hypertension) Study Design: This is a Phase 3, multicenter, international, randomized, double-blind study of oral ibrutinib in combination with prednisone versus placebo in combination with prednisone in subjects with new onset chronic GVHD. Approximately 186 subjects with newly diagnosed moderate or severe | Study Phase: | 3 |
| hard gelatin capsules for oral (PO) administration. Placebo will be supplied as hard gelatin capsules and will look identical to ibrutinib capsules. Primary Objective: To evaluate the efficacy of ibrutinib in combination with prednisone (Arm A) versus placebo in combination with prednisone (Arm B) based on the response rate at 48 weeks (the proportion of responders [CR or PR]) as determined by NIH Consensus Development Project criteria in subjects with new onset moderate to severe cGVHD. Secondary Objectives: To compare the two treatment arms in terms of the following: Efficacy Response rate at 24 weeks (the proportion of responders [CR or PR]) as defined by the NIH Consensus Development Project (2014) Duration of response (DOR) Proportion of subjects obtaining steroid dose level less than 0.15 mg/kg/d at 24 weeks Time to withdrawal of all immunosuppressants (with the exception of ibrutinib/placebo) Overall survival (OS) Lee cGVHD symptom scale improvement Safety Safety and tolerability Differences in steroid-related morbidities (eg, hyperglycemia, hypertension) Study Design: This is a Phase 3, multicenter, international, randomized, double-blind study of oral ibrutinib in combination with prednisone versus placebo in combination with prednisone in subjects with new onset chronic GVHD. Approximately 186 subjects with newly diagnosed moderate or severe | Study Duration: | Estimated to be up to 7 years |
| To evaluate the efficacy of ibrutinib in combination with prednisone (Arm A) versus placebo in combination with prednisone (Arm B) based on the response rate at 48 weeks (the proportion of responders [CR or PR]) as determined by NIH Consensus Development Project criteria in subjects with new onset moderate to severe cGVHD. Secondary Objectives: To compare the two treatment arms in terms of the following: Efficacy Response rate at 24 weeks (the proportion of responders [CR or PR]) as defined by the NIH Consensus Development Project (2014) Duration of response (DOR) Proportion of subjects obtaining steroid dose level less than 0.15 mg/kg/d at 24 weeks Time to withdrawal of all immunosuppressants (with the exception of ibrutinib/placebo) Overall survival (OS) Lee cGVHD symptom scale improvement Safety Safety and tolerability Differences in steroid-related morbidities (eg, hyperglycemia, hypertension) Study Design: This is a Phase 3, multicenter, international, randomized, double-blind study of oral ibrutinib in combination with prednisone versus placebo in combination with prednisone in subjects with new onset chronic GVHD. Approximately 186 subjects with newly diagnosed moderate or severe | C | hard gelatin capsules for oral (PO) administration. Placebo will be supplied as hard gelatin capsules and will look |
| (Arm A) versus placebo in combination with prednisone (Arm B) based on the response rate at 48 weeks (the proportion of responders [CR or PR]) as determined by NIH Consensus Development Project criteria in subjects with new onset moderate to severe cGVHD. Secondary Objectives: To compare the two treatment arms in terms of the following: Efficacy Response rate at 24 weeks (the proportion of responders [CR or PR]) as defined by the NIH Consensus Development Project (2014) Duration of response (DOR) Proportion of subjects obtaining steroid dose level less than 0.15 mg/kg/d at 24 weeks Time to withdrawal of all immunosuppressants (with the exception of ibrutinib/placebo) Overall survival (OS) Lee cGVHD symptom scale improvement Safety Safety and tolerability Differences in steroid-related morbidities (eg, hyperglycemia, hypertension) Study Design: This is a Phase 3, multicenter, international, randomized, double-blind study of oral ibrutinib in combination with prednisone versus placebo in combination with prednisone in subjects with new onset chronic GVHD. Approximately 186 subjects with newly diagnosed moderate or severe | Objectives: | Primary Objective: |
| To compare the two treatment arms in terms of the following: Efficacy Response rate at 24 weeks (the proportion of responders [CR or PR]) as defined by the NIH Consensus Development Project (2014) Duration of response (DOR) Proportion of subjects obtaining steroid dose level less than 0.15 mg/kg/d at 24 weeks Time to withdrawal of all immunosuppressants (with the exception of ibrutinib/placebo) Overall survival (OS) Lee cGVHD symptom scale improvement Safety Safety and tolerability Differences in steroid-related morbidities (eg, hyperglycemia, hypertension) Study Design: This is a Phase 3, multicenter, international, randomized, double-blind study of oral ibrutinib in combination with prednisone versus placebo in combination with prednisone in subjects with new onset chronic GVHD. Approximately 186 subjects with newly diagnosed moderate or severe | | To evaluate the efficacy of ibrutinib in combination with prednisone (Arm A) versus placebo in combination with prednisone (Arm B) based on the response rate at 48 weeks (the proportion of responders [CR or PR]) as determined by NIH Consensus Development Project |
| Efficacy Response rate at 24 weeks (the proportion of responders [CR or PR]) as defined by the NIH Consensus Development Project (2014) Duration of response (DOR) Proportion of subjects obtaining steroid dose level less than 0.15 mg/kg/d at 24 weeks Time to withdrawal of all immunosuppressants (with the exception of ibrutinib/placebo) Overall survival (OS) Lee cGVHD symptom scale improvement Safety Safety Safety and tolerability Differences in steroid-related morbidities (eg, hyperglycemia, hypertension) This is a Phase 3, multicenter, international, randomized, double-blind study of oral ibrutinib in combination with prednisone versus placebo in combination with prednisone in subjects with new onset chronic GVHD. Approximately 186 subjects with newly diagnosed moderate or severe | | Secondary Objectives: |
| Response rate at 24 weeks (the proportion of responders [CR or PR]) as defined by the NIH Consensus Development Project (2014) Duration of response (DOR) Proportion of subjects obtaining steroid dose level less than 0.15 mg/kg/d at 24 weeks Time to withdrawal of all immunosuppressants (with the exception of ibrutinib/placebo) Overall survival (OS) Lee cGVHD symptom scale improvement Safety Safety Safety and tolerability Differences in steroid-related morbidities (eg, hyperglycemia, hypertension) This is a Phase 3, multicenter, international, randomized, double-blind study of oral ibrutinib in combination with prednisone versus placebo in combination with prednisone in subjects with new onset chronic GVHD. Approximately 186 subjects with newly diagnosed moderate or severe | | To compare the two treatment arms in terms of the following: |
| study of oral ibrutinib in combination with prednisone versus placebo in combination with prednisone in subjects with new onset chronic GVHD. Approximately 186 subjects with newly diagnosed moderate or severe | | <ul> <li>Efficacy</li> <li>Response rate at 24 weeks (the proportion of responders [CR or PR]) as defined by the NIH Consensus Development Project (2014)</li> <li>Duration of response (DOR)</li> <li>Proportion of subjects obtaining steroid dose level less than 0.15 mg/kg/d at 24 weeks</li> <li>Time to withdrawal of all immunosuppressants (with the exception of ibrutinib/placebo)</li> <li>Overall survival (OS)</li> <li>Lee cGVHD symptom scale improvement</li> <li>Safety</li> <li>Safety and tolerability</li> <li>Differences in steroid-related morbidities (eg, hyperglycemia,</li> </ul> |
| Criteria, will be randomized in a 1:1 ratio to receive either ibrutinib in combination with prednisone (Arm A) or placebo in combination with prednisone (Arm B). | Study Design: | study of oral ibrutinib in combination with prednisone versus placebo in combination with prednisone in subjects with new onset chronic GVHD. Approximately 186 subjects with newly diagnosed moderate or severe cGVHD, as defined by the NIH Consensus Development Project Criteria, will be randomized in a 1:1 ratio to receive either ibrutinib in combination with prednisone (Arm A) or placebo in combination with |
| Treatment with ibrutinib/placebo will be administered continuously | | Treatment with ibrutinib/placebo will be administered continuously |

| | until unacceptable toxicity, progression of the underlying disease, death, or the start of a new systemic treatment for cGVHD. |
|---|---|
| | Ibrutinib/placebo can be discontinued after response in cGVHD disease symptoms and withdrawal of other systemic immunosuppressants (Section 5.3.1.6). |
| | Corticosteroid therapy will be tapered as per a standard taper regimen with the goal of reducing exposure to high-moderate dose corticosteroids as quickly as possible according to clinical severity of cGVHD. A standard steroid taper schedule is provided in the protocol as guidance for clinicians (Table 4). |
| | The primary endpoint is the response rate at 48 weeks. Response will be defined by the NIH Consensus Development Project Criteria (2014) and must occur: |
| | In the absence of new therapy for cGVHD |
| | In the absence of progression of the underlying disease that was the indication for transplant, or post-transplant lymphoproliferative disease (PTLD), or death |
| | Secondary endpoints will assess for additional clinical benefit including Week-24 response, DOR, corticosteroid dose reduction, time to withdrawal of all immunosuppressants, OS, and Lee cGVHD symptom scale. |
| | The randomization between arms will be stratified according to: |
| | • Age group (12 to <22 years old vs. ≥22 years old) |
| | NIH Global Severity grade (moderate vs. severe) |
| | Ongoing use of systemic immunosuppressants that were initiated for either treatment of or prophylaxis for acute GVHD (Yes vs. No) |
| Population: | Subjects with new onset moderate or severe cGVHD as defined<br>by the NIH Consensus Development Project Criteria<br>(Jagasia 2015) |
| | Subjects must be in need of systemic treatment for cGVHD with corticosteroids |
| Centers: | Multi-center, International |
| Inclusion Criteria: | Eligible subjects will meet all of the following criteria: 1. New onset moderate or severe cGVHD as defined by the NIH Consensus Development Project Criteria (2014, see Appendix M, Appendix N, Appendix O). |
| | 2. History of an allogeneic hematopoietic cell transplant. |
| | 3. Need for systemic treatment with corticosteroids for cGVHD. |
| | 4. No previous systemic treatment for cGVHD (including extracorporeal photopheresis [ECP]). |
| | 5. Participants may be receiving other immunosuppressants for the prophylaxis or treatment of acute GVHD but if the subject is receiving prednisone for prophylaxis or treatment of acute GVHD it must be at or below 0.5 mg/kg/d. |
| | 6. Participants may have received pre-transplant BTK inhibitors for other reasons besides cGVHD such as for the treatment of |

| | leukemia or lymphoma, but must not have received a BTK inhibitor since the time of transplant. 7. Age ≥12 years old. 8. Karnofsky or Lansky (subjects <16 years) performance score ≥60. 9. Adequate renal function defined as an estimated Creatinine Clearance ≥30 mL/min (Cockcroft-Gault formula) 10. Adequate hepatic function as defined by: • Total bilirubin of ≤ 1.5 x ULN (unless of non-hepatic origin or due to Gilbert's Syndrome) or • Total bilirubin of > 1.5 x ULN to 3.0 x ULN if due to GVHD 11. Adequate hematological function defined as: • Absolute neutrophil count ≥1.0 x 10°/L and off growth factor support for 7 days • Platelets ≥30 x 10°/L and no transfusion for 7 days 12. PT/INR <1.5 x ULN and PTT (aPTT) <1.5 x ULN (unless abnormalities are unrelated to coagulopathy or bleeding disorder). When treated with warfarin or other vitamin K antagonist, then INR ≤3.0 (Section 6.2.3). Ethical/Other 13. Male and female subjects of reproductive potential who agree to use both a highly effective methods of birth control (eg, implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], complete abstinence¹, or sterilized partner) and a barrier method (eg, condoms, cervical ring, sponge, etc.) during |
|---|---|
| | the period of therapy and for 90 days for both females and males after the last dose of study drug. |
| <b>Exclusion Criteria:</b> | Subjects are excluded if any of the following criteria are met: |
| | Received any previous systemic treatment for cGVHD with the following exception: |
| | <ul> <li>Corticosteroids for cGVHD received within the 72 hours prior to signing the informed consent form.</li> <li>Inability to begin a prednisone dose ≥0.5 mg/kg/d for the treatment of cGVHD.</li> <li>Presence of single-organ, genito-urinary involvement with cGVHD as the only manifestation of cGVHD.</li> <li>Received any investigational agent ≤28 days before randomization.</li> <li>Received donor lymphocyte infusion (DLI) ≤56 days before randomization.</li> <li>Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or Class 3 or 4 congestive heart</li> </ul> |

<sup>&</sup>lt;sup>1</sup> Complete abstinence is a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject. http://www.hma.eu/fileadmin/dateien/Human\_Medicines/01 About\_HMA/Working\_Groups/CTFG/2014\_09\_HMA\_CTFG\_Contraception.pdf

- failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization.
- 7. Any uncontrolled active systemic infection or active infection requiring systemic treatment that was ongoing ≤7 days before randomization. This does not include secondary prophylaxis of well controlled fungal infections, ongoing treatment of controlled viral reactivations (eg, CMV), or treatment or prophylaxis of controlled low-grade central line infections (eg, Staphylococcus epidermidis).
- 8. Progressive underlying malignant disease or active post-transplant lymphoproliferative disease.
- 9. History of other malignancy (not including the underlying malignancy that was the indication for transplant), with the following exceptions:
  - Malignancy treated with curative intent and with no evidence of active disease present for more than 3 years prior to Screening and felt to be at low risk for recurrence by treating physician
  - Adequately treated nonmelanomatous skin cancer or lentigo maligna melanoma without current evidence of disease
  - Adequately treated cervical carcinoma in situ without current evidence of disease
- 10. Subject has a concurrent illness which in the opinion of the investigator may interfere with the treatment and evaluation of the subject.
- 11. Known bleeding disorders (eg, von Willebrand's disease or hemophilia).
- 12. History of stroke or intracranial hemorrhage within 6 months prior to randomization.
- 13. Known history of human immunodeficiency virus (HIV).
- 14. Subject with chronic liver disease with hepatic impairment per Child-Pugh classification Class C (Appendix E). Please note that acute liver dysfunction due to cGVHD is not applicable to the evaluation of Child-Pugh classification.
- 15. Active hepatitis C virus (HCV) or hepatitis B virus (HBV). Subjects who are positive for hepatitis B core antibody or hepatitis B surface antigen or hepatitis C antibody must have a negative polymerase chain reaction (PCR) result before randomization. Those who are PCR positive will be excluded.
- 16. Vaccinated with live, attenuated vaccines within 4 weeks of randomization.
- 17. Major surgery within 4 weeks of randomization.
- 18. Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk.
- 19. Unable to swallow capsules or malabsorption syndrome, disease

| | significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction. 20. Subjects requiring treatment with a strong CYP3A inducer are not eligible, unless a transition to an agent with less CYP3A induction is planned (Appendix D). 21. Female subject who is pregnant, breastfeeding, or planning to become pregnant while enrolled in this study or within 3 months of last dose of study drug. Male subject who plans to father a child while enrolled in this study or within 3 months after the last dose of study drug. 22. Unwilling or unable to participate in all required study evaluations and procedures. 23. Unable to understand the purpose and risks of the study and to |
|---|---|
| | provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local subject privacy regulations). |
| Study Treatment: | 1:1 Randomization between Arm A and Arm B |
| · | <b>Arm A:</b> Oral ibrutinib 420 mg daily (3 capsules) in combination with oral prednisone starting at 1 mg/kg/day until unacceptable toxicity, progression of underlying disease, death, or the need for a new systemic treatment for progressive cGVHD. |
| | <b>Arm B:</b> Oral matching placebo capsules daily (3 capsules) in combination with oral prednisone starting at 1 mg/kg/day until unacceptable toxicity, progression of underlying disease, death, or the need for a new systemic treatment for progressive cGVHD. |
| Concomitant Therapy: | Refer to Section 6 for information on concomitant therapy. |
| Safety Plan: | The safety of this study will be monitored by an independent data monitoring committee (DMC) as outlined in the DMC charter and in accordance with the Sponsor's Pharmacovigilance procedures. |
| Statistical Methods: | All efficacy analyses will be performed using the intent-to-treat (ITT) population. |
| | Primary Efficacy Analysis: |
| | The primary efficacy endpoint of this study is the response rate at 48 weeks (ie, the proportion of responders [CR or PR]). Response will be defined by the NIH Consensus Development Project Criteria (2014) and must occur: |
| | <ul> <li>In the absence of new systemic therapy for cGVHD</li> <li>In the absence of progression of the underlying disease that was the indication for transplant, or death</li> </ul> |
| | Response rates will be compared between the two treatment arms using the chi-square statistical test. |
| | Secondary Efficacy Analysis: |
| | Response rate at 24 weeks (the proportion of responders [CR or PR]) as defined by the NIH Consensus Development Project |

| | <ul> <li>Duration of response (DOR)</li> <li>Steroid dose reduction to a level of less than 0.15 mg/kg/d at 24 weeks: the proportion of subjects who have steroid dose reduced by 24 weeks will be compared between the two treatment arms</li> <li>Time to withdrawal of all immunosuppressants (with the exception of ibrutinib/placebo) will be compared between the two treatment arms</li> <li>Overall survival (OS): Overall survival will be compared between the two treatment arms using the log rank test</li> <li>Improvement in Lee cGVHD symptom scale scores will be compared between the two treatment arms</li> <li>Safety Analysis:</li> <li>Safety data will be generated from the Safety Population (SP) which consists of all subjects randomized and receiving at least one dose of any study drug (ibrutinib or placebo).</li> <li>Detailed tabulations of safety data (adverse events, clinical laboratory tests and other safety endpoints) will be summarized by treatment arm for all subjects receiving study drug.</li> </ul> |
|---|---|
| Interim Analysis: | An interim review for futility will be performed for the first 50 subjects who complete Week 25 visit or discontinue study drug before this time. |
| Sample Size Determination: | The null hypothesis is that the two treatment arms have the same response rate at 48 weeks and the alternative hypothesis is that the response rates of two arms are different. Assuming a response rate of 30% at 48 weeks for Arm B (placebo + prednisone), a sample size of 186 randomized subjects provides at least an 80% power to detect a 20% difference in the response rates at 48 weeks between the 2 treatment arms (Arm A − Arm B) at an alpha level of 5% (2-sided). The randomization between arms will be stratified according to: • Age group (12 to <22 years old vs. ≥22 years old) • NIH Global Severity grade (moderate vs. severe) • Ongoing use of systemic immunosuppressants that were initiated for either treatment of or prophylaxis for acute GVHD (Yes vs. No) |

#### ABBREVIATIONS

ΑE adverse event

alanine aminotransferase ALT ANC absolute neutrophil count

aPTT activated partial thromboplastin time

American Society for Blood and Marrow Transplantation **ASBMT** 

AST aspartate aminotransferase area under the curve AUC **BAFF** B-cell activating factor

**BCR** B-cell receptor

Bruton's tyrosine kinase **BTK** 

CFR US Code of Federal Regulations chronic graft versus host disease cGVHD chronic lymphocytic leukemia CLL

CRF case report form complete response CR

Common Terminology Criteria for Adverse Events version 4.03 CTCAE v. 4.03

cytochrome P450 **CYP** 

donor lymphocyte infusion DLI data monitoring committee **DMC** Duration of response DOR **ECG** Electrocardiogram

**ECP** extracorporeal photopheresis electronic data capture **EDC** electronic medical records **EMR** Food and Drug Administration FDA forced expiratory volume in 1 second FEV1

Good Clinical Practice **GCP** 

gastrointestinal GI

GVHD graft versus host disease GVT graft versus tumor

hematopoietic cell transplantation **HCT** 

Health Insurance Portability and Accountability Act HIPAA

HIV human immunodeficiency virus **HPA** Hypothalamic-pituitary-adrenal

Investigator's Brochure IΒ

half maximal inhibitor concentration  $IC_{50}$ 

Informed consent form **ICF** 

**ICH** International Conference on Harmonization

**IEC Independent Ethics Committee** 

Immunoglobulin M **IgM** 

ILInterleukin

ILD interstitial lung disease INR international normalized ratio IRB Institutional Review Board IL-2 inducible T-cell kinase **ITK** 

ITT intention-to-treat IV Intravenous

Interactive Web Response System **IWRS KPS** Karnofsky Performance Status

MCL mantle cell lymphoma
mITT modified intention-to-treat
MZL marginal zone lymphoma
SP Safety population

MTD maximum tolerated dose
NCI National Cancer Institute
NIH National Institutes of Health

NRM non-relapse mortality
OS overall survival

PCI-32765 ibrutinib or Imbruvica®
PCR polymerase chain reaction
PCYC Pharmacyclics LLC
PD progressive disease
PK pharmacokinetic

PO oral

PR partial response

PTLD post-transplant lymphoproliferative disease

PT prothrombin time

QD daily

QOD every other day
QTc corrected QT interval
REB Research Ethics Board
SAE serious adverse event

SCARs severe cutaneous adverse reactions

SD stable disease

SF-36 36-Item Short Form Health Survey SJS Stevens - Johnson syndrome

 $t_{1/2}$  half life

TEAE(s) treatment-emergent adverse event(s)

TCR T-cell receptor tumor lysis syndrome

T<sub>max</sub> median time to maximum plasma concentration

ULN upper limit of normal
USPI United States Product Insert
VZIG varicella zoster immune globulin
WM Waldenström's macroglobulinemia

#### 1. <u>BACKGROUND</u>

# 1.1. Disease/Histology

# 1.1.1. Disease Background

Since its first report in 1957, allogeneic hematopoietic cell transplant (HCT) has become a standard therapy for many hematologic malignancies and hematopoietic progenitor cell disorders (Thomas 1957). Hematopoietic cell transplant can cure patients with chemotherapy resistant malignancies through graft versus tumor (GVT) effects generated by the donor's immune system against the recipient's tumor (Appelbaum 2001). However, just as the donor's immune system can sense and attack the recipient's malignant cells, so can it sense and attack the recipient's normal tissues resulting in graft versus host disease (GVHD). In the U.S., approximately 8,000 allogeneic HCTs are now performed each year (Pasquini 2015). Roughly 35% of patients who have undergone HCT will develop cGVHD that requires systemic treatment (Flowers 2011). The prevalence of cGVHD is increasing due to both the increased use of allogeneic transplantation in older adults and the use of peripheral stem cells as a graft source. Chronic GVHD is a serious and life threatening impediment to the otherwise curative potential of HCT (Pidala 2011, Arai 2011, Baird 2006 and Lee 2003) and it is a leading cause of non-relapse mortality (NRM) (Lee 2008). Risk factors for developing cGVHD include prior acute GVHD, older age, use of peripheral blood stem cells, use of unrelated and mismatched donors, and lack of T-cell depletion (Lee 2008).

In the past, timing of manifestations of GVHD were used to classify GVHD into two subsets, acute GVHD classified as occurring within 100 days of HCT and chronic GVHD classified as manifestations beyond 100 days after HCT (Filipovich 2005). In 2005 the National Institutes of Health (NIH) sponsored a consensus development conference that proposed new criteria for diagnosis and classification of cGVHD for clinical trials (Filipovich 2005). The consensus met again in 2014 and proposed minor changes to the diagnostic criteria (Jagasia 2015). The published criteria for diagnosis emphasize the distinction between acute and chronic GVHD as different subsets of GVHD that can be distinguished by clinical manifestations and not time after transplant. The diagnosis of cGVHD is primarily clinical and requires at least one diagnostic sign in a target organ per NIH criteria (ie, a sign found only in cGVHD) or at least one distinctive sign (ie, a sign highly suggestive of cGVHD) in combination with some other laboratory, biopsy, or other test confirmation in the same or another organ. The diagnostic cGVHD findings include collagen-vascular changes involving the skin, mouth, genitalia, gastrointestinal tract, lung, muscle fascia, and joints (Jagasia 2015) (Appendix M). Pathologically, cGVHD is characterized by fibrosis and inflammation of affected organs (Shulman 2006).

#### **Pathogenesis of Chronic Graft Versus Host Disease**

The immunopathology underlying development of cGVHD can be quite variable and is not entirely characterized. Recent information implicates B cells as well as T cells in the generation of cGVHD (Sarantopoulos 2015, Allen 2014, Flynn 2014 and Johnston 2014). T cells have long

been known to be critically important in the development of cGVHD. Higher rates of cGVHD are seen in recipients of colony-stimulating factor mobilized peripheral blood grafts compared with marrow grafts and in patients who receive a higher T cell dose (Anasetti 2011). In vivo T cell depletion with anti-thymocyte globulin or alemtuzumab can reduce the incidence of cGVHD, but at the cost of higher rates of viral or opportunistic infections and relapse of underlying disease (Hale 2012, Perez-Simon 2002). Alloreactive T helper cells, including Th1, Th2, Th17, and T follicular helper cells, produce effector cytokines resulting in antibody deposition, tissue fibrosis, and autoimmunity.

More recently, alloreactive B cells have been implicated in the development of cGVHD (Sarantopoulos 2015, Allen 2014, Flynn 2014, Johnston 2014, Miklos 2005 and Miklos 2004). In addition to the production of alloantibodies, B cells contribute to the immune response via antibody-independent processes, such as antigen presentation, cytokine and chemokine production, and immunoregulatory function (Sahaf 2013). Following activation via the B-cell receptor (BCR) signaling pathways, B cells become potent antigen-presenting cells. Activated B cells produce a variety of inflammatory cytokines, and antigen presentation by autoreactive B cells is critical in autoimmune disorders (Shimabukuro-Vornhagen 2009). Dysfunctional B cells have been identified in cGVHD, where patients have a relatively higher number of activated memory B cells, higher levels of B-cell-activating factor (BAFF) of the tumor necrosis family, and donor-derived alloantibodies (Sarantopoulos 2009).

# 1.1.2. Current Treatment Options

Available therapy for cGVHD is primarily broad-spectrum immunosuppressants which increase the risk of infections and tumor relapse by inhibiting GVT immunity (Holler 2007). The initial and current standard of care treatment for cGVHD is corticosteroids. However, more than 50% of the patients eventually relapse or become refractory, requiring second-line treatment, for which there is no standard of care. Recently, ibrutinib received approval in the United States for the treatment of adult patients with cGVHD after failure of one or more lines of systemic therapy.

Treatment with immunosuppressants is typically needed for a median duration of 2 to 3 years, further contributing to morbidity (Syrjala 2012). During that time patients are likely to experience some or all of the side effects of corticosteroids which include more frequent infections, hypertension, hyperglycemia, decrease in bone density, avascular necrosis, adrenal insufficiency, cataracts and disturbed sleep patterns (Sullivan 1988, Rayos [Prednisone] USPI 2013). Because of the frequent morbidity associated with prolonged corticosteroid use, many other immunosuppressant agents have been investigated in cGVHD, both in the front line and second line setting. Several controlled, phase 3 studies where these agents have been added on to corticosteroid therapy were all unsuccessful in providing benefit despite showing efficacy in early phase studies (Gilman 2012, Martin 2009, Koc 2002, Arora 2001, Koc 2000, and Sullivan 1988). An analysis of clinical trial quality measures in 60 trials in cGVHD primarily conducted before the NIH standardized response criteria (Pavletic 2006) were developed,

revealed that poor study design (eg, lack of rigorous entry criteria, organ response criteria and overall response criteria) likely biased efficacy in the early phase trials (Martin 2011) thereby leading to later unsuccessful controlled studies with the same agents. Agents such as cyclosporine, tacrolimus, sirolimus, and/or mycophenolate mofetil are often added to corticosteroid therapy in both frontline and second line settings despite the lack of efficacy. There is a lack of standard of care and high unmet need for new therapeutic options to effectively suppress immune and fibrotic cascades while preserving GVT and immunity against infection.

While limited progress related to prevention or treatment of cGVHD has been made, the development of the NIH Consensus Criteria for grading and staging of cGVHD represents a significant advancement, providing a clinically useful disease burden measure for use in clinical trials (Jagasia 2015). In addition, the NIH Consensus Response Criteria have been shown to correlate with clinical outcomes (Olivieri 2013, Jacobsohn 2012).

#### 1.2. Ibrutinib Overview

Ibrutinib (IMBRUVICA®) is a first-in-class, potent, orally administered, covalently binding inhibitor of Bruton's tyrosine kinase (BTK) co-developed by Pharmacyclics LLC and Janssen Research & Development LLC for the treatment of B-cell malignancies and cGVHD.

Ibrutinib has been approved in many regions, including the US and EU, for indications including treatment of patients with mantle cell lymphoma (MCL) who have received at least 1 prior therapy, patients with chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL), including CLL/SLL with a deletion of the short arm of chromosome 17 (del17p), patients with Waldenström's macroglobulinemia (WM), Marginal Zone Lymphoma (MZL) who require systemic therapy and have received at least one prior anti-CD20-based therapy, and cGVHD after failure of one or more lines of systemic therapy. For the most up to date and comprehensive nonclinical and clinical information regarding ibrutinib background, safety, efficacy, in vitro and in vivo preclinical activity, and toxicology of ibrutinib, always refer to the latest version of the ibrutinib Investigator's Brochure (IB) and/or the applicable regional labeling information.

#### 1.2.1. Summary of Nonclinical Data

#### 1.2.1.1. Pharmacology

Ibrutinib was designed as a selective and covalent inhibitor of the BTK (Pan 2007). In vitro, ibrutinib is a potent inhibitor of BTK activity (IC $_{50}$  = 0.39 nM). The irreversible binding of ibrutinib to cysteine-481 in the active site of BTK results in sustained inhibition of BTK catalytic activity and enhanced selectivity over other kinases that do not contain a cysteine at this position. When added directly to human whole blood, ibrutinib inhibits signal transduction from the BCR and blocks primary B-cell activation (IC $_{50}$  = 80 nM) as assayed by anti-IgM stimulation followed by CD69 expression (Herman 2011). In addition to BTK activity, ibrutinib inhibits ITK activity with a biochemical IC $_{50}$  of 26.9 nM. Ibrutinib also blocks T cell receptor-induced IL-2 secretion

by a T cell line (Jurkat cells) with an EC<sub>50</sub> of 200 nM. In CLL patients receiving ibrutinib, binding to ITK also has been demonstrated (Dubovsky 2013).

For more detailed and comprehensive information regarding nonclinical pharmacology and toxicology, please refer to the current IB.

#### 1.2.1.2. Safety Pharmacology and Toxicology

No treatment-related effects were observed in the central nervous system or respiratory system in rats at any dose tested. Further, no treatment-related corrected OT interval (OTc) prolongation effect was observed at any tested dose in a cardiovascular study using telemetry-monitored dogs. Based on data from rat and dog including general toxicity studies up to 13 weeks duration, the greatest potential for human toxicity with ibrutinib is predicted to be in lymphoid tissues (lymphoid depletion) and the gastrointestinal tract (soft feces/diarrhea with or without inflammation). Additional toxicity findings seen in only one species with no observed human correlate in clinical studies to date include pancreatic acinar cell atrophy (rat), minimally decreased trabecular and cortical bone (rat) and corneal dystrophy (dog). In studies in pregnant rats and rabbits, ibrutinib administration was associated with malformations (teratogenicity) at ibrutinib doses that result in approximately 14 and 2 times the exposure (area under the concentration-time curve [AUC]) in patients administered the dose of 560 mg daily, respectively. Fetal loss and reduced fetal body weights were also seen in treated pregnant animals. Carcinogenicity studies have not been conducted with ibrutinib. In vitro and in vivo genetic toxicity studies showed that ibrutinib is not genotoxic. No effects on fertility or reproductive capacities were observed in a study in male and female rats.

For the most comprehensive information regarding nonclinical safety pharmacology and toxicology, please refer to the current IB.

#### 1.2.2. Summary of Clinical Data

For the most comprehensive clinical information regarding ibrutinib, please refer to the current version of the IB.

#### 1.2.2.1. Pharmacokinetics and Product Metabolism

Following oral administration of ibrutinib at doses ranging from 420 to 840 mg/day, exposure to ibrutinib increased proportionally to doses increased with substantial intersubject variability. The mean half-life (t<sub>1/2</sub>) of ibrutinib ranged from 4 to 13 hours, with a median time to maximum plasma concentration (T<sub>max</sub>) of 2 hours. Taking into account the approximate doubling in mean systemic exposure when dosed with food and the favorable safety profile, ibrutinib can be dosed with or without food. Ibrutinib is extensively metabolized primarily by cytochrome P450 (CYP) 3A4 enzymes. The on-target effects of metabolite PCI-45227 are not considered clinically relevant. Steady-state exposure of ibrutinib and PCI-45227 was less than 2-fold of single dose exposure. Less than 1% of ibrutinib is excreted renally. Ibrutinib exposure is not

altered in patients with creatinine clearance (CrCl) >30 mL/min. Patients with severe renal impairment or patients on dialysis have not been studied. Following single dose administration, the AUC of ibrutinib increased 2.7-, 8.2- and 9.8-fold in subjects with mild (Child-Pugh class A), moderate (Child-Pugh class B), and severe (Child-Pugh class C) hepatic impairment compared to subjects with normal liver function. A higher proportion of Grade 3 or higher adverse reactions were reported in patients with B-cell malignancies (CLL, MCL and WM) with mild hepatic impairment based on NCI organ dysfunction working group (NCI-ODWG) criteria for hepatic dysfunction compared to patients with normal hepatic function. In the Phase 2 study in subjects with cGVHD, there were no differences in ibrutinib exposure between subjects with normal (n=29) and mild hepatic impairment based on baseline liver function test per NCI criteria (n=13).

For the most comprehensive information regarding pharmacokinetics (PK) and product metabolism, please refer to the current version of the IB.

# 1.2.3. Summary of Clinical Safety

A brief summary of safety data from monotherapy studies, combination therapy studies, and a cGVHD study is provided below.

# 1.2.3.1. Monotherapy Studies

Pooled safety data from a total of 1318 subjects treated with ibrutinib monotherapy in 13 studies that have completed primary analysis or final analysis as of the 31 May 2016 cutoff date for the current Investigator's Brochure update in B-cell malignancies are summarized below.

The most frequently reported treatment-emergent adverse events (TEAEs) in subjects receiving ibrutinib as monotherapy (N=1318):

| Most frequently reported TEAEs ≥15% <sup>a</sup> | Most frequently reported Grade 3 or 4 TEAEs ≥3% <sup>b</sup> | Most frequently reported Serious TEAEs ≥2% ° |
|---|---|---|
| Diarrhea | Neutropenia | Pneumonia |
| Fatigue | Pneumonia | Atrial fibrillation |
| Nausea | Thrombocytopenia | Febrile neutropenia |
| Cough | Anemia | Pyrexia |
| Pyrexia | Hypertension | |
| Anemia | Diarrhea | |
| Neutropenia | Atrial Fibrillation | |
| Upper respiratory tract infection | | |
| Thrombocytopenia | | |
| Oedema peripheral | | |

<sup>&</sup>lt;sup>a</sup> Source is Table 6 of IB (v10), <sup>b</sup> Source is Table 8 of IB (v10), <sup>c</sup> Source is Table 9 of IB (v10).

#### 1.2.3.2. Combination Studies

Pooled safety data from a total of 423 subjects treated with various therapies in combination with ibrutinib from 4 studies conducted in subjects with B-cell malignancies are briefly summarized below. Therapies used in combination with ibrutinib in these studies, included BR (bendamustine and rituximab), FCR (fludarabine, cyclophosphamide, and rituximab), ofatumumab, and R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone).

The most frequently reported TEAEs in subjects receiving ibrutinib in combination therapy (N=423):

| Most frequently reported TEAEs ≥20% <sup>a</sup> | Most frequently reported Grade 3 or 4 TEAEs ≥3% <sup>b</sup> | Most frequently reported<br>Serious TEAEs ≥2% <sup>c</sup> |
|---|---|---|
| Neutropenia | Neutropenia | Pneumonia |
| Diarrhea | Thrombocytopenia | Febrile neutropenia |
| Nausea | Febrile neutropenia | Atrial fibrillation |
| Thrombocytopenia | Pneumonia | Pyrexia |
| Fatigue | Neutrophil count decreased | Cellulitis |
| Anemia | Anemia | |
| Pyrexia | Fatigue | |
| | Hypertension | |
| | Diarrhea | |

<sup>&</sup>lt;sup>a</sup> Source is Table 10 of IB (v10), <sup>b</sup> Source is Table 12 of IB (v10), <sup>c</sup> Source is Table 13 of IB (v10).

#### 1.2.3.3. Chronic GVHD Study

Safety data from the 42 subjects enrolled in the PCYC-1129-CA study demonstrated that 100% of subjects have experienced a treatment-emergent adverse event (TEAE) with a total of 73.8% of subjects reported Grade 3 or higher AEs. Fifty-two percent (52.4%) of subjects reported serious adverse events (SAEs). The most frequent TEAEs and SAEs are summarized below.

Most frequently reported TEAEs in subjects receiving ibrutinib for cGVHD (N=42):

| Most frequently reported TEAEs > 20% | Most frequently reported<br>Grade 3 or 4 TEAEs > 10% | Serious TEAEs occurred in > 1 subject |
|---|---|---|
| Fatigue | Fatigue | Cellulitis |
| Diarrhea | Pneumonia | Headache |
| Muscle spasms | | Pneumonia |
| Nausea | | Pyrexia |
| Increased tendency to bruise | | Septic shock |

Thirty subjects (71.4%) were taking moderate or strong CYP3A inhibitors during the study with 9.5% of subjects taking posaconazole, 42.9% taking fluconazole, and 14.3% taking voriconazole.

Concomitant use of moderate and strong CYP3A inhibitors resulted in higher ibrutinib exposure but there was no association between concurrent CYP3A inhibitor use and dose reductions or discontinuations or with TEAEs leading to dose reductions or discontinuations.

#### 1.2.4. **Risks**

#### 1.2.4.1. Atrial Fibrillation

Atrial fibrillation and atrial flutter have been reported in subjects treated with ibrutinib, particularly in subjects with cardiac risk factors, hypertension, acute infections, and a previous history of atrial fibrillation. Subjects who develop arrhythmic symptoms (eg, palpitations, lightheadedness) or new onset dyspnea should be evaluated clinically, and if indicated, have an ECG performed. For atrial fibrillation which persists, consider the risks and benefits of ibrutinib treatment and follow the protocol dose modification guidelines (see Section 5.3.1.4).

# 1.2.4.2. Bleeding-related Events

There have been reports of hemorrhagic events in subjects treated with ibrutinib, both with and without thrombocytopenia. These include minor hemorrhagic events such as contusion, epistaxis, and petechiae; and major hemorrhagic events, some fatal, including gastrointestinal bleeding, subdural intracranial hemorrhage, and hematuria. Use of ibrutinib in subjects requiring other anticoagulants or medications that inhibit platelet function may increase the risk of bleeding. Subjects with congenital bleeding diathesis have not been studied. See Section 6.2.3 for guidance on concomitant use of anticoagulants, antiplatelet therapy and/or supplements. See Section 6.4 for guidance on ibrutinib management with surgeries or procedures. In an in vitro platelet function study, inhibitory effects of ibrutinib on collagen induced platelet aggregation were observed, refer to Section 6.2.3.

#### 1.2.4.3. Cytopenias

Treatment-emergent Grade 3 or 4 cytopenias (neutropenia, thrombocytopenia, and anemia) were reported in subjects treated with ibrutinib. Subjects should be monitored for fever, weakness, or easy bruising and/or bleeding.

#### **1.2.4.4.** Diarrhea

Diarrhea is the most frequently reported non-hematologic AE with ibrutinib monotherapy and combination therapy. Other frequently reported gastrointestinal events include nausea, vomiting, and constipation. These events are rarely severe. Should symptoms be severe or prolonged follow the protocol dose modification guidelines (see Section 5.3.1.4).

#### 1.2.4.5. Infections

Infections (including sepsis, bacterial, viral, aspergillus or other fungal infections) were observed in subjects treated with ibrutinib therapy. Some of these reported infections have been associated

with hospitalization and death. Consider prophylaxis according to standard of care in subjects who are at increased risk for opportunistic infections (see Section 6.1). Although causality has not been established, cases of progressive multifocal leukoencephalopathy (PML) have occurred in subjects treated with ibrutinib. Subjects should be monitored for symptoms (fever, chills, weakness, confusion) and appropriate therapy should be instituted as indicated.

# 1.2.4.6. Interstitial Lung Disease (ILD)

Cases of interstitial lung disease (ILD) have been reported in subjects treated with ibrutinib. Monitor subjects for pulmonary symptoms indicative of ILD. Should symptoms develop follow the protocol dose modification guidelines (see Section 5.3.1.4).

#### 1.2.4.7. Non-melanoma Skin Cancer

Non-melanoma skin cancers have occurred in subjects treated with ibrutinib. Monitor subjects for the appearance of non-melanoma skin cancer.

#### 1.2.4.8. Rash

Rash has been commonly reported in subjects treated with either single agent ibrutinib or in combination with chemotherapy. Most rashes were mild to moderate in severity. Isolated cases of severe cutaneous adverse reactions (SCARs) including Stevens - Johnson syndrome (SJS) have been reported in subjects treated with ibrutinib. Subjects should be closely monitored for signs and symptoms suggestive of SCAR including SJS. Subjects receiving ibrutinib should be observed closely for rashes and treated symptomatically, including interruption of the suspected agent as appropriate. In addition, hypersensitivity-related events including erythema, urticaria, and angioedema have been reported.

#### 1.2.4.9. Hypertension

Hypertension has been commonly reported in subjects treated with ibrutinib. Monitor subjects for new onset of hypertension or hypertension that is not adequately controlled after starting ibrutinib. Adjust existing anti-hypertensive medications and/or initiate anti-hypertensive treatment as appropriate.

# 1.2.5. Summary of Clinical Data in Chronic GVHD

A Phase 1b/2 study (PCYC-1129-CA) to evaluate the safety and efficacy of ibrutinib treatment in subjects with cGVHD who had failed steroid therapy was initiated in June 2014. The NIH Consensus Panel Response Assessment 2005 was used to determine overall response. As of 01 September 2016, 42 subjects have been recruited and received at least one dose of study drug in the study. The median age is 56 years (19-74 years) with a median duration of GVHD of 13.6 months prior to study entry. The median number of prior therapeutic regimens is 2.0. Thirty-seven subjects have had a response assessment and 5 subjects discontinued prior to the first response assessment. Of the 42 subjects with response assessments or who discontinued

ibrutinib prior to response assessment, 28 subjects are responders (ORR=67%) based on NIH response criteria. Best responses include 9 CRs, 19 PRs, 7 stable disease (SD), 2 progressive disease (PD), and 5 unknown due to the early discontinuation of study drug without post baseline efficacy assessment. Twenty of the 28 responders (71%) achieved a sustained response for at least 20 weeks. Median corticosteroid dose in responding subjects was 0.29 mg/kg/d at baseline, 0.24 mg/kg/d at Week 12, 0.19 mg/kg/d at Week 24, 0.18 mg/kg/d at Week 36, and 0.13 mg/kg/d at Week 48. Five subjects were able to discontinue steroids. Overall response rate results were supported by exploratory analyses of patient-reported symptom bother which showed at least a 7-point decrease in Lee Symptom Scale overall summary score in 24% (10/42) of patients on at least 2 consecutive visits.

These efficacy results are consistent with a response rate and durability that is considered clinically compelling in this high-risk population and with an acceptable safety profile. Based on data from the PCYC-1129 study the US FDA approved ibrutinib for the treatment of adult patients with cGVHD after failure of one or more lines of systemic therapy.

#### 1.3. Prednisone

Prednisone is a glucocorticoid. Glucocorticoids are adrenocortical steroids (corticosteroids), both naturally occurring and synthetic, which are readily absorbed from the gastrointestinal tract. The chemical name for prednisone is pregna-1,4-diene-3,11,20-trione monohydrate,17,21-dihydroxy. Naturally occurring glucocorticoids (hydrocortisone and cortisone), which also have salt-retaining properties, are used as replacement therapy in adrenocortical deficiency states. Their synthetic analogs are primarily used for their potent anti-inflammatory effects in disorders of many organ systems. Glucocorticoids cause profound and varied metabolic effects. In addition, they modify the body's immune responses to diverse stimuli.

# 1.3.1. Summary of Clinical Data

Prednisone is a corticosteroid indicated in the following conditions:

- As an anti-inflammatory or immunosuppressive agent for certain allergic, dermatologic, gastrointestinal, hematologic, ophthalmologic, nervous system, renal, respiratory, rheumatologic, specific infectious diseases or conditions and organ transplantation
- For the treatment of certain endocrine conditions
- For palliating of certain malignant conditions

# 1.3.2. Summary of Clinical Safety

# **Alterations in Endocrine Function**

Hypothalamic-pituitary-adrenal (HPA) axis suppression, Cushing's syndrome, and hyperglycemia. Monitor patients for these conditions with chronic use.

Corticosteroids can produce reversible HPA axis suppression with the potential for corticosteroid insufficiency after withdrawal of treatment. Drug-induced secondary adrenocortical insufficiency may be minimized by gradual reduction of dosage. This type of relative insufficiency may persist for months after discontinuation of therapy; therefore, in any situation of stress occurring during that period, hormone therapy should be reinstituted. If the patient is receiving corticosteroids already, dosage may have to be increased.

Since mineralocorticoid secretion may be impaired, salt and/or a mineralocorticoid should be administered concurrently. Mineralocorticoid supplementation is of particular importance in infancy.

Metabolic clearance of corticosteroids is decreased in hypothyroid patients and increased in hyperthyroid patients. Changes in thyroid status of the patient may necessitate adjustment in dosage.

### **Increased Risks Related to Infection**

Corticosteroids may increase the risks related to infections with any pathogen, including viral, bacterial, fungal, protozoan, or helminthic infections. The degree to which the dose, route and duration of corticosteroid administration correlates with the specific risks of infection is not well characterized, however, with increasing doses of corticosteroids, the rate of occurrence of infectious complications increases.

Corticosteroids may mask some signs of infection and may reduce resistance to new infections.

Corticosteroids may exacerbate infections and increase risk of disseminated infections.

The use of prednisone in active tuberculosis should be restricted to those cases of fulminating or disseminated tuberculosis in which the corticosteroid is used for management of the disease in conjunction with an appropriate anti-tuberculous regimen.

Chickenpox and measles can have a more serious or even fatal course in non-immune children or adults on corticosteroids. In children or adults who have not had these diseases, particular care should be taken to avoid exposure. If a patient is exposed to chickenpox, prophylaxis with varicella zoster immune globulin (VZIG) may be indicated. If patient is exposed to measles, prophylaxis with pooled intramuscular immunoglobulin (IG) may be indicated. If chickenpox develops, treatment with antiviral agents may be considered.

Corticosteroids should be used with great care in patients with known or suspected Strongyloides (threadworm) infestation. In such patients, corticosteroid-induced immunosuppression may lead to Strongyloides hyperinfection and dissemination with widespread larval migration, often accompanied by severe enterocolitis and potentially fatal gram-negative septicemia.

Corticosteroids may exacerbate systemic fungal infections and therefore should not be used in the presence of such infections unless they are needed to control drug reactions.

Corticosteroids may increase risk of reactivation or exacerbation of latent infection.

If corticosteroids are indicated in patients with latent tuberculosis or tuberculin reactivity, close observation is necessary as reactivation of the disease may occur. During prolonged corticosteroid therapy, these patients should receive chemoprophylaxis.

Corticosteroids may activate latent amebiasis. Therefore, it is recommended that latent amebiasis or active amebiasis be ruled out before initiating corticosteroid therapy in any patient who has spent time in the tropics or any patient with unexplained diarrhea.

Corticosteroids should not be used in cerebral malaria.

#### Alterations in Cardiovascular/Renal Function

Corticosteroids can cause elevation of blood pressure, salt, and water retention, and increased excretion of potassium and calcium. These effects are less likely to occur with the synthetic derivatives except when used in large doses. Dietary salt restriction and potassium supplementation may be necessary. These agents should be used with caution in patients with congestive heart failure, hypertension, or renal insufficiency.

Literature reports suggest an apparent association between use of corticosteroids and left ventricular free wall rupture after a recent myocardial infarction; therefore, therapy with corticosteroids should be used with great caution in these patients.

#### **Use in Patients with Gastrointestinal Disorders**

There is an increased risk of gastrointestinal perforation in patients with certain GI disorders. Signs of GI perforation, such as peritoneal irritation may be masked in patients receiving corticosteroids.

Corticosteroids should be used with caution if there is a probability of impending perforation, abscess, or other pyogenic infections; diverticulitis; fresh intestinal anastomoses; and active or latent peptic ulcer.

# **Behavioral and Mood Disturbances**

Corticosteroids use may be associated with central nervous system effects ranging from euphoria, insomnia, mood swings, personality changes, and severe depression, to frank psychotic manifestations. Also, existing emotional instability or psychotic tendencies may be aggravated by corticosteroids.

#### **Decrease in Bone Density**

Corticosteroids decrease bone formation and increase bone resorption both through their effect on calcium regulation (ie, decreasing absorption and increasing excretion) and inhibition of osteoblast function. This, together with a decrease in the protein matrix of the bone secondary to an increase in protein catabolism, and reduced sex hormone production, may lead to inhibition of bone growth in children and adolescents and the development of osteoporosis at any age. Special consideration should be given to patients at increased risk of osteoporosis (ie, postmenopausal women) before initiating corticosteroid therapy and bone density should be monitored in patients on long term corticosteroid therapy.

# **Ophthalmic Effects**

Prolonged use of corticosteroids may produce posterior subcapsular cataracts, glaucoma with possible damage to the optic nerves, and may enhance the establishment of secondary ocular infections due to fungi or viruses.

The use of oral corticosteroids is not recommended in the treatment of optic neuritis and may lead to an increase in the risk of new episodes.

Intraocular pressure may become elevated in some individuals. If corticosteroid therapy is continued for more than 6 weeks, intraocular pressure should be monitored.

Corticosteroids should be used cautiously in patients with ocular herpes simplex because of possible corneal perforation. Corticosteroids should not be used in active ocular herpes simplex.

# **Vaccination**

Administration of live or live, attenuated vaccines is contraindicated in patients receiving immunosuppressive doses of corticosteroids. Killed or inactivated vaccines may be administered; however, the response to such vaccines cannot be predicted. Immunization procedures may be undertaken in patients who are receiving corticosteroids as replacement therapy, eg, for Addison's disease.

While on corticosteroid therapy, patients should not be vaccinated against smallpox. Other immunization procedures should not be undertaken in patients who are on corticosteroids, especially on high dose, because of possible hazards of neurological complications and a lack of antibody response.

#### **Effect on Growth and Development**

Long-term use of corticosteroids can have negative effects on growth and development in children.

Growth and development of pediatric patients on prolonged corticosteroid therapy should be carefully monitored.

# **Use in Pregnancy**

Prednisone can cause fetal harm when administered to a pregnant woman. Human and animal studies suggest that use of corticosteroids during the first trimester of pregnancy is associated with an increased risk of orofacial clefts, intrauterine growth restriction, and decreased birth weight. If this drug is used during pregnancy, or if the patient becomes pregnant while using this drug, the patient should be apprised of the potential hazard to the fetus.

# **Neuromuscular Effects**

Although controlled clinical trials have shown corticosteroids to be effective in speeding the resolution of acute exacerbations of multiple sclerosis, they do not show that they affect the ultimate outcome or natural history of the disease. The studies do show that relatively high doses of corticosteroids are necessary to demonstrate a significant effect.

An acute myopathy has been observed with the use of high doses of corticosteroids, most often occurring in patients with disorders of neuromuscular transmission (eg, myasthenia gravis), or in patients receiving concomitant therapy with neuromuscular blocking drugs (eg, pancuronium). This acute myopathy is generalized, may involve ocular and respiratory muscles, and may result in quadriparesis. Elevation of creatine kinase may occur. Clinical improvement or recovery after stopping corticosteroids may require weeks to years.

#### Kaposi's Sarcoma

Kaposi's sarcoma has been reported to occur in patients receiving corticosteroid therapy, most often for chronic conditions. Discontinuation of corticosteroids may result in clinical improvement.

#### 1.3.3. Summary of Clinical Data in Chronic Graft versus Host Disease

Corticosteroids have been the backbone of treatment of cGVHD for more than 3 decades despite few formal trials to document its efficacy (Flowers 2015, Wolff 2011, Dignan 2012). While effective, prolonged administration of systemic corticosteroids results in substantial morbidity including hypertension, bone loss, weight gain, diabetes, cataracts, and myopathy as well as increasing the risk for underlying malignancy. The administration of alternate day steroids is often attempted to mitigate the risk of these toxicities. In addition, rapid corticosteroid taper and discontinuation is preferred in cGVHD.

#### 1.4. Study Rationale

While corticosteroids are effective in some patients, until the approval of ibrutinib in August 2017 for adult patients with cGHVD after failure of one or more lines of systemic therapy, there

had been no approved therapies for cGVHD as no other immunosuppressant therapy has proven to be effective either in front-line or steroid refractory cGVHD patients. Pre-clinical results have demonstrated a substantial therapeutic benefit of ibrutinib treatment to reduce the prolonged alloimmune effects of cGVHD in animal models and supported investigation in clinical studies. Data supporting the approval of ibrutinib in cGVHD demonstrated that ibrutinib has robust clinical activity with high response rate by NIH criteria as well as an overall favorable safety profile. These data also support the continued clinical evaluation of ibrutinib in combination with prednisone as a treatment option for patients with new onset cGVHD.

# 2. <u>STUDY OBJECTIVES</u>

# 2.1. Primary Objective

To evaluate the efficacy of ibrutinib in combination with prednisone (Arm A) versus placebo in combination with prednisone (Arm B) based on the response rate at 48 weeks (the proportion of responders [CR or PR]) as determined by NIH Consensus Development Project Criteria in subjects with new onset moderate to severe cGVHD (Lee 2015, Jagasia 2015).

# 2.2. Secondary Objective(s)

• To compare the two treatment arms in terms of the following:

# **Efficacy**

- Response rate at 24 weeks (the proportion of responders [CR or PR]) as defined by the NIH Consensus Development Project (2014)
- Duration of response (DOR)
- Proportion of subjects obtaining a steroid dose level less than 0.15 mg/kg/d at 24 weeks
- Time to withdrawal of all immunosuppressants (with the exception of ibrutinib/placebo)
- Overall survival (OS)
- Lee cGVHD symptom scale improvement

# Safety

- Safety and tolerability
- Differences in steroid-related morbidities (eg, hyperglycemia, hypertension)

# 2.3. Exploratory Objective(s)

- Pharmacokinetics of ibrutinib when administered in combination with prednisone in subjects with cGVHD including adolescent subjects
- Pharmacodynamic characteristics of ibrutinib (including BTK and ITK occupancy) in subjects with cGVHD

- Evaluation of biomarkers relevant to disease biology and therapy with ibrutinib for cGVHD
- Improvement in SF-36 patients reported outcome

# 3. <u>STUDY DESIGN</u>

# 3.1. Overview of Study Design

This is a Phase 3, multicenter, international, randomized, double-blind study of oral ibrutinib in combination with prednisone versus placebo in combination with prednisone in subjects with new onset chronic GVHD.

Approximately 186 subjects with newly diagnosed moderate or severe cGVHD, as defined by the 2014 NIH Consensus Development Project Criteria, will be randomized in a 1:1 ratio to receive either ibrutinib in combination with prednisone (Arm A) or placebo in combination with prednisone (Arm B). It is expected that a minimum of 6 subjects in the adolescent group (≥12 and < 22 years of age) will be enrolled.

Treatment with ibrutinib/placebo will be administered continuously until unacceptable toxicity, progression of the underlying disease, death, or the start of a new systemic treatment for cGVHD. Progression of the underlying disease will be defined using standard consensus criteria for the individual malignancy.

Corticosteroid therapy will be tapered as per a standard taper regimen with the goal of reducing exposure to high-moderate dose corticosteroids as quickly as possible according to clinical severity of cGVHD. A standard corticosteroid taper schedule is provided in the protocol as guidance to clinicians (Table 4).

The primary endpoint is the response rate at 48 weeks. Response will be defined by the NIH Consensus Development Project Criteria (2014) and must occur:

- In the absence of new therapy for cGVHD
- In the absence of progression of the underlying disease that was the indication for transplant, or PTLD, or death

Secondary endpoints will assess for additional clinical benefit including Week-24 response, duration of response (DOR), corticosteroid dose reduction, time to withdrawal of all immunosuppressants, OS, and Lee cGVHD symptom scale. Corticosteroid reduction will be determined by a proportion of patients who are on < 0.15 mg/kg of prednisone at week 24, to allow for variations in corticosteroid taper that occur in practice, while at the same time reaching a dose that minimizes the toxicity associated with steroids.

The randomization between arms will be stratified according to:

- Age group (12 to <22 years old vs. ≥22 years old)
- NIH Global Severity grade (moderate vs. severe)
- Ongoing use of systemic immunosuppressants that were initiated for either treatment of or prophylaxis for acute GVHD (Yes vs. No)

The rationale for the study concept is provided in Section 1.4.

# 3.1.1. Study Schema



# 4. <u>SUBJECT SELECTION</u>

#### 4.1. Inclusion Criteria

Prior to randomization, each potential subject must satisfy all of the following inclusion criteria.

#### Disease Related

- 1. New onset moderate or severe cGVHD as defined by the NIH Consensus Development Project Criteria (2014, see Appendix M, Appendix N, and Appendix O).
- 2. History of an allogeneic hematopoietic cell transplant.
- 3. Need for systemic treatment with corticosteroids for cGVHD.
- 4. No previous systemic treatment for cGVHD (including extracorporeal photopheresis [ECP]).
- 5. Participants may be receiving other immunosuppressants for the prophylaxis or treatment of acute GVHD but if the subject is receiving prednisone for prophylaxis or treatment of acute GVHD it must be at or below 0.5 mg/kg/d.
- 6. Participants may have received pre-transplant BTK inhibitors for other reasons besides cGVHD such as for the treatment of leukemia or lymphoma, but must not have received a BTK inhibitor since the time of transplant.

# Demographic

- 7. Age  $\geq$ 12 years old.
- 8. Karnofsky or Lansky (subjects <16 years) performance status ≥60.

#### Laboratory

- 9. Adequate renal function defined as estimated Creatinine Clearance ≥30 mL/min (Cockcroft-Gault formula)
- 10. Adequate hepatic function as defined by:
  - Total bilirubin of  $\leq$  1.5 x ULN (unless of non-hepatic origin or due to Gilbert's Syndrome) or
  - Total bilirubin of > 1.5 x ULN to 3.0 x ULN if due to GVHD
- 11. Adequate hematological function defined as:
  - Absolute neutrophil count  $\ge 1.0 \times 10^9$ /L and off growth factor support for 7 days
  - Platelets  $\ge 30 \times 10^9$ /L and no transfusion for 7 days
- 12. PT/INR <1.5 x ULN and PTT (aPTT) <1.5 x ULN (unless abnormalities are unrelated to coagulopathy or bleeding disorder). When treated with warfarin or other vitamin K antagonist, then INR  $\leq$ 3.0 (Section 6.2.3).

#### Ethical/Other

13. Male and female subjects of reproductive potential who agree to use both a highly effective methods of birth control (eg, implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], complete abstinence<sup>2</sup>, or sterilized partner) and a barrier method (eg, condoms, cervical ring, sponge, etc.) during the period of therapy and for 90 days for both females and males after the last dose of study drug.

#### 4.2. Exclusion Criteria

To be enrolled in the study, potential subjects must meet NONE of the following exclusion criteria:

#### Disease-Related

- 1. Received any previous systemic treatment for cGVHD with the following exception:
  - Corticosteroids for cGVHD received within the 72 hours prior to signing the informed consent form.
- 2. Inability to begin a prednisone dose  $\geq 0.5$  mg/kg/d for the treatment of cGVHD.
- 3. Presence of single-organ, genito-urinary involvement with cGVHD as the only manifestation of cGVHD.

#### Concurrent Conditions

- 4. Received any investigational agent ≤28 days before randomization.
- 5. Received donor lymphocyte infusion (DLI) ≤56 days before randomization.
- 6. Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization.
- 7. Any uncontrolled active systemic infection or active infection requiring systemic treatment that was ongoing ≤7 days before randomization. This does not include secondary prophylaxis of well controlled fungal infections, ongoing treatment of controlled viral reactivations (eg, CMV), or treatment or prophylaxis of controlled low-grade central line infections (eg, Staphylococcus epidermidis).
- 8. Progressive underlying malignant disease or active post-transplant lymphoproliferative disease.
- 9. History of other malignancy (not including the underlying malignancy that was the indication for transplant), with the following exceptions:

<sup>&</sup>lt;sup>2</sup> Complete abstinence is a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject. http://www.hma.eu/fileadmin/dateien/Human\_Medicines/01
About HMA/Working Groups/CTFG/2014\_09\_HMA\_CTFG\_Contraception.pdf

- Malignancy treated with curative intent and with no evidence of active disease present for more than 3 years prior to Screening and felt to be at low risk for recurrence by treating physician
- Adequately treated nonmelanomatous skin cancer or lentigo maligna melanoma without current evidence of disease
- Adequately treated cervical carcinoma in situ without current evidence of disease
- 10. Subject has a concurrent illness which in the opinion of the investigator may interfere with the treatment and evaluation of the subject.
- 11. Known bleeding disorders (eg, von Willebrand's disease or hemophilia).
- 12. History of stroke or intracranial hemorrhage within 6 months prior to randomization.
- 13. Known history of human immunodeficiency virus (HIV).
- 14. Subjects with chronic liver disease with hepatic impairment per Child-Pugh classification Class C (Appendix E). Please note that acute liver dysfunction due to cGVHD is not applicable to the evaluation of Child-Pugh classification.
- 15. Active hepatitis C virus (HCV) or hepatitis B virus (HBV). Subjects who are positive for hepatitis B core antibody or hepatitis B surface antigen or hepatitis C antibody must have a negative polymerase chain reaction (PCR) result before randomization. Those who are PCR positive will be excluded.
- 16. Vaccinated with live, attenuated vaccines within 4 weeks of randomization.
- 17. Major surgery within 4 weeks of randomization.
- 18. Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk.
- 19. Unable to swallow capsules or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction.
- 20. Subjects requiring treatment with a strong CYP3A inducer are not eligible, unless a transition to an agent with less CYP3A induction is planned (Appendix D).
- 21. Female subject who is pregnant, breastfeeding, or planning to become pregnant while enrolled in this study or within 3 months of last dose of study drug. Male subject who plans to father a child while enrolled in this study or within 3 months after the last dose of study drug.
- 22. Unwilling or unable to participate in all required study evaluations and procedures.
- 23. Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local subject privacy regulations).

# 5. TREATMENT OF SUBJECTS

# 5.1. Treatment Allocation and Blinding

#### **5.1.1.** Randomized Double-blind Phase

After the subject provides informed consent on study, site personnel will register the subject in Interactive Web Response System (IWRS) to assign a screening number. After the subject has completed all screening procedures and has met all requirements of the inclusion/exclusion criteria, the site personnel will update IWRS and answer key questions to randomize the subject, and have drug assigned. The first dose of ibrutinib/placebo must be administered after randomization, which should be no more than 72 hours (3 days) after the subject has been randomized by IWRS.

Approximately 186 subjects will be randomized in a 1:1 ratio to each of the 2 treatment arms.

Treatment Arm A: ibrutinib in combination with prednisone

Treatment Arm B: placebo in combination with prednisone

The randomization between arms will be stratified according to:

- Age group (12 to <22 years old vs. ≥22 years old)
- NIH Global Severity grade (moderate vs. severe)
- Ongoing use of systemic immunosuppressants that were initiated for either treatment of or prophylaxis for acute GVHD (yes vs. no)

# **5.1.1.1.** Blinding

This is a double-blind study; therefore, the subjects, the investigators, and the Sponsor's study team members will be blinded to the treatment assignment. The investigator will not be provided with randomization codes. The codes will be maintained within the IWRS, which has the functionality to allow the investigator to break the blind for an individual subject if necessary to appropriately manage or treat the subject. Data that may potentially unblind the treatment assignment (ie, study drug plasma concentrations) will be handled with special care to ensure that the integrity of the blind is maintained and the potential for bias is minimized.

The investigator should contact the Sponsor or its designee to discuss the particular situation before breaking the blind whenever possible. Telephone contact with the Sponsor or its designee will be available 24 hours per day, 7 days per week. In the event the blind is broken, the Sponsor must be informed as soon as possible. The date, time, and reason for the unblinding must be documented in IWRS in the appropriate section of the eCRF and in the source document. The IWRS confirmation indicating the code break must be retained with the subject's source documents in a secure manner. A subject whose treatment assignment has been unblinded may continue the study treatment if the subject is expected to continue receiving clinical benefit. The

subject should continue to return for scheduled study visits. The single-blind (ie, subject remains blinded to treatment assignment) should be maintained provided the subject's safety is not compromised.

At the time of the futility analyses, the randomization codes and, if required, the translation of randomization codes into treatment and control groups will be disclosed to those authorized and only for those subjects included in the interim analyses.

#### 5.2. Study Treatment

**Ibrutinib** (420 mg) or placebo will be given orally once daily continuously starting on Week 1 Day 1 until cGVHD progression, progression of underlying malignancy, subject begins another systemic treatment for cGVHD or unacceptable toxicity.

**Prednisone** 1 mg/kg/d will be given orally once daily continuously starting on Week 1 Day 1 until unacceptable toxicity or until subject is successfully tapered from the prednisone (see Section 5.3.2.2.1). Starting prednisone dose may be as low as 0.5 mg/kg/d if a subject cannot tolerate higher doses.

During Screening, prednisone to treat cGVHD may be started prior to randomization if the clinical condition of the subject necessitates it. If a subject is started on high dose prednisone for treatment of cGVHD prior to randomization, the patient must be randomized within 7 days of starting high dose prednisone.

# **5.3.** Study Medication

#### 5.3.1. Ibrutinib/Placebo

# **5.3.1.1.** Formulation/Packaging/Storage

Ibrutinib capsules are provided as a hard gelatin capsule containing 70 mg and 140 mg of ibrutinib. All formulation excipients are compendial and are commonly used in oral formulations. Refer to the ibrutinib IB for a list of excipients. 70 mg capsules will only be used for subjects who have dose reductions that require a dose of 70 mg and will not be used to constitute a dose larger than 70 mg (eg, 2 x 70 mg capsules to give 140 mg).

The ibrutinib (or placebo) capsules will be packaged in opaque high-density polyethylene plastic bottles with labels bearing the appropriate label text as required by governing regulatory agencies. All study drug will be dispensed in child-resistant packaging.

Refer to the Pharmacy Manual/site investigational product manual for additional guidance on study drug storage, preparation and handling.

Study drug labels will contain information to meet the applicable regulatory requirements.
#### **5.3.1.2.** Dose and Administration

Ibrutinib or placebo is administered orally once daily. It is expected that many subjects commencing therapy with high dose prednisone will require anti-fungal prophylaxis. Please see Section 6.2.1 for dose modification guidelines with concomitant use of CYP3A inhibitors or inducers

The capsules are to be taken around the same time each day with 8 ounces (approximately 240 mL) of water. The capsules should be swallowed intact and subjects should not attempt to open capsules or dissolve them in water. If a dose is not taken at the scheduled time, it can be taken as soon as possible on the same day with a return to the normal schedule the following day. The subject should not take extra capsules to make up the missed dose.

The first dose will be delivered in the clinic on Day 1, after which subsequent dosing is typically on an outpatient basis. Ibrutinib will be dispensed to subjects in bottles at each visit. Unused ibrutinib dispensed during previous visits must be returned to the site and drug accountability records (Section 12.8) updated at each visit. Returned capsules must not be redispensed to anyone.

#### **5.3.1.3.** Overdose

Any dose of study drug administered in excess of 420 mg is considered to be an overdose. Signs and symptoms of an overdose that meet any SAE criterion must be reported as a SAE in the appropriate time frame and documented as clinical sequelae to an overdose.

There is no specific experience in the management of ibrutinib overdose in patients. No maximum tolerated dose (MTD) was reached in the Phase 1 study in which subjects received up to 12.5 mg/kg/day (1400 mg/day). Healthy subjects were exposed up to single dose of 1680 mg. One healthy subject experienced reversible Grade 4 hepatic enzyme increases (AST and ALT) after a dose of 1680 mg. Subjects who ingested more than the recommended dosage should be closely monitored and given appropriate supportive treatment.

Refer to Section 11.4 for further information regarding AE reporting.

## **5.3.1.4.** Dose Modification for Adverse Reactions

The dose of ibrutinib/placebo must be modified according to the dose modification guidance in Table 1 and Table 2 if any of the following toxicities occur:

- Grade 4 neutropenia (ANC  $<500/\mu$ L) for more than 7 days. See Section 6.1 for instructions regarding the use of growth factor support
- Grade 3 thrombocytopenia (platelets  $<50,000/\mu$ L) in the presence of clinically significant bleeding events
- Grade 4 thrombocytopenia (platelets <25,000/μL)

- Grade 3 or 4 nausea, vomiting, or diarrhea if persistent, despite optimal anti-emetic and/or anti-diarrheal therapy
- Any other Grade 4 or unmanageable Grade 3 toxicity

Adverse events that are considered related to concomitant high dose corticosteroids (eg, hyperglycemia, insomnia) do not require dose modification or holding of ibrutinib. For Grade 3 or 4 atrial fibrillation or persistent atrial fibrillation of any grade, consider the risks and benefits of ibrutinib treatment. *If clinically indicated, the use of anticoagulants or antiplatelet agents may be considered for the thromboprophylaxis of atrial fibrillation* (Section 6.2.3).

For other AEs not listed above, including Grade 2 AEs that are deemed per the investigator potentially manageable by dose reduction, these can be managed with a one dose level reduction.

In the event that the investigator feels deviation from the recommendations above is required, please consult the medical monitor to discuss for approval.

If the dose of ibrutinib/placebo is reduced for an adverse event, at the investigator's discretion, the dose of ibrutinib may be re-escalated after 4 weeks of a dose reduction in the absence of a recurrence of the toxicity that led to the reduction. Dose changes must be recorded in the Dose Administration eCRF.

Table 1. Ibrutinib/Placebo Dose Modifications

| Occurrence | Action to be Taken |
|---|---|
| First | Withhold study drug until recovery to Grade ≤1 or baseline; may restart at original dose level |
| Second | Withhold study drug until recovery to Grade ≤1 or baseline; may restart at 1 dose level lower (eg, 280 mg/day for 420 mg/day dose) |
| Third | Withhold study drug until recovery to Grade ≤1 or baseline; may restart at 1 dose level lower (eg, 140 mg/day for 420 mg/day dose) |
| Fourth | Discontinue study drug |

Table 2. Ibrutinib/Placebo Dose Reduction Levels

| Starting Dose Level | 420 mg | 280 mg | 140 mg |
|------------------------|-------------|-------------|-------------|
| Dose Reduction Level 1 | 280 mg | 140 mg | 70 mg |
| Dose Reduction Level 2 | 140 mg | 70 mg | Discontinue |
| Dose Reduction Level 3 | Discontinue | Discontinue | |

For required dose modification for hepatic impairment refer to Section 5.3.1.5 and for concomitant treatment with CYP3A inhibitors refer to Section 6.2.1.

# **5.3.1.5.** Dose Modification for Subjects with Hepatic Impairment

Dose modifications for hepatic impairment will depend on baseline total bilirubin level and subsequent changes in bilirubin levels per Table 3 below. If the elevation of bilirubin is due to a non-hepatic cause or Gilbert's Syndrome, then no dose modifications are necessary.

 Table 3.
 Ibrutinib/Placebo Dose Modifications for Subjects with Hepatic Impairment

| Starting Dose Level by<br>Bilirubin Levels | Bili ≤1.5 x ULN at baseline:<br>420 mg | Bili >1.5-3 x ULN at baseline: 140 mg |
|---|---|---|
| On-study bilirubin level ≤1.5 x ULN | Continue 420 mg | Increase to 420 mg |
| On-study bilirubin level >1.5-3 x ULN | Reduce to 140 mg | Continue 140 mg |
| On-study bilirubin level >3 x ULN | <ul> <li>Hold* until bili level &gt;1.5-3 x ULN restart at 140mg</li> <li>When bili level ≤1.5 x ULN</li> </ul> | <ul> <li>Hold* until bili level &gt;1.5-3 x ULN restart at 140mg</li> <li>When bili level ≤1.5 x ULN</li> </ul> |
| | restart at 420mg | restart at 420mg |

Bili = bilirubin

## 5.3.1.6. Ibrutinib/Placebo Hold after Withdrawal of All Immunosuppressants

At the physician's discretion, ibrutinib/placebo may be held if ALL of the following conditions are met:

- All systemic immunosuppressants used for the treatment of cGVHD have been discontinued. (The continued use of very low doses of corticosteroids used only for physiologic adrenal replacement is allowed)
- cGVHD response has been maintained for 12 weeks after complete withdrawal of all immunosuppressants (not including ibrutinib/placebo)
- The subject has received a minimum of 48 weeks of ibrutinib/placebo

If cGVHD returns/worsens after ibrutinib/placebo has been held for the above criteria, ibrutinib/placebo may be re-started after consulting with the medical monitor.

<sup>\*</sup> In cases where the investigator wishes to restart ibrutinib/placebo after ibrutinib/placebo has been held for more than 28 days for hepatic impairment, please contact the medical monitor for approval. In the event a patient has had a dose reduction due to a non-hepatic toxicity and then develops elevated bilirubin level (or vice versa) that requires a dose reduction, the lower of the two dose reductions should be used. The medical monitor should be consulted for any questions involving dose reductions

#### 5.3.2. Prednisone

# 5.3.2.1. Formulation/Packaging/Storage

Prednisone tablets for oral administration are available in multiple strengths. Commercially available prednisone will be supplied by the Sponsor where applicable. The commercial material will be relabeled for clinical trial use.

For situations where a subject who must receive an IV or alternate formulation of corticosteroid (eg, hospitalization for AE), the dose should be equivalent to the subject's prednisone dose using the prednisone equivalency table (Appendix K) unless the subjects clinical condition warrants a different dose (eg, stress doses of steroids for sepsis). All doses of corticosteroids must be entered into the eCRF.

Refer to the Pharmacy Manual for additional guidance on prednisone storage, preparation and handling.

#### **5.3.2.2.** Dose and Administration

Prednisone will be given orally at 1.0 mg/kg/d with rounding to multiples of 5 mg (eg, 15, 20, 25, etc.).

If a prednisone dose of 1.0 mg/kg/d is contraindicated (eg, poorly controlled diabetes, major mood disturbances) then the starting dose of prednisone may be reduced to 0.5-1.0 mg/kg/d. Subjects unable to receive a starting dose of prednisone of at least 0.5 mg/kg/d are ineligible for the study.

If, during Screening, the clinical condition of the subject requires immediate initiation of treatment with prednisone, prednisone may be started prior to randomization. If the subject begins prednisone during Screening and prior to randomization the eligible subject must be randomized within 7 days of starting prednisone.

If a subject has started corticosteroids within the 72 hours prior to consent, then the subject is eligible and can continue corticosteroids after signing consent but must be randomized within 7 days of signing consent.

# 5.3.2.2.1. Prednisone Taper

Prednisone taper should be attempted by the schedule outlined in Table 4:

Table 4. Prednisone Taper Schedule

| Study Week # | Dose (mg/kg, body weight) |
|--------------|---------------------------|
| 0 | 1.0 qd |
| 2 | 0.75 qd |
| 4 | 0.65 qd |
| 6 | 0.50 qd |
| 8 | 0.70 qod* |
| 10 | 0.55 qod |
| 12 | 0.45 qod |
| 14 | 0.35 qod |
| 16 | 0.25 qod |
| 18 | 0.20 qod |
| 20 | 0.15 qod |
| 22 | 0.10 qod |
| 24 | 0.0 |

<sup>\*</sup>qod=every other day. \*Timing of steroid taper is defined by when the first dose of prednisone is given.

The prednisone taper should commence by week 2, but it is understood that considerable variation in prednisone taper will occur depending on the subjects' response and other intercurrent illnesses. More rapid tapering of prednisone doses is allowed if clinically appropriate. Rounding of corticosteroid doses is acceptable. Decisions about the use of qod or alternative dosing schedules (eg, Mon/Wed/Fri) may follow institutional practice. Prednisone taper should be completed prior to tapering of other immunosuppressants unless the clinical condition of the subject dictates tapering/discontinuing other medications sooner (eg, toxicity associated with the use of the medication).

#### **5.3.2.2.2.** Flares in cGVHD

Exacerbation of cGVHD symptoms may occur during prednisone taper or with intercurrent illnesses. Temporary re-escalation of prednisone dose is allowed at the physician's discretion. Tapering of increased prednisone dose for a flare should begin within 4 weeks.

#### **5.3.2.3.** Overdose

The effects of accidental ingestion of large quantities of prednisone over a very short period of time have not been reported, but prolonged use of the drug can produce mental symptoms, moon face, abnormal fat deposits, fluid retention, excessive appetite, weight gain, hypertrichosis, acne, striae, ecchymosis, increased sweating, pigmentation, dry scaly skin, thinning scalp hair, increased blood pressure, tachycardia, thrombophlebitis, decreased resistance to infection, negative nitrogen balance with delayed bone and wound healing, headache, weakness, menstrual disorders, accentuated menopausal symptoms, neuropathy, fractures, osteoporosis, peptic ulcer,

decreased glucose tolerance, hypokalemia, and adrenal insufficiency. Hepatomegaly and abdominal distention have been observed in children.

Treatment of acute overdosage is by immediate gastric lavage or emesis followed by supportive and symptomatic therapy. For chronic overdosage in the face of severe disease requiring continuous steroid therapy the dosage of prednisone may be reduced only temporarily, or alternate day treatment may be introduced.

#### **5.3.2.4.** Dose Modification for Adverse Reactions

Prednisone will be tapered by study design according to clinical response in cGVHD (Table 4). Prednisone suppresses the hypothalamic-pituitary-adrenal (HPA) axis and, therefore, doses must be tapered slowly after long-term use. The occurrence of unmanageable adverse reactions from prednisone (eg, poorly controlled hypertension) may require a more rapid reduction in prednisone dosing, but may not necessitate a change in dose of study drug (ibrutinib/placebo). Dose modifications will be at the discretion of the physician and should reflect a balance of appropriately treating cGVHD and minimizing adverse effects.

#### 5.4. Criteria for Permanent Discontinuation of Ibrutinib/Placebo

Investigators are encouraged to keep a subject who is experiencing clinical benefit in the study unless significant toxicity puts the subject at risk or routine noncompliance puts the study outcomes at risk. For a complete list of criteria for permanent discontinuation of ibrutinib/placebo, refer to Section 9.2.

An End-of-Treatment visit (Section 8.2.3) is required for all subjects except for those subjects who have withdrawn full consent.

# 6. <u>CONCOMITANT MEDICATIONS/PROCEDURES</u>

Concomitant therapies must be recorded from 30 days prior to signing of the ICF through 30 days after the last dose of study treatment (ibrutinib/placebo or corticosteroids), start of another therapy for cGVHD, or start of a new therapy for progression for the underlying malignancy.

## **6.1.** Permitted Concomitant Medications

## 6.1.1. Ancillary Therapy and Supportive Care

Ancillary therapy and supportive care for cGVHD is permitted as outlined in the NIH Consensus Development Project 2014 Ancillary Therapy and Supportive Care Working Group Report (Carpenter 2015, Appendix L). In particular, the use of regimen to specifically treat or prevent bronchiolitis obliterans are allowed (eg, inhaled steroids/azithromycin/montelukast) and will not be considered systemic treatment for cGVHD.

Other supportive medications in accordance with standard clinical practice (such as for emesis, diarrhea, etc.) are permitted. Use of neutrophil growth factors (filgrastim and pegfilgrastim) or red blood cell growth factors (erythropoietin) is permitted per institutional policy. Transfusions may be given in accordance with institutional policy. Anti-fungal prophylaxis should be given as outlined in Appendix L.

After consultation with the medical monitor the following may be considered; localized hormonal or bone sparing treatment for malignancies, and localized radiotherapy for medical conditions other than the underlying disease.

# 6.1.2. Systemic Immunosuppressant Therapy

During the Screening period, the physician will have the discretion to start prednisone while eligibility for the study is being confirmed, however, the subject must be randomized within 7 days of initiating treatment with prednisone.

Addition of any other new systemic immunosuppressant therapy (including ECP) to treat cGVHD is prohibited during Screening and subsequent enrollment into the study. Addition of a new systemic immunosuppressant for cGVHD will be considered a treatment failure and ibrutinib/placebo will be discontinued.

At enrollment, subjects may be receiving other immunosuppressants for the prophylaxis or treatment of acute GVHD. Tapering of these other immunosuppressants upon start of ibrutinib/placebo or prednisone is permitted (see Section 5.3.2.2.1).

Use of immunosuppressants for reasons other than treatment for cGVHD should be discussed with the medical monitor.

## **6.2.** Medications to be Used with Caution

# 6.2.1. CYP3A Enzyme Inhibitors/Inducers

Ibrutinib is metabolized primarily by CYP3A4. The dose of ibrutinib/placebo should be adjusted for concomitant use of CYP3A inhibitors per Table 5 below:

Table 5. Ibrutinib/Placebo Dose Modifications for Concomitant Use of CYP3A Inhibitors

| CYP inhibitor class | Dose modification instructions |
|---|---|
| Mild CYP3A inhibitors | 420 mg once daily. No dose adjustment required. |
| Moderate CYP3A inhibitors | 420 mg once daily. No dose adjustment required. |
| <ul> <li>Voriconazole at any dose or</li> <li>Posaconazole at doses less than or equal to suspension 200 mg BID or delayed-release tablet 300 mg QD</li> </ul> | 280 mg once daily |
| <ul> <li>Strong CYP3A inhibitors or</li> <li>Posaconazole at higher doses</li> </ul> | 140 mg once daily or consider alternative with less<br>CYP3A inhibitory potential |

Avoid concomitant use of strong CYP3A inducers (Appendix D). Consider alternative agents with less CYP3A induction and transition to a new agent within 4 weeks of randomization.

A list of common CYP3A inhibitors and inducers is provided in Appendix D. For further information, please refer to the current version of the ibrutinib IB and examples of inhibitors, inducers, and substrates can be found at http://medicine.iupui.edu/clinpharm/ddis/main-table/. This website is continually revised and should be checked frequently for updates.

## 6.2.2. Drugs That May Have Their Plasma Concentrations Altered by Ibrutinib

In vitro studies indicated that ibrutinib is not a substrate of P-glycoprotein (P-gp), but is a mild inhibitor. Ibrutinib is not expected to have systemic drug-drug interactions with P-gp substrates. However, it cannot be excluded that ibrutinib could inhibit intestinal P-gp after a therapeutic dose. There is no clinical data available. Therefore, to avoid a potential interaction in the GI tract, narrow therapeutic range P-gp substrates such as digoxin, should be taken at least 6 hours before or after ibrutinib/placebo.

# 6.2.3. Antiplatelet Agents and Anticoagulants

Supplements such as fish oil and vitamin E preparations should be avoided. Use ibrutinib/placebo with caution in subjects requiring anticoagulants or medications that inhibit platelet function. Subjects with congenital bleeding diathesis have not been studied. For guidance on ibrutinib/placebo and the use of anticoagulants during procedures/surgeries see Section 6.4.

Subjects requiring the use of therapeutic anticoagulation therapy (eg, atrial fibrillation), consider the risks and benefits of continuing ibrutinib treatment. Subjects treated with warfarin (or other

vitamin K antagonists) should maintain an INR  $\leq$  3.0 and if unable to maintain this level another anticoagulant agent should be considered. If therapeutic anticoagulation is clinically indicated, treatment with ibrutinib/placebo should be held while anticoagulation is being initiated and not be restarted until the subject is clinically stable and has no signs of bleeding. Subjects should be observed closely for signs and symptoms of bleeding. No dose reduction is required when study drug is restarted.

## 6.3. Other Systemic Immunosuppressant Therapy for cGVHD

Addition of any other *new* systemic immunosuppressant therapy (including ECP) to treat cGVHD is prohibited during Screening and subsequent enrollment into the study. The addition of other systemic immunosuppressant therapy to treat cGHVD will not allow for the appropriate assessment of response attributable to ibrutinib/placebo. The Sponsor must be notified in advance (or as soon as possible thereafter) of any instances in which prohibited therapies are administered.

# 6.4. Guidelines for Ibrutinib Management with Surgeries or Procedures

Ibrutinib may increase risk of bleeding with invasive procedures or surgery. The following guidance should be applied to the use of ibrutinib/placebo in the perioperative period for subjects who require surgical intervention or an invasive procedure while receiving ibrutinib/placebo.

## **6.4.1.** Minor Surgical Procedures

For minor procedures (such as a central line placement, skin or needle biopsy, lumbar puncture [other than shunt reservoir access], thoracentesis, or paracentesis) ibrutinib/placebo should be held for at least 3 days prior to the procedure and should not be restarted for at least 3 days after the procedure. For bone marrow biopsies that are performed while the subject is on ibrutinib/placebo, it is not necessary to hold ibrutinib/placebo.

# **6.4.2.** Major Surgical Procedures

For any surgery or invasive procedure requiring sutures or staples for closure, ibrutinib/placebo should be held at least 7 days prior to the intervention (except for emergency procedures) and should be held at least 7 days after the procedure and restarted at the discretion of the investigator when the surgical site is reasonably healed without serosanguineous drainage or the need for drainage tubes.

# 7. <u>STUDY EVALUATIONS</u>

# 7.1. Description of Procedures

## 7.1.1. Assessments

## 7.1.1.1. Informed Consent Form (ICF)

Adult subjects must read, understand, and sign the Institutional Review Board/Research Ethics Board/Independent Ethics Committee (IRB/REB/IEC) approved ICF confirming his or her willingness to participate in this study before any study-specific screening procedures are performed. Consent of minors consists of signed parental permission form and minor's assent. Subjects must also grant permission to use protected health information per the Health Insurance Portability and Accountability Act (HIPAA). In addition, subjects must sign all approved ICF amendments per the site IRB/REB/IEC guidelines during the course of the study.

## 7.1.1.2. Confirm Eligibility

All necessary procedures and evaluations must be performed to document that the subject meets all of the inclusion criteria and none of the exclusion criteria prior to first dose on Day 1 (Section 4). Details of establishing diagnosis of moderate or severe cGVHD are listed in Appendix M, Appendix N, and Appendix O. Please refer to NIH Staging and Response Assessment Manual for further details.

All subjects with prior malignancy as the indication for transplantation must be assessed prior to randomization to rule out progression of underlying malignancy. Assessments are to be performed and collected as deemed appropriate for the follow-up and management for routine standard of care of the underlying malignancy. The results of these assessments do not have to be known prior to randomization.

An enrollment eligibility form must be completed prior to enrollment into the trial.

## 7.1.1.3. Medical History and Demographics

The subject's relevant medical history through review of medical records and by interview will be collected and recorded. Concurrent medical signs and symptoms must be documented to establish baseline severities. A disease history, including the date of initial diagnosis will be recorded. For subjects <22 years of age at the time of enrollment, medical history will include surveillance for potential late effects (Appendix P).

## 7.1.1.4. Prior and Concomitant Medications

All medications from 30 days prior to signing of ICF through 30 days after the last dose of ibrutinib/placebo or prednisone, start of another therapy for cGVHD, or start of a new therapy for progression of underlying malignancy will be documented.

## 7.1.1.5. Adverse Events

The accepted regulatory definition for an AE is provided in Section 11.1. The occurrence of an AE from the time the ICF is signed until first dose should be recorded under medical history in the eCRF form. All medical occurrences after the first dose of ibrutinib/placebo or prednisone until 30 days after the last dose of ibrutinib/placebo or prednisone, start of new medication for cGVHD or start of a new therapy for progression of the underlying malignancy that meet the AE definition must be recorded as AEs in the eCRF. If the subject rolls over into a follow-up study, AE collection will stop after the last dose is given as part of that study. Laboratory abnormalities designated clinically significant by the investigator will also be documented as AEs. Assessment for corticosteroid-related AEs, in particular (Appendix Q), should be performed. Additional important requirements for AE and SAE reporting are explained in Section 11.4.

## 7.1.1.6. Physical Examination

The physical examination will include height (at Screening for adults, and at Screening and annually for subjects <22 years at the time of enrollment), weight, and examination per clinical practice.

## 7.1.1.7. Karnofsky/Lansky Performance Scale

The Karnofsky/Lansky Performance Scale is provided in Appendix C. The Lansky scale is to be used for all subjects less than 16 years of age.

## **7.1.1.8.** Vital Signs

Vital signs will include blood pressure, heart rate, respiratory rate, and body temperature.

## 7.1.2. Laboratory

## 7.1.2.1. Hematology

Hematology will be evaluated by a central laboratory and parameters will include a complete blood count: white blood cells, red blood cells, hemoglobin, hematocrit, platelets, neutrophils, lymphocytes, monocytes, eosinophils, basophils.

## 7.1.2.2. Chemistry (Serum)

Serum chemistry will be evaluated by a central laboratory and parameters will include sodium, potassium, chloride, blood urea nitrogen (BUN)/Urea, creatinine, glucose, calcium, total protein, albumin, AST, ALT, alkaline phosphatase, total bilirubin, lactate dehydrogenase (LDH), phosphate, uric acid, magnesium and bicarbonate.

#### 7.1.2.3. Infection Surveillance

Subjects should be monitored closely for signs or symptoms of aspergillus infection and other opportunistic infections. Screening for infectious agents, including fungal (eg, aspergillus) and viral (eg, CMV) infections as appropriate for the subjects' clinical course and medical history, should be performed.

## 7.1.2.4. Coagulation Studies

Measurement of PT/INR and aPTT will be performed at Screening using a local laboratory.

# 7.1.2.5. Hepatitis Serologies

Hepatitis serologies will be evaluated by a local laboratory and include hepatitis C antibody, hepatitis B surface antigen, and hepatitis B core antibody. If hepatitis B core antibody, hepatitis B surface antigen, or hepatitis C antibody is positive, then PCR to quantitate hepatitis B DNA or hepatitis C RNA must be performed and must be negative prior to randomization. Hepatitis serologies and/or PCR obtained as part of standard of care within 28 days prior to randomization are acceptable for use in establishing eligibility.

## 7.1.2.6. Serum Immunoglobulins

Serum immunoglobulins will be evaluated by a central laboratory and include IgA, IgG and IgM levels.

## 7.1.2.7. Pregnancy Test

Serum pregnancy test will be required at Screening by local laboratory only for women of childbearing potential. A urine pregnancy test will also be performed on Day 1 prior to first dose. If positive, pregnancy must be ruled out by ultrasound to be eligible. This test may be performed more frequently if required by local regulatory authorities.

## 7.1.3. Diagnostics/Procedures

## 7.1.3.1. Electrocardiograms (ECG)

Electrocardiograms should be performed at the investigator's discretion, particularly in subjects with arrhythmic symptoms (eg. palpitations, lightheadedness) or new onset dyspnea.

During visits in which both ECGs and blood draws are performed, ECGs should be performed first.

At Screening, a 12-lead ECG is required.

Abnormalities noted at Screening should be included in the medical history. Subjects <22 years of age at enrollment will have a second ECG on Week 2 Day 1 during PK testing. This ECG should be done 2-4 hours after ibrutinib/placebo has been taken.

## 7.1.3.2. Forced Expiratory Volume in 1 Second (FEV1)

Forced expiratory volume in 1 second (FEV1) should be measured using spirometry and FEV1 measurement should be obtained prior to randomization. FEV1 values obtained as standard of care within 56 days prior to randomization can be used to fulfill the requirement for a baseline FEV1 measurement. If FEV1 results are abnormal at baseline, then subsequent FEV1 measurements should be obtained every 12 weeks. If the FEV1 result is normal at baseline, then subsequent FEV1 measurements should be obtained every 24 weeks. The NIH Lung score should be ascertained with every cGVHD activity assessment regardless of whether a FEV1 is performed.

## 7.1.4. Pharmacokinetics/Biomarkers

#### 7.1.4.1. Pharmacokinetics

Plasma concentrations of ibrutinib and metabolite PCI-45227 after repeated dosing will be determined using a validated analytical method. Other potential metabolites of ibrutinib may be explored. Refer to Appendix B for PK sample collection schedule.

If ibrutinib/placebo is on hold or missed at the Week 2 or Week 25 PK evaluation, PK testing should be obtained on the next scheduled visit after ibrutinib dose has been stable for a minimum of 7 days.

# 7.1.4.2. Biomarkers and Pharmacodynamic Studies

Biological specimens collected at specified timepoints during the study may be used for pharmacodynamic and biomarker assessments as indicated as well as sequencing expression analysis, immunophenotyping and secreted protein analyses. Refer to Appendix B for pharmacodynamic, biomarker and T/B/NK sample collection schedule.

Samples collected in this study may be stored at a biorepository for up to 10 years (or according to local regulations) for additional research as new assays are developed for ibrutinib and cGVHD. Samples will be used to better understand the effects of ibrutinib, cGVHD, sensitivity and/or resistance to the investigational treatment regimen in this study. The research may begin at any time during the study or the post-study storage period. Stored samples will be coded throughout the sample storage and analysis process and will not be labeled with personal identifiers.

Specific analysis and platforms may include, but are not limited to, soluble protein isolation including chemokine and cytokine, protein identification and quantification, viable cell manipulation, stimulation and co-culture, kinase drug occupancy studies, flow cytometric or

CyTOF based cell identification, and phospho-protein analyses. New analysis platforms and assays directed at protein specific outputs may be considered as technologies develop and improve or as new relevant disease or therapy markers are recognized.

# 7.1.4.3. Biomarker DNA and RNA Sequencing

T-cell and B-cell genetic functional diversity will be determined using a combination of TCR and BCR sequencing platform data alongside functional and immunophenotyping assays. The goal of these studies will be to establish study drug related changes to the systemic immune environment of the subjects.

RNA and DNA species analysis and or RNA/DNA sequencing may be performed on cells obtained from biomarkers specimens in an effort to quantify the expression or mutation of specific genes implicated in cGVHD disease pathogenesis and or therapy response.

# 7.2. Sample Collection and Handling

The actual dates and times of sample collection must be recorded in source documents for transcription to the eCRF or central laboratory requisition form. Refer to the Schedule of Assessments (Appendix A and Appendix B) for the timing and frequency of all sample collections.

Instructions for the collection, handling, and shipment of samples are found in the Central Laboratory Manual.

## 7.3. Efficacy Evaluations

## 7.3.1. NIH Consensus Panel Response Criteria

Response will be defined using the NIH Consensus Panel Chronic GVHD Activity Assessment (Appendix H and Appendix I).

## **Overall Response:**

Skin, mouth, liver, upper and lower GI, esophagus, lung, eye, and joint/fascia are the organs or sites considered in evaluating overall response.

- Complete Response (CR) is defined as resolution of all manifestations in each organ or site.
- Partial Response (PR) is defined as improvement in at least 1 organ or site without progression in any other organ or site.
- Disease Progression is defined as clinically meaningful worsening in one or more organs regardless of improvement in other organs. Note that mixed response (ie, improvement in at least 1 organ accompanied by progression in another organ) is considered disease progression.

• Stable disease (SD): response that does not meet the criteria for CR, PR, or disease progression.

Please refer to NIH Staging and Response Assessment Manual and Appendix I for further details

## 7.3.2. Lee cGVHD Symptom Scale and SF-36 Questionnaire

All subjects in the study will complete the Lee cGVHD Symptom Scale (Appendix F) and SF-36 questionnaire (Appendix G) at all cGVHD activity assessment visits. These questionnaires should be administered before other study procedures.

## 7.3.3. Late effects surveillance for adolescents (<22 years at randomization)

Late effects surveillance for adolescents will consist of the collection of data on growth and development (height, weight, and Tanner Stage) and medical records review for late effects of transplantation. This assessment will be performed at Screening and annually up to 5 years post randomization (Appendix P).

## 8. <u>STUDY PROCEDURES</u>

## 8.1. Screening Phase

# 8.1.1. Screening/Consenting Visit

The following procedures will be performed at the Screening Visit within 28 days prior to randomization unless otherwise noted:

- Obtain signed, written informed consent and if applicable, child assent, and parental permission
- Medical history including demographic information
- Record history related to late effect surveillance for subjects <22 years of age at the time of enrollment using the Late-Effects surveillance form (Appendix P)
- Collection of transplant history, including indication
- cGVHD Diagnosis and staging (NIH) (Appendix M, Appendix N, and Appendix O)
- Assessment for relapse/progressive disease for subjects receiving transplant for malignant disorders
- Infection surveillance
- Evaluation of Karnofsky/Lansky performance status (Appendix C)
- Physical examination including, height and weight. Document Tanner stage for subjects <22 years of age (subjects ≥22 years may use prior height measurement if available in source documents) (Appendix P)
- Record AEs since signing the ICF

- Record concomitant medication history including corticosteroids requirement, over-the-counter drugs, vitamins and herbs since 30 days prior to signing ICF
- cGVHD activity assessment (eg, NIH assessments [Appendix H and Appendix J]). For subjects who begin prednisone prior to randomization, cGVHD activity assessment should be completed prior to start of prednisone. If prednisone is started at the time that ibrutinib/placebo is started (Day 1) then activity assessment can be completed any time during Screening up until the day of first dose of ibrutinib/placebo (Day 1).
- Lee cGVHD Symptom Scale (Appendix F)/SF-36 questionnaire (Appendix G). Perform at the same time as cGVHD assessment.
- FEV1 (see Section 7.1.3.2)
- Obtain vital signs (including blood pressure, heart rate, respiratory rate, and body temperature) after the subject has rested in the sitting position for ≥3 minutes
- Obtain blood specimens for the following laboratory tests:
  - Hematology
  - Serum chemistry
  - o Coagulation studies: PT/INR, aPTT
  - Hepatitis serologies/PCR
- T/B/NK sampling (Appendix B)
- Biomarker sampling (Appendix B)
- Obtain 12-lead ECG after the subject has been in a supine position and resting for at least 10 minutes
- Obtain serum pregnancy test for women of childbearing potential only
- Complete eligibility form prior to randomization in Treatment Phase
- Obtain subject number in the IWRS system

At any time from consent throughout the treatment period, the subject may be called to discuss potential prednisone dosing changes. The phone call will be documented in the source documentation and will be entered in the CRF.

## **8.2.** Treatment Phase

## 8.2.1. Treatment Visits

## 8.2.1.1. Week 1 Day 1

Following completion of the Screening Visit and once eligibility has been confirmed, subjects are randomized. Randomization should occur as close to the time of the expected first dose as possible, ie, not more than 3 days prior to expected first dose with study drug.

#### **Predose**

- Physical examination
- Vital signs
- Performance status (KPS/Lansky) (Appendix C)
- cGVHD activity assessment per NIH (Appendix H and Appendix J). Only perform if not performed previously during Screening (see Section 8.1.1 above).
- Lee cGVHD Symptom Scale (Appendix F)/SF-36 Questionnaire (Appendix G). Only perform if not performed previously during Screening (see Section 8.1.1 above).
- FEV1. Only perform if not performed previously during Screening (see Section 7.1.3.2)
- Hematology
- Serum chemistry
- Urine pregnancy test for women of childbearing potential
- Quantitative serum immunoglobulins (IgA, IgM, IgG)
- Review of baseline AEs and concomitant medications (including corticosteroid requirements)
- Review of inclusion and exclusion criteria to re-confirm subject eligibility prior to first dosing
- Pharmacodynamic sampling (Appendix B)
- T/B/NK sampling (Appendix B)
- Biomarker sampling (Appendix B)

## **Postdose**

- Administer ibrutinib/placebo at specified dose level, and then dispense remaining amount to subject for at-home dosing
- Provide drug diary and dosing instructions to subject
- Review AEs

### 8.2.1.2. Week 2

## **Predose**

- Physical examination
- Hematology
- Serum chemistry
- Vital signs
- Review AEs and concomitant medications (including corticosteroid requirements)
- Pharmacokinetic sampling (Appendix B)

#### **Postdose**

- Administer ibrutinib/placebo at specified dose level
- Pharmacokinetic sampling at 1, 2, 4, and 6 hours postdose (Appendix B)
- For subjects <22 years of age at enrollment: Obtain 12-lead ECG approximately 2-4 hours post ibrutinib/placebo dose, after the subject has been in a supine position and resting for at least 10 minutes

## 8.2.1.3. Week 5, 9, 13, 17, 21, 25

#### **Predose**

- Physical examination
- Vital signs
- Performance status (KPS/Lansky) (Appendix C)
- Hematology
- Serum chemistry
- cGVHD activity assessment per NIH (Appendix H and Appendix J) (Weeks 5, 13 and 25 only)
- cGVHD response assessment (Appendix I) (Weeks 5, 13 and 25 only)
- Lee cGVHD Symptom Scale (Appendix F)/SF-36 Questionnaire (Appendix G) (Weeks 5, 13 and 25 only)
- FEV1 (Week 13 if abnormal at Screening, Week 25 for all subjects, see Section 7.1.3.2)
- Quantitative serum immunoglobulins (IgA, IgG, and IgM) (Weeks 13 and 25 only)
- Pharmacokinetic sampling (Appendix B) (Week 25 only)
- Pharmacodynamic sampling (Appendix B)
- T/B/NK sampling (Appendix B)
- Biomarker sampling
- Review returned subject dosing diary
- Drug accountability
- Review AEs and concomitant medications (including corticosteroid requirements)

## **Postdose**

- Administer ibrutinib/placebo at specified dose level, and then dispense remaining amount to subject
- Pharmacokinetic sampling at 1, 2, 4, and 6 hours postdose (Week 25 only)

# 8.2.1.4. Week 37, 49, and every 12 weeks thereafter ( $\pm$ 7 days)

## **Predose**

- Physical examination
- Vital signs
- Performance status (KPS/Lansky) (Appendix C)
- Hematology
- Serum chemistry
- cGVHD activity assessment per NIH (Appendix H and Appendix J)
- cGVHD response assessment (Appendix I)
- Lee cGVHD Symptom Scale (Appendix F)/SF-36 Questionnaire (Appendix G)
- FEV1 every 12 weeks if prior FEV1 was abnormal, every 24 weeks if prior FEV1 was normal (see Section 7.1.3.2)
- Quantitative serum immunoglobulins (IgA, IgG, and IgM)
- Pharmacodynamic sampling (Appendix B) (Weeks 49, 73, and 97 only)
- T/B/NK sampling (Appendix B) (Weeks 37, 49, 73 and 97 only)
- Biomarker sampling (Appendix B) (Weeks 37, 49, 73 and 97 only)
- Review returned subject dosing diary
- Drug accountability
- Review AEs and concomitant medications (including corticosteroid requirements)

## **Postdose**

• Administer ibrutinib/placebo at specified dose level, and then dispense remaining amount to subject

## 8.2.2. Progressive Disease Visit

Progressive Disease visit should be performed at any time during the study, if based on clinical and/or laboratory evaluation, the Investigator suspects progressive disease. If possible, the visit should be performed within 72 hours after the subject's previous dose.

- Physical examination
- Vital signs
- Performance status (KPS/Lansky) (Appendix C)
- Hematology
- Serum chemistry
- cGVHD activity assessment per NIH (Appendix H and Appendix J)
- cGVHD response assessment (Appendix I)
- Lee cGVHD Symptom Scale (Appendix F)/SF-36 Questionnaire (Appendix G)

- FEV1 (if not obtained within the previous 12 weeks, see Section 7.1.3.2)
- Quantitative serum immunoglobulins (IgA, IgG, and IgM)
- Review AEs and concomitant medications (including corticosteroid requirements)
- Review returned subject dosing diary
- Final drug accountability
- Pharmacodynamic sampling (Appendix B)
- T/B/NK sampling (Appendix B)
- Biomarker sampling (Appendix B)

## 8.2.3. End-of-Treatment Visit

An End-of-Treatment visit should occur 30 days (±7 days) from the last dose of study drug or prior to the start of a new cGVHD treatment. If the subject starts a new cGVHD treatment less than 7 days after the Progressive Disease visit, only those procedures not conducted at the Progressive Disease visit should be performed at the End-of-Treatment visit. If ibrutinib/placebo is held after Week 48 due to response (see Section 5.3.1.6), the End-of-Treatment visit should occur 30 days after ibrutinib/placebo was put on hold.

The following procedures will be performed at the End-of-Treatment visit:

- Physical examination
- Vital signs
- Performance status (KPS/Lansky) (Appendix C)
- Hematology
- Serum chemistry
- cGVHD activity assessment per NIH (Appendix H and Appendix J) (if not performed within previous 30 days)
- cGVHD response assessment (Appendix I) (if not performed within previous 30 days)
- Lee cGVHD Symptom Scale (Appendix F)/SF-36 Questionnaire (Appendix G) (if not performed within previous 30 days)
- FEV1 (if not obtained within previous 12 weeks)
- Quantitative serum immunoglobulins (IgA, IgG, and IgM)
- Review AEs and concomitant medications (including corticosteroid requirements and any new cGVHD treatment if applicable)
- Review returned subject dosing diary
- Final drug accountability

# 8.3. Follow-up Phase

Once a subject has completed the End-of-Treatment visit they will enter the Follow-up Phase. Subjects that withdraw from treatment for reasons other than progressive cGVHD or progression of their underlying malignancy will participate in ongoing response follow-up.

## 8.3.1. Response Follow-up

Subjects who discontinue ibrutinib/placebo for reasons other than progressive cGVHD or progression of underlying malignancy will be followed at pre-specified response assessment time points (Weeks 5, 13, 25 and every 12 weeks thereafter) by clinic visit until progressive disease or progression of underlying malignancy. During this period, the following procedures will be performed:

- Physical examination
- Vital signs
- Performance status (KPS/Lansky) (Appendix C)
- Hematology
- Serum chemistry
- cGVHD activity assessment per NIH (Appendix H and Appendix J)
- cGVHD response assessment (Appendix I)
- Lee cGVHD Symptom Scale (Appendix F)/SF-36 Questionnaire (Appendix G)
- FEV1 every 12 weeks if prior FEV1 abnormal, every 24 weeks if prior FEV1 normal
- Review corticosteroid requirements and any new cGVHD treatment if applicable

# 8.3.2. Long-Term Follow-up

Once subjects have cGVHD progression, or have progression of their underlying malignancy (for subjects who have not withdrawn consent), they will be contacted approximately every 12 weeks (±14 days) by clinic visit or telephone to assess survival and the use of alternative cGVHD therapy. In addition, subjects who have progressive cGVHD will continue to have the Lee Symptom Scale and SF-36 assessments until the week 60 visit. Subjects will be contacted until death, subject withdrawal, lost to follow-up, or study termination by the Sponsor, whichever occurs first.

## 8.3.3. Expected length of participation on study

The Sponsor will continue to follow adult subjects up to approximately 3 years after the first subject was randomized. Adolescents (<22 years of age at the time of randomization) will be followed for up to 5 years after randomization; however, the study may close after the last patient below 18 years of age has exited the study if all other participating subjects have completed a minimum of 1 year of follow-up. Subjects may be rolled over to a long-term extension study for long-term follow-up.

## 9. SUBJECT COMPLETION AND WITHDRAWAL

# 9.1. Completion

A subject will be considered to have completed the study if he or she has died before the end of the study, has not been lost to follow up, or has not withdrawn consent before the end of study.

## 9.2. Discontinuation from Ibrutinib/Placebo

Ibrutinib/placebo will be discontinued in the event of any of the following events:

- Subject begins treatment with another systemic therapy (including ECP) for cGVHD
- cGVHD progression
- Progression or relapse of the malignancy that was the indication for transplantation or development of PTLD
- Unacceptable toxicity: an intercurrent illness or AE that prevents further ibrutinib/placebo administration despite dose adjustment
- Noncompliance with study medication
- Investigator's decision (such as chronic noncompliance, significant protocol deviation, or best interest of the subject)
- Withdrawal of consent for treatment by subject
- Unblinding at primary efficacy analysis
- Study termination by Sponsor
- Subject becomes pregnant
- Death

All subjects, regardless of reason for discontinuation of ibrutinib/placebo will undergo an End-of-Treatment visit and be followed as outlined under Section 8.3

The investigator should notify the Sponsor within 24 hours if a subject discontinues ibrutinib/placebo treatment due to cGVHD progression and should provide documentation of cGVHD progression for review by the Sponsor's medical monitor.

## 9.3. Withdrawal from Study

Withdrawal from study (including all follow-up) will occur under the following circumstances:

- Withdrawal of consent for follow-up observation by the subject
- Lost to follow-up
- Study completion / termination
- Death

If a subject is lost to follow-up, every reasonable effort should be made by the study site personnel to contact the subject. The measures taken to follow up should be documented.

When a subject withdraws before completing the study, the following information should be documented in the source documents:

- Reason for withdrawal;
- Whether the subject withdraws full consent (ie, withdraws consent to treatment and all further contact) or partial consent (ie, withdraws consent to treatment but agrees to participate in follow-up visits); and/or, withdraws consent from future biomarker research.

# 10. STATISTICAL METHODS AND ANALYSIS

Statistical analysis will be done by the Sponsor or under the authority of the Sponsor. A general description of the statistical methods to be used to analyze the efficacy and safety data is outlined below. Specific details will be provided in the Statistical Analysis Plan.

# 10.1. Analysis Sets

## **10.1.1.** Intention-to-Treat Population (ITT)

The ITT Population is defined as all subjects who are randomized in the study. The ITT population will be used for all efficacy analyses.

The mITT Population is defined as all subjects who are randomized in the study (ITT) and who do not have evidence of progression of underlying malignancy from measurements made at or before the time of randomization. If indicated, the mITT population may be used for additional efficacy analyses.

## 10.1.2. Safety Population (SP)

The Safety Population will consist of all randomized subjects who received at least one dose of any study drug.

# **10.2.** Sample Size Determination

The null hypothesis is that the two treatment arms have the same response rate at 48 weeks and the alternative hypothesis is that the response rates of two arms are different.

Assuming a response rate of 30% at 48 weeks for Arm B (placebo + prednisone), a sample size of 186 randomized subjects provides at least 80% power to detect a 20% difference in the response rates at 48 weeks between the 2 treatment arms (Arm A – Arm B) at an alpha level of 5% (2-sided).

No replacement of subjects will be implemented.

# **10.3.** Subject Information

The distribution of subjects by treatment arm for each of the analysis populations will be provided. The number of subjects randomized, dosed, and discontinued will be summarized. Treatment discontinuation will be summarized according to the reasons for discontinuation and by treatment arm.

Demographic and baseline variables and baseline disease characteristics will be summarized by treatment arm.

# 10.4. Efficacy Analyses

# 10.4.1. Primary Efficacy Endpoint

The primary efficacy endpoint of this study is the response rate at 48 weeks (ie, the proportion of responders [CR or PR]). Response will be defined by the NIH Consensus Development Project Criteria (2014).

A subject will not be considered as a responder at 48 weeks if the response was not CR or PR, or if he/she meets any of following criteria:

- Starts a second-line systemic therapy for cGVHD at or prior to the response assessment at 48 weeks
- Has evidence of progression of the underlying malignancy that was the indication for transplant at or prior to response assessment at 48 weeks

Subjects who withdraw from the study prior to, or are missing the response at, 48 weeks will not be considered responders.

The primary efficacy analysis will be performed using the ITT population. The chi-square test will be used to compare the proportions between the two treatment arms.

# **10.4.2.** Secondary Endpoints for Efficacy

The secondary efficacy endpoints are:

- Response rate at 24 weeks (the proportion of responders [CR or PR]) as defined by the NIH Consensus Development Project (2014)
- Duration of response (DOR) will be defined from the time of initial partial or complete response until progression of cGVHD
- Proportion of subjects with steroid dose reduction to a level of less than 0.15 mg/kg/d at 24 weeks
- Time to withdrawal of all immunosuppressants (with the exception of ibrutinib/placebo)

- Overall survival (OS) is defined as the time from randomization until death due to any cause
- Improvement in Lee cGVHD Symptom Scale scores will be compared between the two treatment arms

Proportion of subjects with improvement in overall score on the Lee cGVHD Symptom Scale and the proportion of subjects with steroid dose reduction will be analyzed using the same method for the primary efficacy endpoint. The Kaplan Meier methodology will be used to estimate the distribution of OS for each treatment group. The log-rank test will be used to compare the OS between the 2 treatment arms. Time to withdrawal of all immunosuppressants will be analyzed using the same method used for OS.

Duration of response is defined as the interval between the date of initial documentation of a response (PR or better), and the date of first documented evidence of progressive cGVHD or death for responders only. Responders will include subjects who achieve response (PR or better) based on NIH 2014 cGVHD criteria. Non-responders will be excluded from the analysis for DOR. Median duration of response will be estimated using Kaplan Meier methodology.

## 10.4.3. Exploratory Endpoints

- Pharmacokinetics (PK) parameters of ibrutinib when administered in combination with prednisone in subjects with cGVHD including adolescent subjects
- Pharmacodynamic characteristics (including BTK and ITK occupancy) of ibrutinib in subjects with cGVHD
- Biomarkers relevant to disease biology and therapy with ibrutinib for cGVHD
- Summary scales of SF-36 patient reported outcome

## **Pharmacokinetic**

Ibrutinib and PCI-45227 bioanalytical data will be used in non-compartmental PK analysis. Plasma concentrations below the lowest quantifiable concentration will be treated as zero in the summary statistics. All subjects and samples excluded from the analysis will be clearly documented in the PK report.

Descriptive statistics will be used to summarize ibrutinib and PCI-45227 concentrations at each sampling time point and PK parameters of ibrutinib and PCI-45227 (including, but not limited to:  $C_{max}$ ,  $t_{max}$ ,  $AUC_{last}$ , and  $t_{1/2}$ ).

Individual and mean plasma ibrutinib and PCI-45227 concentration time profiles will be plotted.

Ibrutinib data from this study may also be combined with data from other studies performed with ibrutinib in subjects with hematologic malignancies as part of a population-PK analysis using nonlinear mixed effects models. For the population-PK analysis, covariates that could potentially

correlate with plasma PK parameters will be evaluated. The results of the population-PK analyses (if performed) will be presented in a separate report.

# **Biomarker and Pharmacodynamics**

The following biomarker assessments will be undertaken:

- 1. Sequence-directed Immune Function Assessment
- 2. Cytokine, Chemokine, and Soluble Biomarker Assessment
- 3. Co-culture Immunologic Function Tests
- 4. CyTOF-based Phospho-immunophenotyping

PK/PD and biomarkers will be evaluated separately and will not be covered in the statistical analysis plan (SAP).

## **Patient Reported Outcomes**

SF-36 summary scores will be evaluated; detailed analyses will be covered in the statistical analysis plan (SAP).

## 10.5. Safety Analysis

Analysis of safety data will be conducted on the safety population, which includes randomized subjects who receive at least 1 dose of ibrutinib/placebo. The baseline value is defined as the last value collected on or prior to the first dose date of ibrutinib/placebo, whichever comes first.

The safety variables to be summarized include exposure to ibrutinib/placebo and prednisone, AEs, clinical laboratory test results (hematology and chemistry), Karnofsky/Lansky performance status, and vital sign measurements. In general, safety data will be tabulated or listed. No formal statistical testing is planned.

Growth and development and late effects will be summarized in adolescent subjects.

## **Adverse Events**

The verbatim terms used in the eCRF by investigators to identify AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA).

Treatment-emergent period is defined as the period of time from the first dose of study treatment, until the earlier of:

• Thirty days following the last dose of ibrutinib/placebo or prednisone whichever occurs later

OR

• The start date of a new therapy for cGVHD or for the progression of the underlying malignancy.

The TEAEs are those events that:

- Are not present prior to the treatment-emergent period and occur during the treatment-emergent period,
- Are considered related to study drug by the investigator regardless of the start dates of the events, or
- Are present prior to the treatment-emergent period but worsen in severity during the treatment-emergent period or are subsequently considered related to study drug by the investigator.

All treatment-emergent AEs will be summarized. For each AE, the number and percentage of subjects who experience at least one occurrence of the given event will be summarized. The number and percent of subjects with TEAEs will be summarized according to intensity (CTCAE, v4.03) and drug relationship, as well as categorized by system organ class and preferred term. Summaries and listings may be provided, as appropriate, for those subjects who die, who discontinue treatment due to an AE, or who experience a severe or a SAE.

## **Clinical Laboratory Tests**

Laboratory tests will be summarized separately for hematology and serum chemistry. All laboratory values will be graded using the NCI CTCAE v4.03. The worst toxicity grade during the study will be tabulated.

## **Steroid-related Toxicities**

Treatment-emergent steroid-related AEs will be summarized by the two study arms (Appendix Q). The number and percent of subjects with steroids related TEAEs will be summarized according to intensity (CTCAE, v4.03) and will be categorized by system organ class and preferred term.

## 10.6. Interim Futility Review

An interim analysis (for futility only) will be performed for the first 50 subjects who complete the Week 25 visit or discontinue study drug before this time. The independent DMC will review the interim futility analysis results and make a recommendation accordingly. Details regarding the interim futility review will be described in the DMC charter.

# **10.7.** Data Monitoring Committee (DMC)

An independent DMC will be established to monitor data on an ongoing basis to ensure the continuing safety of the subjects enrolled in this study and to meet efficacy objectives. The committee will meet periodically to review interim data. After the review, the DMC will make

recommendations regarding the continuation of the study. The DMC will also oversee the interim futility review. This review will be performed for the first 50 subjects who complete the Week 25 visit or discontinue study drug before this time. Available pharmacokinetics data will be provided to the DMC for the interim futility review.

The DMC will consist of at least one medical expert in the relevant therapeutic area and at least one statistician. The DMC responsibilities, authorities, and procedures will be documented in a separate charter.

## 11. ADVERSE EVENT REPORTING

Timely, accurate, and complete reporting and analysis of safety information from clinical studies are crucial for the protection of subjects, investigators, and the Sponsor, and are mandated by regulatory agencies worldwide. The Sponsor has established Standard Operating Procedures in conformity with regulatory requirements worldwide to ensure appropriate reporting of safety information; all clinical studies conducted by the Sponsor or its affiliates will be conducted in accordance with those procedures.

#### 11.1. Definitions

## 11.1.1. Adverse Events

An AE is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of an investigational study drug, whether or not considered related to the study drug (ICH-E2A 1995).

For the purposes of this clinical study, AEs include events which are either new or represent detectable exacerbations of pre-existing conditions.

The term "disease progression" should not be reported as an AE term. As an example, "worsening of underlying disease" or the clinical diagnosis that is associated with disease progression should be reported.

Adverse events may include, but are not limited to:

- Subjective or objective symptoms provided by the subject and/or observed by the investigator or study staff including laboratory abnormalities of clinical significance.
- Any AEs experienced by the subject through the completion of final study procedures.
- AEs not previously observed in the subject that emerge during the protocol-specified AE reporting period, including signs or symptoms associated with the underlying disease that were not present before the AE reporting period.

• Complications that occur as a result of protocol-mandated interventions (eg, invasive procedures such as biopsies).

The following are NOT considered AEs:

- **Pre-existing Condition:** A pre-existing condition (documented on the medical history CRF) is not considered an AE unless the severity, frequency, or character of the event worsens during the study period.
- **Pre-planned or Elective Hospitalization:** A hospitalization planned before signing the ICF is not considered an SAE, but rather a therapeutic intervention. However, if during the pre-planned hospitalization an event occurs, which prolongs the hospitalization or meets any other SAE criteria, the event will be considered an SAE. Surgeries or interventions that were under consideration, but not performed before enrollment in the study, will not be considered serious if they are performed after enrollment in the study for a condition that has not changed from its baseline level. Elective hospitalizations for social reasons, solely for the administration of chemotherapy, or due to long travel distances are also not SAEs.
- **Diagnostic Testing and Procedures:** Testing and procedures should not be reported as AEs or SAEs, but rather the cause for the test or procedure should be reported.

## 11.1.2. Serious Adverse Events

A SAE based on International Conference on Harmonisation (ICH) and EU Guidelines on Pharmacovigilance for Medicinal Products for Human Use is any untoward medical occurrence that at any dose:

- Results in death (ie, the AE actually causes or leads to death).
- Is life-threatening. Life-threatening is defined as an AE in which the subject was at risk of death at the time of the event. It does not refer to an event which hypothetically might have caused death if it were more severe. If either the investigator or the Sponsor believes that an AE meets the definition of life-threatening, it will be considered life-threatening.
- Requires in-patient hospitalization >24 hours or prolongation of existing hospitalization.
- Results in persistent or significant disability/incapacity (ie, the AE results in substantial disruption of the subject's ability to conduct normal life functions).
- Is a congenital anomaly/birth defect.
- Is an important medical event that may not result in death, be immediately life-threatening or require hospitalization, but may be considered an SAE when, based upon appropriate medical judgment, the event may jeopardize the subject or subject may require intervention to prevent one of the other outcomes listed in this definition. Examples of such events are intensive treatment in an emergency department or at home for allergic bronchospasm, blood dyscrasias, or convulsion that does not result in hospitalization; or development of drug dependency or drug abuse.

Given that the investigator's perspective may be informed by having actually observed the event, and the Sponsor is likely to have broader knowledge of the drug and its effects to inform its

evaluation of the significance of the event, if either the Sponsor or the investigator believes that the event is serious, the event will be considered serious.

# 11.1.3. Severity Criteria (Grade 1-5)

Definitions found in the Common Terminology Criteria for Adverse Events version 4.03 (CTCAE v4.03) will be used for grading the severity (intensity) of AEs. The CTCAE v4.03 displays Grades 1 through 5 with unique clinical descriptions of severity for each referenced AE. Should a subject experience any AE not listed in the CTCAE v4.03, the following grading system should be used to assess severity:

- Grade 1 (Mild AE) experiences which are usually transient, requiring no special treatment, and not interfering with the subject's daily activities
- Grade 2 (Moderate AE) experiences which introduce some level of inconvenience or concern to the subject, and which may interfere with daily activities, but are usually ameliorated by simple therapeutic measures
- Grade 3 (Severe AE) experiences which are unacceptable or intolerable, significantly interrupt the subject's usual daily activity, and require systemic drug therapy or other treatment
- Grade 4 (Life-threatening or disabling AE) experiences which cause the subject to be in imminent danger of death
- Grade 5 (Death related to AE) experiences which result in subject death

## 11.1.4. Causality (Attribution)

The investigator is to assess the causal relation (ie, whether there is a reasonable possibility that the study drug caused the event) using the following definitions:

**Not Related:** Another cause of the AE is more plausible; a temporal sequence

cannot be established with the onset of the AE and administration of the investigational product; or, a causal relationship is considered

biologically implausible.

**Unlikely:** The current knowledge or information about the AE indicates that a

relationship to the investigational product is unlikely.

**Possibly Related:** There is a clinically plausible time sequence between onset of the AE

and administration of the investigational product, but the AE could also be attributed to concurrent or underlying disease, or the use of other drugs or procedures. Possibly related should be used when the investigational product is one of several biologically plausible AE

causes.

**Related:** The AE is clearly related to use of the investigational product.

# 11.2. Unexpected Adverse Events

An "unexpected" AE is an AE that is not listed in the IB/package insert or is not listed at the specificity or severity that has been observed. For example, hepatic necrosis would be "unexpected" (by virtue of greater severity) if the IB referred only to elevated hepatic enzymes or hepatitis. Similarly, cerebral thromboembolism and cerebral vasculitis would be "unexpected" (by virtue of greater specificity) if the IB/package insert listed only cerebral vascular accidents. "Unexpected" also refers to AEs that are mentioned in the IB as occurring with a class of drugs or as anticipated from the pharmacological properties of the drug, but are not specifically mentioned as occurring with the study drug under investigation.

# 11.3. Special Reporting Situations

Special reporting situation on a Sponsor study may require expedited reporting and/or safety evaluation include, but are not limited to:

- Overdose of any study drug
- Suspected abuse/misuse of a study drug
- Inadvertent or accidental exposure to a study drug
- Medication error involving a product (with or without subject exposure to the study drug, eg, name confusion)

Occurrence of any special reporting situations should be recorded in the eCRF. If any special reporting situation meets the criteria of an AE, it should be recorded on the AEs eCRF. If the AE is considered serious, it should be recorded on the AEs eCRF as serious and should be reported on the Serious Adverse Event Report Form. The Serious Adverse Event Report Form should be sent via email or fax to Pharmacyclics Drug Safety or designee within 24 hours of awareness.

# 11.4. Documenting and Reporting of Adverse Events and Serious Adverse Events by Investigators

## 11.4.1. Assessment of Adverse Events

Investigators will assess the occurrence of AEs and SAEs at all subject evaluation timepoints during the study. All AEs and SAEs whether volunteered by the subject, discovered by study personnel during questioning, detected through physical examination, clinically significant laboratory test, or other means, will be recorded in the subject's medical record and on the AEs CRF and, when applicable, on the Serious Adverse Event Report Form.

Each recorded AE or SAE will be described by its duration (ie, start and end dates), severity, regulatory seriousness criteria (if applicable), suspected relationship to the investigational product, and any actions taken.

# 11.4.2. Adverse Event Reporting Period

All AEs whether serious or non-serious, will be documented from the time signed and dated ICF is obtained until 30 days following the last dose of study drug (ibrutinib/placebo or prednisone) or the start date of a new therapy for cGVHD. The occurrence of AE at the time the ICF is signed until first dose should be recorded under medical history in the eCRF form. All medical occurrences after the first dose of study drug until 30 days after the last dose of study drug that meet the AE definition must be recorded as AEs in the eCRF. SAEs will be reported to the Sponsor Drug Safety via an SAE reporting form and will be recorded in the eCRF from the time of ICF signing. Serious adverse events reported after 30 days following the last dose of study drug should also be reported if considered related to study drug. Resolution information after 30 days should be provided.

Progression of cGVHD should NOT be reported as an event term, but instead symptoms/clinical signs of disease progression may be reported (see Section 11.1.1).

All AEs, regardless of seriousness, severity, or presumed relationship to study drug, must be recorded using medical terminology in the source document. All records will need to capture the details of the duration and the severity of each episode, the action taken with respect to the study drug, investigator's evaluation of its relationship to the study drug, and the event outcome. Whenever possible, diagnoses should be given when signs and symptoms are due to a common etiology (eg, cough, runny nose, sneezing, sore throat, and head congestion should be reported as "upper respiratory infection"). Investigators must record in the CRF their opinion concerning the relationship of the AE to study therapy. All measures required for AE management must be recorded in the source document and reported according to Sponsor instructions.

All deaths should be reported with the primary cause of death as the AE term, as death is typically the outcome of the event, not the event itself. Autopsy and postmortem reports must be forwarded to the Sponsor, or designee, as outlined above, if allowed per local regulatory guidelines.

If a death occurs within 30 days after the last dose of study drug, the death must be reported to the Sponsor as a SAE.

# 11.4.3. Expediting Reporting Requirements for Serious Adverse Events

All SAEs (initial and follow-up information) will be reported on the Serious Adverse Event Report Form and sent via email or fax to Pharmacyclics Drug Safety, or designee, within 24 hours of the discovery of the event or information. Pharmacyclics may request follow-up and other additional information from the investigator (eg, hospital admission/discharge notes and laboratory results). The contact information (phone, email and fax) for Pharmacyclics Drug Safety can be found on the Serious Adverse Event Report Form and instructions.

All SAEs that have not resolved by the end of the study, or that have not resolved upon discontinuation of the subject's participation in the study, must be followed until any of the following occurs:

- The event resolves
- The event stabilizes
- The event returns to baseline, if a baseline value/status is available
- The event can be attributed to agents other than the study drug or to factors unrelated to study conduct
- It becomes unlikely that any additional information can be obtained (subject or health care practitioner refusal to provide additional information, lost to follow up after demonstration of due diligence with follow-up efforts)

The Sponsor assumes responsibility for appropriate reporting of AEs to the regulatory authorities and governing bodies according to the local regulations.

The investigator (or Sponsor where required) must report these events to the appropriate Independent Ethics Committee/Institutional Review Board (IEC/IRB) that approved the protocol unless otherwise required and documented by the IEC/IRB.

# 11.4.4. Pregnancy

Before study enrollment, subjects must agree to take appropriate measures to avoid pregnancy. However, should a pregnancy occur in a female study subject, consent to provide follow-up information regarding the outcome of the pregnancy and the health of the infant until 30 days old will be requested.

A female subject or female partner of a male subject must immediately inform the investigator if she becomes pregnant from the time of consent to 90 days after the last dose of study drug (s). Any female subjects receiving study drug (s) who become pregnant must immediately discontinue study drug. The investigator should counsel the subject, discussing any risks of continuing the pregnancy and any possible effects on the fetus.

Although pregnancy itself is not regarded as an AE, the outcome will need to be documented. Any pregnancy occurring in a female subject or female partner of a male subject must be reported from the time of first dose up until 90 days after the last dose of study drug (s). Any occurrence of pregnancy must be recorded on the Pregnancy Report Form Part I and sent via email or fax to Pharmacyclics Drug Safety, or designee, within 24 hours of learning of the event. All pregnancies will be followed for outcome, which is defined as elective termination of the pregnancy, miscarriage, or delivery of the fetus. For pregnancies with an outcome of live birth, the newborn infant will be followed until 30 days old by completing the Pregnancy Report Form Part II. Any congenital anomaly/birth defect noted in the infant must be reported as a SAE.

# 11.4.5. Other Malignancies

All new malignant tumors including solid tumors, skin malignancies and hematologic malignancies will be reported for the duration of study treatment and during any protocol-specified follow-up periods including post-progression follow-up for OS. If observed, enter data in the corresponding eCRF. Relapse of underlying malignancy will not be considered a new malignancy.

## 11.4.6. Eye-Related Adverse Events

New or worsening eye-related symptoms that are Grade 2 or higher, or a symptom that was Grade 2 or higher at baseline worsens, should be evaluated by an ophthalmologist whose findings should be reported on the ophthalmologic eCRF.

# 11.4.7. Adverse Events of Special Interest (AESI)

Specific AEs, or groups of AEs, will be followed as part of standard safety monitoring activities by the Sponsor. These events (regardless of seriousness) should be reported on the Serious Adverse Event Report Form and sent via email or fax to Pharmacyclics Drug Safety, or designee, within 24 hours of awareness.

# 11.4.7.1. Major Hemorrhage

Major hemorrhage is defined as any of the following:

- Any treatment-emergent hemorrhagic AEs of Grade 3 or higher\*
- Any treatment-emergent serious adverse events of bleeding of any grade
- Any treatment-emergent central nervous system hemorrhage/hematoma of any grade

Events meeting the definition of major hemorrhage will be captured as an event of special interest according to Section 11.4.7 above.

## 12. STUDY ADMINISTRATION AND INVESTIGATOR OBLIGATIONS

## 12.1. Regulatory and Ethical Compliance

This clinical study was designed and will be implemented in accordance with the protocol, the ICH Harmonized Tripartite Guidelines for Good Clinical Practices, with applicable local regulations (including US Code of Federal Regulations [CFR] Title 21 and European Directive 2001/20/EC), and with the ethical principles laid down in the Declaration of Helsinki.

<sup>\*</sup>All hemorrhagic events requiring transfusion of red blood cells should be reported as Grade 3 or higher AE per CTCAE v4.03.

# 12.2. Institutional Review Board (IRB), Research Ethics Board (REB) and Independent Ethics Committee (IEC) Approval

The investigator will submit this protocol, the ICF, IB, and any other relevant supporting information (eg, all advertising materials or materials given to the subject during the study) to the appropriate IRB/REB/IEC for review and approval before study initiation. Amendments to the protocol and ICF must also be approved by the IRB/REB/IEC before the implementation of changes in this study.

The investigator is responsible for providing the IRB/REB/IEC with any required information before or during the study, such as SAE expedited reports or study progress reports.

The IRB/REB/IEC must comply with current United States (US) regulations (§21 CFR 56) as well as country-specific national regulations and/or local laws.

The following documents must be provided to Pharmacyclics or its authorized representative before entering subjects in this study: (1) a copy of the IRB/REB/IEC letter that grants formal approval; and (2) a copy of the IRB/REB/IEC-approved ICF.

## 12.3. Informed Consent

The ICF and process must comply with the US regulations (§ 21 CFR Part 50) as well as country specific national regulations and/or local laws. Parental permission will be obtained for subjects who are below the age of legal consent and assent procedures for minors will follow country specific national regulations. The ICF will document the study-specific information the investigator or his/her designee provides to the subject and the subject's agreement to participate.

The investigator or designee (designee must be listed on the Delegation of Authority log), **must** explain in terms understandable to the subject the purpose and nature of the study, study procedures, anticipated benefits, potential risks, possible AEs, and any discomfort participation in the study may entail. This process must be documented in the subject's source record. Each subject must provide a signed and dated ICF before any study-related (nonstandard of care) activities are performed. The original and any amended signed and dated consent forms must remain in each subject's study file at the study site and be available for verification by study monitors at any time. A copy of each signed consent form must be given to the subject at the time that it is signed by the subject.

# 12.4. Quality Control and Quality Assurance

Sponsor shall implement and maintain quality control and quality assurance procedures to ensure that the study is conducted and data are generated, documented and reported in compliance with the protocol, GCP, and applicable regulatory requirements. This study shall be conducted in accordance with the provisions of the Declaration of Helsinki (October 2008) and all revisions thereof, and in accordance with the Food and Drug Administration (FDA) regulations (21 CFR

Parts 11, 50, 54, 56, and 312, Subpart D – Responsibilities of Sponsors and investigators) and with the ICH guidelines on GCP (ICH E6).

## 12.5. Protected Subject Health Information Authorization

Information on maintaining subject confidentiality in accordance to individual local and national subject privacy regulations must be provided to each subject as part of the informed consent process (refer to Section 7.1.1.1), either as part of the ICF or as a separate signed document (for example, in the US, a site-specific HIPAA consent may be used). The investigator or designee **must** explain to each subject that for the evaluation of study results, the subject's protected health information obtained during the study may be shared with Pharmacyclics and its designees, regulatory agencies, and IRBs/REBs/IECs. As the study Sponsor, Pharmacyclics will not use the subject's protected health information or disclose it to a third party without applicable subject authorization. It is the investigator's or designee's responsibility to obtain written permission to use protected health information from each subject. If a subject withdraws permission to use protected health information, it is the investigator's responsibility to obtain the withdrawal request in writing from the subject **and** to ensure that no further data will be collected from the subject. Any data collected on the subject before withdrawal will be used in the analysis of study results.

During the review of source documents by the monitors or auditors, the confidentiality of the subject will be respected with strict adherence to professional standards and regulations.

## 12.6. Study Files and Record Retention

The investigator **must** keep a record of **all** subjects who have consented to enroll in the study. For those subjects subsequently excluded from enrollment, the reason(s) for exclusion is to be recorded.

The investigator/study staff must maintain adequate and accurate records to enable the conduct of the study to be fully documented and the study data to be subsequently verified. Essential documentation includes, but is not limited to, the IB, signed protocols and amendments, IRB/REB/IEC approval letters (dated), signed Form FDA 1572 and Financial Disclosures, signed ICFs (including subject confidentiality information), drug dispensing and accountability records, shipping records of investigational product and study-related materials, signed (electronically), dated and completed case report forms (CRFs), and documentation of CRF corrections, SAE forms transmitted to Pharmacyclics and notification of SAEs and related reports, source documentation, normal laboratory values, decoding procedures for blinded studies, curricula vitae for study staff, and all relevant correspondence and other documents pertaining to the conduct of the study.

All essential documentation will be retained by the investigator for at least 2 years after the date the last marketing application is approved for the drug for the indication for which it is being investigated and until there are no pending or contemplated marketing applications; or, if no
application is to be filed or if the application is not approved for such indication, until 2 years after formal discontinuation of clinical development of the drug.

The investigator must notify Pharmacyclics and obtain written approval from Pharmacyclics before destroying any clinical study documents or images (eg, scan, radiograph, ECG tracing) at any time. Should an investigator wish to assign the study records to another party or move them to another location, advance written notice will be given to Pharmacyclics. Pharmacyclics will inform the investigator of the date that study records may be destroyed or returned to Pharmacyclics.

Pharmacyclics must be notified in advance of, and Pharmacyclics must provide express written approval of, any change in the maintenance of the foregoing documents if the investigator wishes to move study records to another location or assign responsibility for record retention to another party. If the investigator cannot guarantee the archiving requirements set forth herein at his or her study site for all such documents, special arrangements must be made between the investigator and Pharmacyclics to store such documents in sealed containers away from the study site so that they can be returned sealed to the investigator for audit purposes.

#### 12.7. Case Report Forms and Record Maintenance

The case report forms will be used to collect the clinical study data and must be completed for each enrolled subject with all required study data accurately recorded such that the information matches the data contained in medical records (eg, physicians' notes, nurses' notes, clinic charts and other study-specific source documents). Authorized study site personnel (ie, listed on the Delegation of Authority log) will complete CRFs designed for this study according to the completion guidelines that will be provided. The investigator will ensure that the CRFs are accurate, complete, legible, and completed within a reasonable period of time. At all times, the investigator has final responsibility for the accuracy and authenticity of all clinical data.

The CRFs exists within an electronic data capture (EDC) system with controlled access managed by Pharmacyclics or its authorized representative for this study. Study staff will be appropriately trained in the use of CRFs and application of electronic signatures before the start of the study and before being given access to the EDC system. Original data and any changes of data will be recorded using the EDC system, with all changes tracked by the system and recorded in an electronic audit trail. The investigator attests that the information contained in the CRFs is true by providing electronic signature within the EDC system. After database lock, the investigator will receive a copy of the subject data (eg, paper, CD, or other appropriate media) for archiving at the study site.

#### 12.8. Investigational Study Drug Accountability

Ibrutinib and any comparator used must be kept in a locked limited access room. The study drug must not be used outside the context of the protocol. Under no circumstances should the investigator or other site personnel supply ibrutinib or comparator to other investigators,

subjects, or clinics or allow supplies to be used other than as directed by this protocol without prior authorization from Pharmacyclics.

Accountability records for ibrutinib and any comparator must be maintained and readily available for inspection by representatives of Pharmacyclics and are open to inspections by regulatory authorities at any time.

An Investigational Drug Accountability Log must be used for drug accountability. For accurate accountability, the following information must be noted when drug supplies are used during the study:

- 1. Study identification number (PCYC-1140-IM)
- 2. Subject identification number
- 3. Lot number(s) of ibrutinib or placebo dispensed for that subject
- 4. Date and quantity of drug dispensed
- 5. Any unused drug returned by the subject

At study initiation, the monitor will evaluate and approve the site's procedure for investigational product disposal/destruction to ensure that it complies with Pharmacyclics' requirements. If the site cannot meet Pharmacyclics' requirements for disposal/destruction, arrangements will be made between the site and Pharmacyclics or its representative, for return of unused investigational product. Before disposal/destruction, final drug accountability and reconciliation must be performed by the monitor.

All study supplies and associated documentation will be regularly reviewed and verified by the monitor.

#### 12.9. Study Monitoring/Audit Requirements

Representatives of Pharmacyclics or its designee will monitor this study until completion. Monitoring will be conducted through personal visits with the investigator and site staff, remote monitoring, as well as any appropriate communications by mail, fax, email, or telephone. The purpose of monitoring is to ensure that the study is conducted in compliance with the protocol, standard operating procedures (SOPs), and other written instructions and regulatory guidelines, and to ensure the quality and integrity of the data. This study is also subject to reviews or audits.

To assure the accuracy of data collected in the CRFs, it is mandatory that the monitor/auditor have access to all original source documents, including all electronic medical records (EMR) at reasonable times and upon reasonable notice. If access to the EMR cannot be granted to the monitor, the site must ensure that all certified copies of documents are available during monitoring visits for all screened and enrolled subjects. During the review of source documents, every effort will be made to maintain the anonymity and confidentiality of all subjects during

this clinical study. However, because of the experimental nature of this treatment, the investigator agrees to allow the IRB/REB/IEC, representatives of Pharmacyclics, its designated agents and authorized employees of the appropriate Regulatory Authority to inspect the facilities used in this study and, for purposes of verification, allow direct access to the hospital or clinic records of all subjects enrolled into this study. A statement to this effect will be included in the informed consent and permission form authorizing the use of protected health information.

Pharmacyclics or its authorized representative may perform an audit at any time during or after completion of this study. All study-related documentation must be made available to the designated auditor. In addition, a representative of the FDA or other Regulatory Agencies may choose to inspect a study site at any time before, during, or after completion of the clinical study. In the event of such an inspection, Pharmacyclics will be available to assist in the preparation. All pertinent study data should be made available as requested to the Regulatory Authority for verification, audit, or inspection purposes.

#### 12.10. Investigator Responsibilities

A complete list of investigator responsibilities are outlined in the clinical trial research agreement and the Statement of Investigator Form FDA 1572, both of which are signed by the investigator before commencement of the study. In summary, the investigator will conduct the study according to the current protocol; will read and understand the IB; will obtain IRB/REB/IEC approval to conduct the study; will obtain informed consent from each study participant; will maintain and supply to the Sponsor or designee, auditors and regulatory agencies adequate and accurate records of study activity and drug accountability for study-related monitoring, audits, IRB/REB/IEC reviews and regulatory inspections; will report SAEs to the Sponsor or designee and IRB/REB/IEC according to the specifics outlined in this protocol; will personally conduct or supervise the study; and will ensure that colleagues participating in the study are informed about their obligations in meeting the above commitments.

#### 12.11. Sponsor Responsibilities

A complete list of the Sponsor responsibilities is outlined in the clinical trial research agreement and in the laws and regulation of the country in which the research is conducted. In summary, the Sponsor will select qualified investigators, provide them with the information they need to properly conduct the study, ensure adequate monitoring of the study, conduct the study in accordance with the general investigational plan and protocols and promptly inform investigators, health and regulatory agencies/authorities as appropriate of significant new adverse effects or risks with respect to the drug.

#### 12.12. Financial Disclosure

A separate financial agreement will be made between each principal investigator and Pharmacyclics or its authorized representative before the study drug is delivered.

For this study, each investigator and sub-investigator (as designated on the Form FDA1572) will provide a personally signed Financial Disclosure Form in accordance with § 21 CFR 54. Each investigator will notify Pharmacyclics or its authorized representative of any relevant changes in financial disclosure information during the conduct of the study and for 1 year after the study has been completed.

#### 12.13. Liability and Clinical Trial Insurance

In the event of a side effect or injury, appropriate medical care as determined by the investigator/designee will be provided.

The ICF will include a description of treatment in the event of a study related injury and handling of the costs associated therewith, incorporating country-specific national regulations and/or local laws. Financial compensation for lost wages, disability or discomfort due to the study is not available.

Clinical trial insurance has been undertaken according to the laws of the countries where the study will be conducted. An insurance certificate will be made available to the participating sites at the time of study initiation.

#### 12.14. Protocol Amendments

Pharmacyclics will initiate any change to the protocol in a protocol amendment document. The amendment will be submitted to the IRB/REB/IEC together with, if applicable, a revised model ICF. Written documentation of IRB/REB/IEC and required site approval must be received by Pharmacyclics before the amendment may take effect at each site. Additionally, under this circumstance, information on any change in risk and/or change in scope must be provided to subjects already actively participating in the study, and they must read, understand and sign each revised ICF, confirming willingness to remain in the trial.

No other significant or consistent change in the study procedures, except to eliminate an immediate hazard, shall be effected without the mutual agreement of the investigator and Pharmacyclics.

#### 12.15. Publication of Study Results

Pharmacyclics may use the results of this clinical study in registration documents for Regulatory Authorities in the US or abroad. The results may also be used for papers, abstracts, posters, or other material presented at scientific meetings or published in professional journals or as part of an academic thesis by an investigator. In all cases, to avoid disclosures that could jeopardize proprietary rights and to ensure accuracy of the data, Pharmacyclics reserves the right to preview all manuscripts and abstracts related to this study, allowing Pharmacyclics sufficient time to make appropriate comments before submission for publication.

In most cases, the investigators at the sites with the highest accruals of eligible subjects shall be listed as lead authors on manuscripts and reports of study results. The medical monitor, study director and/or lead statistician may also be included in the list of authors. This custom can be adjusted upon mutual agreement of the authors and Pharmacyclics and in accordance with current standards for authorship as recorded in professional conference and journal submission instructions.

#### 12.16. Study Discontinuation

The Sponsor reserves the right to terminate the study at any time. Should this be necessary, both the Sponsor and the investigator will arrange discontinuation procedures. In terminating the study, the Sponsor and the investigator will assure that adequate consideration is given to the protection of the subjects' interests.

#### 13. REFERENCES

Allen JL, Tata PV, Fore MS et al. Increased BCR responsiveness in B cells from patients with chronic GVHD. Blood. 2014;123:2108-15.

Anasetti C, Logan BR, Lee SJ, et al. Increased incidence of chronic graft-versus-host disease (GVHD) and no survival advantage with filgrastim-mobilized peripheral blood stem cells (PBSC) compared to bone marrow (BM) transplants from unrelated donors: results of Blood and Marrow Transplant Clinical Trials Network (BMT CTN) Protocol 0201, a Phase III, prospective, randomized trial. ASH Annual Meeting Abstracts 2011;118: Abstract 1.

Appelbaum FR, Haematopoietic cell transplantation as immunotherapy. Nature 2001; 411:385-9.

Arai S, Jagasia M, Storer B, et al. Global and organ-specific chronic graft-versus-host disease severity according to the 2005 NIH Consensus Criteria. Blood. 2011;118:4242-49.

Arora M, Wagner JE, Davies SM, et al. Randomized clinical trial of thalidomide, cyclosporine, and prednisone versus cyclosporine and prednisone as initial therapy for chronic graft-versus-host disease. Biol Blood Marrow Transplant. 2001;7:265-73.

Baird K, Pavletic SZ. Chronic graft versus host disease. Curr Opin Hematol. 2006;13:426-435.

Brunton LL, Chabner BA, Knollmann BC (Eds). The Pharmacological Basis of Therapeutics, 12th ed. McGraw Hill, New York 2011. p.1216.

Carpenter PA, Kitko CL, Elad S, et al. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: V. The 2014 Ancillary Therapy and Supportive Care Working Group Report. Biol Blood Marrow Transplant. 2015;21:1167-87.

Child CG, Turcotte JG. "Surgery and portal hypertension". In Child CG. The liver and portal hypertension. Philadelphia: Saunders. 1964. pp. 50-64.

Dignan FL, Amrolia P, Clark A, et al. Diagnosis and management of chronic graft-versus-host disease. Br J Haematol. 2012;158:46-61.

Dubovsky JA, Beckwith KA, Natarajan G, et al. Ibrutinib is an irreversible molecular inhibitor of ITK driving a Th1-selective pressure in T lymphocytes. Blood 2013;122:2539–49.

Filipovich AH, Weisdorf D, Pavletic S, et al. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: I. Diagnosis and staging working group report. Biol Blood Marrow Transplant 2005;11:945-956.

Flowers ME, Martin PJ. How we treat chronic graft-versus-host disease. Blood. 2015;125:606-15. Review.

Flowers ME, Inamoto Y, Carpenter PA, et al. Comparative analysis of risk factors for acute graft-versus-host disease and for chronic graft-versus-host disease according to National Institutes of Health consensus criteria. Blood. 2011;117:3214-9.

Flynn R, Du J, Veenstra RG, et al. Increased T follicular helper cells and germinal center B cells are required for cGVHD and bronchiolitis obliterans. Blood. 2014;123:3988-98.

Gilman AL, Schultz KR, Goldman FD, et al. Randomized trial of hydroxychloroquine for newly diagnosed chronic graft-versus-host disease in children: a Children's Oncology Group study. Biol Blood Marrow Transplant. 2012;18:84-91.

Hale GA, Shrestha S, Le-Rademacher J, et al. Alternate donor hematopoietic cell transplantation (HCT) in non-Hodgkin lymphoma using lower intensity conditioning: A Report from the CIBMTR. Biol Blood Marrow Transplant 2012;18:1036-1043.

Herman SE, Gordon AL, Hertlein E, et al. Bruton tyrosine kinase represents a promising therapeutic target for treatment of chronic lymphocytic leukemia and is effectively targeted by PCI-32765. Blood. 2011;117:6287-96.

Holler E. Risk assessment in haematopoietic stem cell transplantation: GvHD prevention and treatment. Best Pract Res Clin Haematol. 2007;20:281-294.

International Conference on Harmonization (ICH) Guideline for Industry: Clinical Safety Data Management: Definitions and Standards for Expedited Reporting (ICH-E2A). March 1995.

International Conference on Harmonisation (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use: ICH Harmonised Tripartite Guideline: Guidance for Good Clinical Practice (ICH-E6)(R1). June 1996.

Inamoto Y, Savani BN, Shaw BE, et al. Secondary solid cancer screening following hematopoietic cell transplantation. Bone Marrow Transplant. 2015.[Epub ahead of print].

Investigator's Brochure. Ibrutinib. Version 12.0: 11 December 2018. Pharmacyclics LLC; Janssen Research & Development, LLC.

Jacobsohn DA, Kurland BF, Pidala J, et al. Correlation between NIH composite skin score, patient-reported skin score, and outcome: results from the Chronic GVHD Consortium. Blood. 2012;120:2545-52.

Jagasia MH, Greinix HT, Arora M, et al. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: I. The 2014 Diagnosis and Staging Working Group report. Biol Blood Marrow Transplant. 2015;21:389-401.

Johnston HF, Xu Y, Racine JJ, et al. Administration of anti-CD20 mAb is highly effective in preventing but ineffective in treating chronic graft-versus-host disease while preserving strong graft-versus-leukemia effects. Biol Blood Marrow Transplant. 2014;20:1089-103.

Koc S, Leisenring W, Flowers ME, et al. Thalidomide for treatment of patients with chronic graft-versus-host disease. Blood. 2000;96:3995-6.

Koc S, Leisenring W, Flowers ME, et al. Therapy for chronic graft-versus-host disease: a randomized trial comparing cyclosporine plus prednisone versus prednisone alone. Blood 2002;100:48-51.

Lee SJ, Wolff D, Kitko C, et al. Measuring Therapeutic Response in Chronic Graft-versus-Host Disease. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: IV. The 2014 Response CriteriaWorking Group Report. Biol Blood Marrow Transplant. 2015;21:984-999.

Lee JW, Deeg HJ. Prevention of chronic GVHD. Best Pract Res Clin Haematol. 2008;21:259-270.

Lee SJ, Vogelsang G, Flowers ME. Chronic graft-versus-host disease. Biol Blood Marrow Transplant. 2003;9:215-233.

Majhail NS, Rizzo JD, Lee SJ, et al. Recommended screening and preventive practices for long-term survivors after hematopoietic cell transplantation. Biol Blood Marrow Transplant. 2012;18:348–71.

Martin PJ, Inamoto Y, Carpenter PA, Lee SJ, Flowers ME. Treatment of chronic graft-versus-host disease: Past, present and future. Korean J Hematol. 2011;46(3):153-63.

Martin PJ, Storer BE, Rowley SD, et al. Evaluation of mycophenolate mofetil for initial treatment of chronic graft-versus-host disease. Blood 2009;113:5074-82.

Miklos DB, Kim H, Zorn E, et al. Antibody Response to DBY minor histocompatibility antigen is induced after allogenic stem cell transplantation and in normal female donors. Blood 2004;103:353-359.

Miklos DB, Kim HT, Miller KH et al. Antibody responses to H-Y minor histocompatibility antigens correlate with chronic graft-versus-host disease and disease remission. Blood 2005;105:2973-2978.

NCI Common Terminology Criteria for Adverse Events. Version 4.03. 2010.

Olivieri A, Cimminiello M, Corradini P, et al. Long-term outcome and prospective validation of NIH response criteria in 39 patients receiving imatinib for steroid-refractory chronic GVHD. Blood. 2013;122:4111-8.

Pan Z, Scheerens H, Li SJ, et al. Discovery of selective irreversible inhibitors for Bruton's tyrosine kinase. ChemMedChem 2007;2:58-61.

Pasquini MC, Zhu X. Current uses and outcomes of hematopoietic stem cell transplantation: CIBMTR Summary Slides, 2015 (http://www.cibmtr.org).

Pavletic SZ, Martin P, Lee SJ, et al. Measuring therapeutic response in chronic graft-versus-host-disease: national institutes of health consensus development project on criteria for clinical trials in chronic graft-versus-host-disease: IV. Response criteria working group report. Biol. Blood Marrow Transplant. 2006;12:252-66.

Perez-Simon JA, Kottaridis PD, Martino R, et al. Nonmyeloablative transplantation with or without alemtuzumab: comparison between 2 prospective studies in patients with lymphoproliferative disorders. Blood. 2002;100:3121-3127.

Pidala J, Kurland B, Chai X, et al. Patient-reported quality of life is associated with severity of chronic graft-versus-host disease as measured by NIH criteria: report on baseline data from the Chronic GVHD Consortium. Blood. 2011;117:4651-4657.

Pugh RN, Murray-Lyon IM, Dawson L, et al. "Transection of the oesophagus for bleeding oesophageal varices". The British Journal of Surgery, 1973;60: 646-9.

RAYOS (prednisone) delayed-release tablets. Prescribing Information. Horizon Pharma USA Inc. Deerfield, IL; 2013.

Sahaf B, Arai S, Otani J, et al. Rituximab Provides Steroid-Sparing Therapy in New-Onset Chronic Graft-Versus-Host Disease. ASBMT 2013;19,S140. Abstract 55.

Sarantopoulos S, Blazar BR, Cutler C, et al. B cells in chronic graft-versus-host disease. Biol Blood Marrow Transplant. 2015;21:16-23.

Sarantopoulos S, Stevenson KE, Kim HT, et al. Altered B-cell homeostasis and excess BAFF in human chronic graft-versus-host disease. Blood. 2009;113:3865-3874.

Shimabukuro-Vornhagen A, Hallek MJ, Storb RF, von Bergwelt-Baildon MS. The role of B cells in the pathogenesis of graft-versus-host disease. Blood. 2009;114:4919-4927.

Shulman HM, Kleiner D, Lee SJ, et al. Histopathologic diagnosis of chronic graft-versus-host disease: National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: II. Pathology Working Group Report. Biol Blood Marrow Transplant 2006;12:31-47.

Smith EM, Pang H, Cirrincione C, et al. Effect of duloxetine on pain, function, and quality of life among patients with chemotherapy-induced painful peripheral neuropathy: a randomized clinical trial. JAMA. 2013;309:1359–67.

Sullivan KM, Witherspoon RP, Storb R, et al. Prednisone and azathioprine compared with prednisone and placebo for treatment of chronic graft-v-host disease: prognostic influence of prolonged thrombocytopenia after allogeneic marrow transplantation. Blood 1988;72:546-54.

Syrjala KL, Martin PJ, Lee SJ. Delivering care to long-term adult survivors of hematopoietic cell transplantation. J Clin Oncol. 2012;30:3746-51.

Thomas ED, Lochte HL Jr, Lu WC, Ferrebee JW. Intravenous infusion of bone marrow in patients receiving radiation and chemotherapy. N Engl J Med. 1957; 257:491-6.

USPI IMBRUVICA® (ibrutinib) revised August 2017, Pharmacyclics LLC.

Wolff D, Schleuning M, von Harsdorf S, et al. Consensus Conference on Clinical Practice in Chronic GVHD: Second-Line Treatment of Chronic Graft-versus-Host Disease. Biol Blood Marrow Transplant.2011;17:1-17.

#### 14. <u>APPENDICES</u>

06 February 2019 FINAL

Appendix A. Schedule of Assessments

| | | | | | | | | | | | Late effects |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | Post-Treatment/ | atment/ | surveillance |
| | Screening Phase | | | | Tre | Treatment Phase | | | Follow-up Phase | p Phase | (adolescents only) |
| | | | | | | | | End-of-<br>Treatment | Response<br>Follow-up | | Month 12, 24, 36, 48, and 60 |
| | | | | | 9, 13, 17, | 37, 49 | Progressive | Visit<br>(30 days<br>from | Visits<br>(Until<br>progressive | Survival | |
| Study Weeks | | Ţ | 2 | S | 21, 25<br>q4 weeks | q12 weeks | Disease<br>Visit | last dose of<br>study drug) | disease) | Follow-up<br>q12 weeks | |
| Study Day of | | | - | - 10 <del>-</del> | + | - | | | | | |
| Study Windows | -28 days | On time | ime | 1 | ±3 days | $\pm 7 davs$ | anytime | ±7, | ± 7 days | ± 14 days | ± 30 days |
| Administrative Procedures | cedures | | | | | | | | , | | |
| Informed | X | | | | | | | | | | |
| consent/Child | | | | | | | | | | | |
| Assent/Parental permission | | | | | | | | | | | |
| Confirm eligibility | × | qX | | | | | | | | | |
| Randomization | | qX | | | | | | | | | |
| cGVHD diagnosis<br>& staging (NIH) | x | | | | | | | | | | |
| Medical history<br>and demographics | X | | | | | | | | | | |
| Malignancy relapse<br>evaluation | x | | | | | | | | | | |
| Infection<br>surveillance | x | 2 5 | 2 | | | | | | | 35 | |
| GVHD/Transplant<br>history | x | | | | | | | | | | |
| Physical exam | pХ | Xª | Xª | Xª | Xg | Xg | вX | Xg | ęX | | |
| KPS/Lansky status | x | X | | X | x | X | x | x | X | | |
| Vital signs | X | X | X | X | X | X | X | X | X | | |
| Survival | | | | | | | | | | X | |
| ECG. | X | | Xc | | If cl | If clinically indicated (eg, subjects with palpitations, lightheadedness) | (eg, subjects wit | h palpitations, | lightheadednes | s) | |

06 February 2019 FINAL

| | Screening Phase | S 5 | | | Tre | Treatment Phase | | | Post-Treatment/<br>Follow-up Phase | atment/<br>p Phase | Late effects<br>surveillance<br>(adolescents only) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Weeks | | - | | vo | 9, 13, 17,<br>21, 25<br>a4 weeks | 37, 49<br>q12 weeks | Progressive<br>Disease<br>Visit | End-of-<br>Treatment<br>Visit<br>(30 days<br>from<br>last dose of<br>study drug) | Response Follow-up Visits (Until progressive disease) | Survival<br>Follow-up<br>a12 weeks | Month 12, 24, 36, 48, and 60 |
| Study Day of<br>Study Week | | 1 | 1 | 1 | 1 | 1 | | ò | ė. | | |
| Study Windows | -28 days | On time | ime | | ±3 days | $\pm$ 7 days | anytime | ±7, | $\pm$ 7 days | $\pm$ 14 days | $\pm 30 days$ |
| Documentation of<br>height, weight, and<br>Tanner Stage | אַ | | | | E | 3 | | | | 8 | χ |
| Surveillance for late effects (adolescents only) | · K | | | | | | | | | | ' <sub>[X</sub> |
| Clinical Laboratory Assessments | Assessments | | | | | | | | | | |
| Hematology | X | Σg | X | X | X | X | X | X | x | Q1 | |
| Serum chemistry | X | Xg | X | X | X | X | X | x | X | | |
| Coagulation (PT,<br>INR,<br>and aPTT) | ĸ | | | | | | | | | | |
| Pregnancy test <sup>d</sup> | × | × | | | | | | | | . 8 | |
| Hepatitis serologies<br>and/or PCR | x | | | | | | | | | | |
| Quantitative serum<br>immunoglobulins<br>(IgA, IgG and IgM) | | X | | | Weeks 13, 25 | x | x | x | | | |
| PK/PD, T/B/NK<br>cell counts,<br>biomarkers <sup>f</sup> | Pleas | e see A | ppendi | x B for | r sample requirer | Please see Appendix B for sample requirements and timing for these assays | for these assays | | | | |
| Efficacy Assessments | ts | | | | | | | | | | |
| cGVHD activity<br>assessment<br>(NIH Form) | <sub>¥</sub> X | | | x | Weeks 13,<br>25 <sup>h</sup> | чх | x | $\mathbf{x}_1$ | x | | |
| cGVHD response | | | | x | Weeks 13,<br>25 <sup>h</sup> | $\mathbf{x}^{\mathbf{p}}$ | x | $\mathbf{x}_{\mathbf{l}}$ | x | | |

| | | | | | 1 | l | | | Post-Treatment/ | atment/ | Late effects<br>surveillance |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening Phase | | | | Tre | Treatment Phase | | | Follow-up Phase | p Phase | (adolescents only) |
| | | | N. | | | | | End-of-<br>Treatment<br>Visit<br>(30 days | Response<br>Follow-up<br>Visits<br>(Until | | Month 12, 24, 36, 48, and 60 |
| Study Weeks | | - | 2 | vo | 9, 13, 17,<br>21, 25<br>94 weeks | 37, 49<br>q12 weeks | Progressive<br>Disease<br>Visit | from<br>last dose of<br>study drug) | progressive<br>disease)<br>a12 weeks <sup>m</sup> | Survival<br>Follow-up<br>a12 weeks | |
| Study Day of<br>Study Week | | 1 | - | 1 | | 1 | | à | | | |
| Study Windows | -28 days | On time | me | | ±3 days | $\pm$ 7 days | anytime | $\pm$ 7 days | lays | $\pm 14 days$ | $\pm 30 days$ |
| Lee cGVHD<br>Symptom Scale/<br>SF-36 e | <sup>4</sup> X | | | × | Weeks 13,<br>25 <sup>h</sup> | vх | x | $\mathbf{x}_{l}$ | × | (x) | м |
| FEV1 by<br>spirometry <sup>h</sup> | X | | | | Weeks 13,<br>25 <sup>h</sup> | хp | x | x | x | | |
| Corticosteroid requirements | x | X | X | X | X | X | x | x | × | | |
| Ongoing Subject Assessments | sessments | | | | | | | | | | |
| Concomitant<br>medications | х | 30 day | rs prior | r to Inf | ormed Consent t | o 30 days after la<br>prednisone | 30 days prior to Informed Consent to 30 days after last dose of ibrutinib/placebo or prednisone | ib/placebo or | | | |
| Prednisone dosing<br>changes – phone<br>contacts | м | Conti | nuonu | from h | nformed Consen | nt to 30 days after<br>or prednisone | Continuous from Informed Consent to 30 days after last dose of ibrutinib/placebo or prednisone | inib/placebo | | | |
| Adverse events | X | Conti | snonu | from Ir | nformed Consen | nt to 30 days after<br>or prednisone | Continuous from Informed Consent to 30 days after last dose of ibrutinib/placebo or prednisone | inib/placebo | | | |
| Study Drug Admini | Study Drug Administration and Dispensation | sation | | | | | | | | 9.0 | |
| Prednisone<br>1 mg/kg/day | | Disp | ensed | Continon West | Continuous daily dosing Dispensed on Week 1 D1, Week 5 and every on treatment visit thereafter | ng<br>and every on<br>er | | | | | |
| Ibrutinib/Placebo<br>420 mg PO | | Disp | ensed | Contin<br>on Wet<br>treatm | Continuous daily dosing Dispensed on Week 1 D1, Week 5 and every on treatment visit thereafter | ng<br>and every on<br>er | | | | | |
| Drug diary dispensing, review, and drug accountability | | | Ö | ontinuc | Continuous throughout study | ndy | , x | , x | | | |

Abbreviations: AEs = adverse events; aPTT = activated partial thromboplastin time; ECG = electrocardiogram; KPS = Karnofsky Performance Status; EOT = end-of-treatment; INR = international normalized ratio; PD = pharmacodynamic; PK = pharmacokinetics; PO = orally; PT = prothrombin time; q4 weeks = every 4 weeks; q8 weeks = every 8 weeks; q12 weeks = every 12 weeks

FINAL

### Footnote:

- The physical examination will include, height (at Screening for adults, and at Screening and annually for subjects <22 years of age at the time of enrollment), weight, and examination per clinical practice.
- b Confirm eligibility and randomize within 3 days prior to first dose.
- ECG's may be performed at the investigator's discretion, particularly in subjects with arrhythmic symptoms (eg, palpitations, lightheadedness) or new onset of dyspnea. At Week 2 12-lead ECG (subject in supine position and resting for at least 10 min prior to ibrutinib dose) performed on subjects <22 years of age at
- Women of childbearing potential only. Serum pregnancy test required at Screening and urine pregnancy test required at Day 1 prior to first dose. If the test result is positive, the pregnancy must be ruled out by ultrasound to be eligible.
  - Pharmacokinetic (PK) samples will be drawn for all subjects according to the schedule in Appendix B predose specimen is required. Pharmacodynamic (PD), Lee cGVHD Symptom Scale and SF-36 should be completed prior to any assessments, and before being clinically evaluated by the study nurse or physician.
    - T/B/NK and Biomarker sampling will be performed on selected days. Refer to Appendix B for more details. Hematology and Serum Chemistry may be done within 3 days of Day 1.
- The cGVHD Response assessment, Lee cGVHD Symptom Scale, SF-36, and FEV1 may be done from 7 days prior to Week 25/49 to 21 days after Week 25/49. If FEV1 results are abnormal at Screening FEV1 should be obtained every 12 weeks, and if normal at Screening repeat every 24 weeks. Lung score should be obtained with every cGVHD assessment.
  - Drug diary review and drug accountability only. Must be done at End of Treatment Visit if not already done at Progressive Disease visit.
- Tanner stage and late effects are needed annually up to 60 months post enrollment only for subjects <22yrs of age at enrollment. Adolescents (<22 years of age at the time of enrollment) will be followed for up to 5 years after enrollment and may be rolled-over to a long-term extension study during late-effects follow-up.
  - cGVHD should be evaluated prior to start of prednisone (if initiated during Screening) or prior to Week1 Day 1 start of prednisone and ibrutinib/placebo. cGVHD response assessments and PRO measures at EOT visit need not be repeated if performed within the previous 30 days.
- Subjects in Response follow-up should be evaluated at all pre-specified response assessment time points, including week 5, week 13, week 25, and every 12 weeks afterward

Appendix B. Schedule of Assessments for Pharmacokinetics, Pharmacodynamics, Biomarker and T/B/NK

| Day 1, | | | | | |
|---|---|---|---|---|---|
| Week | Time | Pharmacokinetics | Pharmacodynamics | Biomarkers | T/B/NK |
| Screening | | | | X <sup>€, α</sup> | X |
| 1 | Predose | | X | X €, α, N | X |
| | Predose <sup>a</sup> (trough value) | X | | | |
| | 1h post dose <sup>b</sup> (± 15 min) | X | | | |
| 2 | 2 h post dose <sup>b</sup> (± 15 min) | X | | | |
| | 4 h post dose <sup>b</sup> (± 30 min) | X | | | |
| | 6 h post dose <sup>b</sup> (± 1 h) | X | | | |
| 5 | Predose | | X | X €, α | X |
| 9 | Predose | | X | X €, α, N | X |
| 13 | Predose | | X | X <sup>€</sup> , α | X |
| 17 | Predose | | X | X €, α, N | X |
| 21 | Predose | | X | X <sup>€</sup> , α | X |
| | Predose <sup>a</sup> (trough value) | X | X | X €, α, N | X |
| | 1h post dose <sup>b</sup> (± 15 min) | X | | | |
| 25 | 2 h post dose <sup>b</sup> (± 15 min) | X | | | |
| | 4 h post dose <sup>b</sup> (± 30 min) | X | | | |
| | 6 h post dose <sup>b</sup> (± 1 h) | X | | | |
| 37 | Predose | | | Χ <sup>ε</sup> | X |
| 49 | Predose | | X | X €, α, N | X |
| 73 | Predose | | X | X ε | X |
| 97 | Predose | | X | X <sup>€</sup> , α | X |
| Progressive<br>Disease Visit | | | X | Χ €, α | X |
| Sample Collect | ion Tube Type | NaHep<br>(2mL) | ACD<br>(8.5 mL) | €=EDTA<br>(10 mL), | EDTA<br>(10 ml) |

a Sample collected 24 hours (± 2 hours) after last intake and prior to dosing on that PK day (applies only on days when PK is collected).

The same timepoints as Week 2 and Week 25 PK sample collection will be followed. If ibrutinib/placebo is on hold during scheduled Week 2 and 25 Week PK evaluation, PK testing should be obtained on the next scheduled visit after ibrutinib dose has been stable for 7 days.

Record actual time of sample collection (applies only on days when PK is collected).

#### Appendix C. Karnofsky/Lansky Performance Status

| Karno | fsky Scale (recipient age ≥16 years) | Lansk | y Scale (recipient age <16 years) |
|---|---|---|---|
| Able to | carry on normal activity; no special care | | o carry on normal activity; no special needed |
| 100 | Normal, no complaints, no evidence of disease | 100 | Fully active |
| 90 | Able to carry on normal activity | 90 | Minor restriction in physically strenuous play |
| 80 | Normal activity with effort | 80 | Restricted in strenuous play, tires more easily, otherwise active |
| most p | e to work, able to live at home, cares for<br>ersonal needs, a varying amount of<br>nce is needed | Mild to | o moderate restriction |
| 70 | Cares for self, unable to carry on normal activity or to do active work | 70 | Both greater restrictions of, and less time spent in active play |
| 60 | Requires occasional assistance but is able to care for most needs | 60 | Ambulatory up to 50% of time, limited active play with assistance/supervision |
| 50 | Requires considerable assistance and frequent medical care | 50 | Considerable assistance required for any active play, fully able to engage in quiet play |
| institut | to care for self, requires equivalent of ional or hospital care, disease may be ssing rapidly | Modei | rate to severe restriction |
| 40 | Disabled, requires special care and assistance | 40 | Able to initiate quiet activities |
| 30 | Severely disabled, hospitalization indicated, although death not imminent | 30 | Needs considerable assistance for quiet activity |
| 20 | Very sick, hospitalization necessary | 20 | Limited to very passive activity initiated by others (eg, TV) |
| 10 | Moribund, fatal process progressing rapidly | 10 | Completely disabled, not even passive play |

#### Appendix D. Inhibitors and Inducers of CYP3A

Inhibitors and inducers of CYP3A enzymes are defined as follows. Refer to Section 6.2.1 on instructions for concomitant use of CYP3A inhibitors and inducers with ibrutinib. Further information can be found at the following website: http://medicine.iupui.edu/clinpharm/ddis/main-table/.

| Inhibitors of CYP3A | Inducers of CYP3A |
|---|---|
| Strong inhibitors: | carbamaze |
| indinavir | nevirapine |
| nelfinavir | barbiturates |
| ritonavir | glucocorticoids |
| clarithromycin | modafinil |
| Itraconazole | oxcarbazepine |
| Ketoconazole | pioglitazone |
| nefazodone | troglitazone |
| saquinavir | pioglitazone |
| suboxone | Strong CYP3A inducers |
| telithromycin | avasimibe |
| cobicistat | carbamazepine |
| boceprevir | phenobarbital |
| mibefradil | phenytoin |
| telaprevir | rifabutine |
| troleandomycin | rifampin |
| posaconazole | St. John's Wort |
| voriconazole | St. John S Wort |
| Moderate inhibitors: | |
| aprepitant | |
| amprenavir | |
| amiodarone | |
| atazanavir | |
| ciprofloxacin | |
| isavuconazole | |
| crizotinib | |
| darunavir | |
| dronedarone | |
| erythromycin | |
| diltiazem | |
| fluconazole | |
| fosamprenavir | |
| grapefruit juice | |
| Seville orange juice | |
| verapamil | |
| imatinib | |
| Weak inhibitors: | |
| cimetidine | |
| fluvoxamine | |
| All other inhibitors: | |
| chloramphenicol | |
| delavirdine | |
| gestodene | |
| mifepristone | |
| norfloxacin | |
| star fruit | |
| Tunner 11 days | d. Mr. Johnson d. Const. d. v. Disster |

<sup>&</sup>lt;sup>a</sup> Itraconazole and ketoconazole will be replaced with voriconazole for study subjects

#### Appendix E. Child-Pugh Score for Subjects with Chronic Liver Impairment

| Measure | 1 point | 2 points | 3 points |
|---|---|---|---|
| Total bilirubin, μmol/L (mg/dL) | <34 (<2) | 34-50 (2-3) | >50 (>3) |
| Serum albumin, g/L (g/dL) | >35 (>3.5) | 28-35 (2.8-3.5) | <28 (<2.8) |
| PT/INR | <1.7 | 1.71-2.30 | >2.30 |
| Ascites | None | Mild | Moderate to Severe |
| Hepatic encephalopathy | None | Grade I-II (or suppressed with medication) | Grade III-IV<br>(or refractory) |

| Points | Class |
|--------|-------|
| 5-6 | A |
| 7-9 | В |
| 10-15 | С |

#### Appendix F. Lee cGVHD Symptom Scale

| Identification (Name): | Date: |
|------------------------|-------|
|------------------------|-------|

#### chronic GVHD Symptom Scale

By circling one (1) number per line, please indicate how much you have been bothered by the following problems in the past month:

| SKIN: | | Not at all | Slightly | Moderately | Quite a<br>bit | Extremely |
|---|---|---|---|---|---|---|
| 1. | Abnormal skin color | 0 | 1 | 2 | 3 | 4 |
| 2. | Rashes | 0 | 1 | 2 | 3 | 4 |
| 3. | Thickened skin | 0 | 1 | 2 | 3 | 4 |
| 4. | Sores on skin | 0 | 1 | 2 | 3 | 4 |
| 5. | Itchy skin | 0 | 1 | 2 | 3 | 4 |
| EYES | AND MOUTH: | Not at all | Slightly | Moderately | Quite a bit | Extremely |
| 6. | Dry eyes | 0 | 1 | 2 | 3 | 4 |
| 7. | Need to use eye drops frequently | 0 | 1 | 2 | 3 | 4 |
| 8. | Difficulty seeing clearly | 0 | 1 | 2 | 3 | 4 |
| 9. | Need to avoid certain foods due to mouth pain | 0 | 1 | 2 | 3 | 4 |
| 10. | Ulcers in mouth | 0 | 1 | 2 | 3 | 4 |
| 11. | Receiving nutrition from an intravenous line or feeding tube | 0 | 1 | 2 | 3 | 4 |
| BREA | THING: | Not at all | Slightly | Moderately | Quite a<br>bit | Extremely |
| 12. | Frequent cough | 0 | 1 | 2 | 3 | 4 |
| 13. | Colored sputum. | 0 | 1 | 2 | 3 | 4 |
| 14. | Shortness of breath with exercise | 0 | 1 | 2 | 3 | 4 |
| 15. | Shortness of breath at rest | 0 | 1 | 2 | 3 | 4 |
| 16. | Need to use oxygen | 0 | 1 | 2 | 3 | 4 |

| EATI | NG AND DIGESTION: | Not at all | Slightly | Moderately | Quite a<br>bit | Extremely |
|---|---|---|---|---|---|---|
| 17. | Difficulty swallowing solid foods | 0 | 1 | 2 | 3 | 4 |
| 18. | Difficulty swallowing liquids | 0 | 1 | 2 | 3 | 4 |
| 19. | Vomiting | 0 | 1 | 2 | 3 | 4 |
| 20. | Weight loss | 0 | 1 | 2 | 3 | 4 |
| MUSO | CLES AND JOINTS: | Not at all | Slightly | Moderately | Quite a<br>bit | Extremely |
| 21. | Joint and muscle aches | 0 | 1 | 2 | 3 | 4 |
| 22. | Limited joint movement | 0 | 1 | 2 | 3 | 4 |
| 23. | Muscle cramps | 0 | 1 | 2 | 3 | 4 |
| 24. | Weak muscles | 0 | 1 | 2 | 3 | 4 |
| Energ | y: | Not at all | Slightly | Moderately | Quite a<br>bit | Extremely |
| 25. | Loss of energy | 0 | 1 | 2 | 3 | 4 |
| 26. | Need to sleep more/take naps | 0 | 1 | 2 | 3 | 4 |
| 27. | Fevers | 0 | 1 | 2 | 3 | 4 |
| MEN' | TAL AND EMOTIONAL: | Not at all | Slightly | Moderately | Quite a<br>bit | Extremely |
| 28. | Depression | 0 | 1 | 2 | 3 | 4 |
| 29. | Anxiety | 0 | 1 | 2 | 3 | 4 |
| 30. | Difficulty sleeping | 0 | 1 | 2 | 3 | 4 |

#### Source:

 $http://www.uniklinikum-regensburg.de/imperia/md/content/kliniken-institute/haematologie-onkologie/gvhd/deutsch/lee-symptom\_scale.pdf$ 

#### Appendix G. SF-36 Questionnaire

#### Your Health and Well-Being

This survey asks for your views about your health. This information will help keep track of how you feel and how well you are able to do your usual activities. Thank you for completing this survey!

For each of the following questions, please mark an  $\boxtimes$  in the one box that best describes your answer.

1. In general, would you say your health is:

| Excellent | Very good | Good | Fair | Poor |
|-----------|-----------|------|------|------|
| • | | | | |
| 1 | 2 | 3 | 4 | 5 |

2. <u>Compared to one year ago</u>, how would you rate your health in general now?

| Much better<br>now than one<br>year ago | Somewhat<br>better<br>now than one | About the same as one year ago | Somewhat<br>worse<br>now than one | Much worse<br>now than one<br>year ago |
|---|---|---|---|---|
| | year ago | _ | year ago | _ |
| _ | _ | _ | _ | _ |
| 1 | 2 | 3 | 4 | 5 |

SF-36v2\* Health Survey © 1992, 1996, 2000 Medical Outcomes Trust and QualityMetric Incorporated. All rights reserved. SF-36\* is a registered trademark of Medical Outcomes Trust. (SF-36v2\* Health Survey Standard, United States (English)) 3. The following questions are about activities you might do during a typical day. Does your health now limit you in these activities? If so, how much?

| | | Yes,<br>limited<br>a lot | Yes,<br>limited<br>a little | No, not<br>limited<br>at all |
|---|---|---|---|---|
| a | Vigorous activities, such as running, lifting heavy objects, participating in strenuous sports | | 2 | 3 |
| ь | Moderate activities, such as moving a table, pushing a vacuum cleaner, bowling, or playing golf | | 2 | 3 |
| c | Lifting or carrying groceries | 🗌 1 | 2 | 3 |
| d | Climbing several flights of stairs | 1 | 2 | 3 |
| e | Climbing one flight of stairs | 1 | 2 | 3 |
| ſ | Bending, kneeling, or stooping | 🗆 1 | 2 | 3 |
| 8 | Walking more than a mile | 🗆 1 | 2 | 3 |
| h | Walking several hundred yards | 🔲 1 | 2 | 3 |
| i | Walking one hundred yards | 🔲 1 | 2 | 3 |
| | Bathing or dressing yourself | | | |

SF-36v2<sup>®</sup> Health Survey © 1992, 1996, 2000 Medical Outcomes Trust and QualityMetric Incorporated. All rights reserved. SF-36<sup>®</sup> is a registered trademark of Medical Outcomes Trust. (SF-36v2<sup>®</sup> Health Survey Standard, United States (English))

| 4. | During the past 4 weeks, how much of the time have you had any of the |
|---|---|
| | following problems with your work or other regular daily activities as a |
| | result of your physical health? |

| | | All of<br>the time | Most of<br>the time | Some of<br>the time | A little of<br>the time | None of<br>the time |
|---|---|---|---|---|---|---|
| | · | | | | | |
| а | Cut down on the amount of time you spent on work or other activities | 1 | 2 | 3 | 4 | 5 |
| ь | Accomplished less than you would like | 1 | 2 | 3 | 4 | s |
| c | Were limited in the <u>kind</u> of work or other activities | 1 | 2 | 3 | 4 | s |
| d | Had <u>difficulty</u> performing the<br>work or other activities (for<br>example, it took extra effort) | 1 | 2 | 3 | 4 | 5 |
| | During the past 4 weeks, l | ow much | of the time | have you | had any of | the |

5. During the <u>past 4 weeks</u>, how much of the time have you had any of the following problems with your work or other regular daily activities <u>as a result of any emotional problems</u> (such as feeling depressed or anxious)?

| | | All of<br>the time | Most of<br>the time | Some of the time | A little of<br>the time | None of<br>the time |
|---|---|---|---|---|---|---|
| | · | | | | | |
| | Cut down on the <u>amount of</u><br>time you spent on work or<br>other activities | 1 | 2 | 3 | 4 | 5 |
| , | Accomplished less than you would like | 1 | 2 | 3 | 4 | 5 |
| = | Did work or other activities<br>less carefully than usual | 1 | 2 | 3 | 4 | 5 |

 $SF-36v2^B$  Health Survey  $\otimes$  1992, 1996, 2000 Medical Outcomes Trust and QualityMetric Incorporated. All rights reserved.  $SF-36^B$  is a registered trademark of Medical Outcomes Trust. ( $SF-36v2^B$  Health Survey Standard, United States (English))

6. During the <u>past 4 weeks</u>, to what extent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups?



7. How much bodily pain have you had during the past 4 weeks?



8. During the <u>past 4 weeks</u>, how much did <u>pain</u> interfere with your normal work (including both work outside the home and housework)?

| Not a | nt all A | little bit | Moderately | Quite a bit | Extremely |
|-------|----------|------------|------------|-------------|-----------|
| • | 7 | | | | |
| | 1 | 2 | 3 | 4 | 5 |

SF-36v2<sup>®</sup> Health Survey © 1992, 1996, 2000 Medical Outcomes Trust and QualityMetric Incorporated. All rights reserved. SF-36<sup>®</sup> is a registered trademark of Medical Outcomes Trust. (SF-36v2<sup>®</sup> Health Survey Standard, United States (English))

These questions are about how you feel and how things have been with you
during the past 4 weeks. For each question, please give the one answer that
comes closest to the way you have been feeling. How much of the time
during the past 4 weeks...

| | _ | | | | | |
|---|---|---|---|---|---|---|
| | | All of<br>the time | Most of<br>the time | Some of the time | A little of the time | None of<br>the time |
| , D | oid you feel full of life? | 1 | 2 | 3 | 4 | 5 |
| ь Н | ave you been very nervous? | 1 | 2 | 3 | | 5 |
| dı | ave you felt so down in the umps that nothing could neer you up? | 1 | 2 | 3 | 4 | 5 |
| d Н | ave you felt calm and<br>eaceful? | | 2 | 3 | 4 | 5 |
| e D | old you have a lot of energy? | 1 | 2 | 3 | 4 | 5 |
| r H | ave you felt downhearted<br>and depressed? | 1 | 2 | 3 | 4 | 5 |
| 8 D | oid you feel worn out? | П 1 | 2 | 3 | 4 | 5 |
| ь Н | ave you been happy? | 1 | 2 | 3 | 4 | 5 |
| , D | id you feel tired? | 1 | 2 | 3 | 4 | 5 |
| <u>e1</u> | uring the <u>past 4 weeks,</u> l<br><u>motional problems</u> interf<br>iends, relatives, etc.)? | | | | | |
| | All of Most of<br>the time the time | | | little of<br>he time | None of<br>the time | |
| | <b>V</b> | _ | 7 | | _ | I |
| | 1 2 | | 3 | 4 | 5 | |

SF-36v2\* Health Survey © 1992, 1996, 2000 Medical Outcomes Trust and QualityMetric Incorporated. All rights reserved. SF-36\* is a registered trademark of Medical Outcomes Trust. (SF-36v2\* Health Survey Standard, United States (English))

#### 11. How TRUE or FALSE is each of the following statements for you?

| | | Definitely<br>true | Mostly<br>true | Don't<br>know | Mostly<br>false | Definitely<br>false |
|---|---|---|---|---|---|---|
| a | I seem to get sick a little easier than other people | 1 | 2 | 3 | | 5 |
| b | I am as healthy as<br>anybody I know | 🔲 1 | 2 | 3 | 4 | 5 |
| c | I expect my health to get worse | 🔲 1 | 2 | 3 | 4 | 5 |
| d | My health is excellent | 1 | 2 | 3 | | 5 |

Thank you for completing these questions!

SF-36v2® Health Survey © 1992, 1996, 2000 Medical Outcomes Trust and QualityMetric Incorporated. All rights reserved. SF-36® is a registered trademark of Medical Outcomes Trust. (SF-36v2® Health Survey Standard, United States (English))

# Appendix H. Chronic GVHD Activity Assessment - Clinician

| FORM A Current | Current Patient Weight: | | | 1 | | Today's Date: | 8 | | | MR#/Name: | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 93 | | CHI | SONIC | GVHI | ACTIV | TTY ASSES | SME | RONIC GVHD ACTIVITY ASSESSMENT- CLINICIAN | | | | |
| Health Care Provider<br>Global Ratings: | Where w following most sev | Where would you rate the severity of this patient's chronic GvHD symptoms on the following scale, where 0 is cGVHD symptoms that are not at all severe and 10 is the most severe cGVHD symptoms possible: | cGVHD syoms poss | f this pa<br>ymptom<br>ible: | tient's chr<br>s that are | everity of this patient's chronic GvHD symptoms on the cGVHD symptoms that are not at all severe and 10 is the oms possible: | ptoms of and 10 | h 828 | <time>&gt; w&lt;</time> | Over the < <ti>cGvHD is<br/>cGvHD is<br/>+3= Very much better</ti> | his patient' | S |
| 0=none<br>1= mild<br>2=moderate | cGvHD sympton | CGVHD symptoms | 4 | 5 | 2 9 | 8 9 Most s | 9 10<br>Most severe cGvHD | | ately better<br>better<br>he same | | | |
| 3=severe | | | | | | and the second | | -1=A little worse<br>-2=Moderately worse<br>-3=Very much worse | orse<br>ely worse<br>ich worse | | | 10 |
| Mouth | | Erythema | None | 0 | Mild en<br>modera | Mild erythema or moderate erythema | - | Moderate (≥25%) or Severe erythema | or 2 | Severe erythema<br>(≥25%) | еша | 3 |
| | | Lichenoid | None | 0 | Lichen-I | Lichen-like changes<br>(<25%) | - | Lichen-like changes (25-50%) | s 5 | Lichen-like changes (>50%) | anges | 3 |
| | | Ulcers | None | 0 | | | | Ulcers involving (<20%) | 3 | Severe ulcerations (>20%) | tions | 9 |
| | | | | | | | | | Total score | Total score for all mucosal changes | hanges | |
| Gastrointestinal-Esophageal • Dysphagia OR Odynophagia | ageal | 0= no esophageal symptoms<br>1=Occasional dysphagia or odynophagia with solid food or pills <u>during the past week</u><br>2=Intermittent dysphagia or odynophagia with solid foods or pills, but not for liquids o<br>3=Dysphagia or odynophagia for almost all oral intake, <u>on almost every day of the p</u> e | symptoms<br>chagia or o<br>phagia or o<br>dynophagia | s<br>odynoph<br>odynoph<br>a for alm | agia with s<br>agia with s<br>ost all oral | olid food or pills o<br>olid foods or pills<br>intake, <u>on almos</u> | during the<br>s, but not<br>st every o | 0= no esophageal symptoms<br>1=Occasional dysphagia or odynophagia with solid food or pills <u>during the past week</u><br>2=Intermittent dysphagia or odynophagia with solid foods or pills, but not for liquids or soft foods, <u>during the past week</u><br>3=Dysphagia or odynophagia for almost all oral intake, <u>on almost every day of the past week</u> | ds, <u>during</u> t | he past week | | 7 |
| Gastrointestinal-Upper GI Early satiety OR Anorexia OR Nausea & Vomiting | ច | 0= no symptoms<br>1=mild, occasional symptoms, with little reduction in oral intake <u>during the past week</u><br>2=moderate, intermittent symptoms, with some reduction in oral intake <u>during the pa</u><br>3=more severe or persistent symptoms throughout the day, with marked reduction in | l symptom<br>nittent syn<br>persistent | s, with lings<br>optoms,<br>symptor. | ttle reduction with some ms through | on in oral intake or<br>reduction in oral<br>out the day, with | during th<br>intake d<br>marked | 0= no symptoms<br>1=mild, occasional symptoms, with little reduction in oral intake <u>during the past week</u><br>2=moderate, intermittent symptoms, with some reduction in oral intake <u>during the past week</u><br>3=more severe or persistent symptoms throughout the day, with marked reduction in oral intake, <u>on almost every day of the past week</u> | ke, <u>on almo</u> | st every day of the L | oast week | |
| Gastrointestinal-Lower Gl Diarrhea | ច | 0= no loose or liquid stools <u>during the past week</u> 1= occasional loose or liquid stools, on some days <u>during the past week</u> 2=intermittent loose or liquid stools throughout the day, <u>on almost every</u> correct volume depletion 3=voluminous diarrhea on almost every day of the past week, <b>requiring</b> | iid stools case or liquid se or liquid oletion | uring the<br>stools, c<br>stools th | e past weel<br>on some de<br>nroughout t | k<br>yys <u>during the pa</u><br>he day, <u>on almo</u><br>he past week. <b>re</b> | st week | 0= no loose or liquid stools <u>during the past week</u> 1= occasional loose or liquid stools, on some days <u>during the past week</u> 2=intermittent loose or liquid stools throughout the day, <u>on almost every day of the past week, without requiring</u> intervention to prevent or correct volume depletion 3=voluminous diarrhea on almost every day of the past week, requiring intervention to prevent or correct volume depletion | without re | quiring intervention | ı to prevent | or |
| Lungs (Liters and % predicted) Bronchiolitis Obliterans | edicted) | FEV1 | | FVC | 77 | Single Breath DLCO (adjusted for hemoglobin) | CO (ad | justed for | TLC | | RV | 0 |
| Liver Values | | Total serum bilirubin mg/dL | | NTN | mg/dL | ALT U/L | | ULN | Alkaline | Alkaline Phosphatase<br>U/L | NTN | U/L |
| Baseline Values | | | | | | Karnofsky or<br>Lansky | <u>a</u> | Platelet Count<br>K/uL | Total WBC | SC<br>K/uL | Eosinophils | ls<br>% |
| | | ☐ Abnormality pre: ☐ Abnormality pre: ☐ Abnormality pre: ☐ Abnormality pres | sent but ex<br>sent but ex<br>sent but ex | plained<br>plained<br>plained | entirely by<br>entirely by<br>entirely by | non-GVHD docu<br>non-GVHD docu<br>non-GVHD docu | mented<br>mented<br>mented | <ul> <li>□ Abnormality present but explained entirely by non-GVHD documented cause (specify site/alternate cause):</li> <li>□ Abnormality present but explained entirely by non-GVHD documented cause (specify site/alternate cause):</li> <li>□ Abnormality present but explained entirely by non-GVHD documented cause (specify site/alternate cause):</li> </ul> | temate cau<br>temate cau<br>temate cau | se): | 111 | |

#### CHRONIC GVHD ACTIVITY ASSESSMENT- CLINICIAN (FORM A)

| | SCORE 0 | SCORE 1 | SCORE 2 | SCORE 3 |
|---|---|---|---|---|
| | SCORE | SCORE 1 | SCORE 2 | SCORE 3 |
| SKIN | □ No BSA involved | ☐ 1-18% BSA | ☐ 19-50% BSA | □ >50% BSA |
| GVHD features to be scored by BSA: Check all that apply: Maculopapular rash/erythema Lichen planus-like features Sclerotic features Papulosquamous lesions or ichthyosis Keratosis pilaris-like | | | | |
| ☐ Abnormality present b<br>(specify): | out explained entirely | y by non-GVHD doc | umented cause | |
| SKIN FEATURES<br>SCORE | ☐ No sclerotic features | | ☐ Superficial sclerotic features "not hidebound" (able to pinch) | Check all that apply: Deep sclerotic features "Hidebound" (unable to pinch) Impaired mobility Ulceration |
| is not at all severe ar | the severity of this | patient's skin and/or<br>vere symptoms possib | joint tightening on the fo | |
| EYES | □ No symptoms | ☐ Mild dry eye symptoms not affecting ADL (requirement of lubricant eye drops ≤3 x per day) | ☐ Moderate dry eye symptoms partially affecting ADL (requiring lubricant eye drops >3 x per day or punctal plugs), WITHOUT new vision impairment due to KCS | ☐ Severe dry eye symptoms significantly affecting ADL (special eyewear to relieve pain) OR unable to work because of ocular symptoms OR loss of vision due to KCS |
| ☐ Abnormality present b (specify): | out explained entirely | y by non-GVHD doc | umented cause | |

| | SCORE 0 | SCORE 1 | SCORE 2 | SCORE 3 |
|---|---|---|---|---|
| LUNGS | No symptoms | Mild<br>symptoms<br>(shortness of<br>breath after<br>climbing one<br>flight of steps) | Moderate<br>symptoms<br>(shortness of<br>breath after<br>walking on flat<br>ground) | Severe symptoms (shortness of breath at rest; requiring $0_2$ ) |
| Abnormality present b (specify): | ut explained entirely | y by non-GVHD doc | umented cause | |
| JOINTS AND<br>FASCIA | No symptoms | Mild tightness<br>of arms or<br>legs, normal or<br>mild decreased<br>range of<br>motion (ROM)<br>AND not<br>affecting ADL | Tightness of arms or legs OR joint contractures, erythema thought due to fasciitis, moderate decrease ROM AND mild to moderate limitation of ADL | Contractures WITH significant decrease of ROM AND significant limitation of ADL (unable to tie shoes, button shirts, dress self, etc.) |
| Abnormality present b (specify): | ut explained entirely | y by non-GVHD doc | umented cause | |



#### ☐ Abnormality present but explained entirely by non-GVHD documented cause (specify):

#### Reference:

Lee SJ, Wolff D, Kitko C, et al. Measuring Therapeutic Response in Chronic Graft-versus-Host Disease. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: IV. The 2014 Response CriteriaWorking Group Report. Biol Blood Marrow Transplant. 2015;21:984-999.

FINAL

Appendix I. Response Determination for Chronic GVHD Clinical Trials based on Clinician Assessments

| Organ | Complete Response | Partial Response | Progression |
|---|---|---|---|
| Skin | NIH Skin Score 0 after | Decrease in NIH Skin Score | Increase in NIH Skin Score by 1 or |
| | previous involvement | by 1 or more points | more points, except 0 to 1 |
| Eyes | NIH Eye Score 0 after | Decrease in NIH Eye Score | Increase in NIH Eye Score by 1 or |
| | previous involvement | by 1 or more points | more points, except 0 to 1 |
| Mouth | NIH Modified OMRS 0 after | Decrease in NIH Modified OMRS | Increase in NIH Modified OMRS |
| | previous involvement | of 2 or more points | of 2 or more points |
| Esophagus | NIH Esophagus Score 0 after | Decrease in NIH Esophagus | Increase in NIH Esophagus Score |
| | previous involvement | Score by 1 or more points | by 1 or more points, except 0 to 1 |
| Upper GI | NIH Upper GI Score 0 after | Decrease in NIH Upper GI | Increase in NIH Upper GI Score |
| | previous involvement | Score by 1 or more points | by 1 or more points, except 0 to 1 |
| Lower GI | NIH Lower GI Score 0 after | Decrease in NIH Lower GI | Increase in NIH Lower GI Score by 1 |
| | previous involvement | Score by 1 or more points | or more points, except from 0 to 1 |
| Liver | Normal ALT, alkaline | Decrease by 50% | Increase by $2 \times ULN$ |
| | phosphatase, and Total | | |
| | bilirubin after previous | | |
| | elevation of 1 or more | | |
| Lungs | - Normal %FEV1 after | <ul> <li>Increase by 10% predicted</li> </ul> | <ul> <li>Decrease by 10% predicted</li> </ul> |
| | previous involvement | absolute value of %FEV1 | absolute value of %FEV1 |
| | <ul> <li>If PFTs not available, NIH</li> </ul> | <ul> <li>If PFTs not available, decrease</li> </ul> | <ul> <li>If PFTs not available, increase in</li> </ul> |
| | Lung Symptom Score 0 | in NIH Lung Symptom Score | NIH Lung Symptom Score by 1 |
| | after previous involvement | by 1 or more points | or more points, except 0 to 1 |
| Joints and fascia | Both NIH Joint and Fascia | Decrease in NIH Joint and Fascia | Increase in NIH Joint and Fascia |
| | Score 0 and P-ROM score | Score by 1 or more points or | Score by 1 or more points or |
| | 25 after previous involvement | increase in P-ROM score by 1 | decrease in P-ROM score by 1 |
| | by at least 1 measure | point for any site | point for any site |
| Global | Clinician overall severity score 0 | Clinician overall severity score | Clinician overall severity score |
| | | decreases by 2 or more points | increases by 2 or more points |
| | | on a 0-10 scale | on a 0-10 scale |
| I manage by timil again actually in IVIII | - constant | | |

ULN indicates upper limit of normal.

## Overall Response:

Skin, mouth, liver, upper and lower GI, esophagus, lung, eye, and joint/fascia are the organs or sites considered in evaluating overall

- Complete Response (CR) is defined as resolution of all manifestations in each organ or site
- Partial Response (PR) is defined as improvement in at least 1 organ or site without progression in any other organ or site.
- Disease Progression is defined as clinically meaningful worsening in one or more organs regardless of improvement in other organs. Mixed Response: CR or PR in at least 1 organ accompanied by progression in another organ is considered disease progression.
- Stable disease (SD): response that does not meet the criteria for CR, PR, or disease progression.

assessments coinciding with chronic GVHD flares (transient worsening of organs that were previously involved) will be inevaluable progression will be calculated using first date of disease progression. Lack of Response includes categories of disease progression or If a patient shows overall cGVHD improvement while organ responses indicate progression in one or more organs, cGVHD and should be repeated as soon as the flare resolves or at the next assessment time point. If progression is confirmed, time to assessment should be repeated at a different time point, to confirm progression, before discontinuing study drug. Response stable disease. Lee SJ, Wolff D, Kitko C, et al. Measuring Therapeutic Response in Chronic Graft-versus-Host Disease. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: IV. The 2014 Response Criteria Working Group Report. Biol Blood Marrow Transplant. 2015;21:984-999.

#### Appendix J. Chronic GVHD Activity Assessment – Patient Self Report

| FORM B Today's Date: MR#/Name: |
|--------------------------------|
|--------------------------------|

#### CHRONIC GVHD ACTIVITY ASSESSMENT-PATIENT SELF REPORT

| Please rate how severe the following symptoms have been in the <u>last seven days</u> . Please fill in the circle below from 0 (symptom has not been present) to 10 (the | | | Not<br>You<br>Present<br>Imagine | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| symptom was as bad as imagine it could be) for e | 0<br>10 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | | |
| Your <b>skin itching</b> at its W | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | |
| Your <b>skin and/or joint tightening</b> at their WORST? | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Your mouth sensitivity at its WORST? | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Your <b>genital discomfort</b> at its WORST? (Women – vagina, vulva, or labia) (Men – penis) | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Eyes | What is your i | | | | ur main complaint with regard to your eyes? | | | | | | | |
| | thow severe this symptom is, from 0 (not e) to 10 (most severe): 0 1 2 3 4 5 6 7 8 10 10 (most severe): | | | | | | | | 8 9 | | | |

| Patient Global Ratings: | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| 1. Overall, do you think that your chronic graft versus host disease is mild, moderate or severe? 1= mild 2=moderate 3=severe | | | | | | | | | | |
| | | | | | | | | | | host disease symptoms are, where 0 is c GvHD symptoms possible. |
| 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| cGvHD sym<br>not at all se | | | | | | | | | | Most severe cGvHD symptoms possible |
| 3. Compared to a month ago, overall would you say that your cGvHD symptoms are: | | | | | | | | | | |
| +3= Very much better +2= Moderately better +1=A little better 0= About the same | | | | | | | | | | |

#### Reference:

-1=A little worse -2=Moderately worse -3=Very much worse

Lee SJ, Wolff D, Kitko C, et al. Measuring Therapeutic Response in Chronic Graft-versus-Host Disease. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: IV. The 2014 Response Criteria Working Group Report. Biol Blood Marrow Transplant. 2015;21:984-999.

#### Appendix K. Prednisone Equivalents Table

Corticosteroid Doses Equivalent to 20 mg Prednisone

| Corticosteroid | Equivalent dose (mg) |
|--------------------|----------------------|
| Prednisone | 20 |
| Cortisone | 100 |
| Cortisol | 80 |
| Hydrocortisone | 80 |
| Prednisolone | 20 |
| Methylprednisolone | 16 |
| Triamcinolone | 16 |
| Betamethasone | 3 |
| Dexamethasone | 3 |

#### Source:

Brunton LL, Chabner BA, Knollmann BC (Eds). The Pharmacological Basis of Therapeutics, 12<sup>th</sup> ed. McGraw Hill, New York 2011. p.1216.

Appendix L. Summary of Ancillary Therapy and Supportive Care Interventions

| Organ System | Organ-Specific Intervention* | |
|---|---|---|
| | Prevention | Treatment |
| Skin and appendages | Photoprotection -sun avoidance and physical sunblocks (eg, protective clothing, UVA, and UVB sunscreens). Avoidance of photosensitizing agents (eg, voriconazole). Surveillance for malignancy [Inamoto 2015, Majhail 2012]. | For intact skin topical emollients including urea containing products, corticosteroids, antipruritic agents, and others (eg, PUVA or narrow band UVB, calcineurin inhibitors). For erosions/ulcerations e microbiologic cultures, topical antimicrobials, protective films or other dressings, debridement, hyperbaric oxygen, wound care specialist consultation. |
| Mouth and oral cavity | Maintain good oral/dental hygiene.<br>Routine dental cleaning and<br>radiographs. Surveillance for<br>infection and malignancy.<br>Nutritional counseling, if needed. | Topical high and ultra-high potency corticosteroids and topical calcineurin inhibitors. Topical analgesics. Therapy for oral dryness (eg, salivary stimulants, sialogogues) and for prevention of related complications (ie, dental decay). |
| Eyes | Photoprotection. Surveillance for infection, cataract formation, and increased intraocular pressure. | Artificial tears, ocular ointments, topical corticosteroids or cyclosporine, punctal occlusion, humidified environment, occlusive eye wear, moisture chamber eyeglasses, cevimeline, pilocarpine, gas-permeable scleral contact lens, autologous serum, microbiologic cultures, topical antimicrobials, doxycycline. |
| Vulva and vagina | Surveillance for estrogen deficiency, infection (HSV, HPV, yeast, bacteria) and malignancy [Majhail 2012]. | Water-based or silicone lubricants, topical estrogens, topical corticosteroids or calcineurin inhibitors, dilators or vibrators, surgery for extensive synechiae or obliteration, early gynecology consultation. Avoid glycerin, paraben, fragrance, and other additive products. |
| Gastrointestinal tract and liver | Surveillance for infection (viral, bacterial, fungal, parasites) | Rule out other potential etiologies. Dietary modification, enzyme supplementation for pancreatic insufficiency, bile salt resins, gastroesophageal reflux management, esophageal dilatation, ursodeoxycholic acid, topical glucocorticoids, limitation of ethanol intake, avoidance of hepatotoxins. |

| Organ System | Organ-Specific Intervention* | |
|---|---|---|
| | Prevention | Treatment |
| Lungs | Surveillance for infection<br>(Pneumocystis jiroveci, viral,<br>fungal, bacterial). | Rule out other potential etiologies (eg, infection, gastroesophageal reflux). Inhaled corticosteroids, bronchodilators, supplementary oxygen, pulmonary rehabilitation. Consideration of lung transplantation in appropriate candidates. |
| Hematopoietic | Surveillance for infection (CMV, parvovirus) | Rule out other potential etiologies (eg, drug toxicity, infection). Hematopoietic growth factors, immunoglobulin for immune cytopenias |
| Neurologic | Calcineurin drug level monitoring. Seizure prophylaxis as indicated, including blood pressure control, electrolyte replacement, anticonvulsants. EMG monitoring and staging in symptomatic patients taking medications known to cause neuropathy. Close monitoring of distal extremities for wounds in insensate patients. | Occupational and physical therapy to prevent falls and improve function, treatment of neuropathic syndromes with tricyclic antidepressants, SSRI, or anticonvulsants [Smith 2013]. Orthotics and assistive devices (canes and walkers). Bracing, splinting or surgical release for entrapment neuropathies. |
| Immunologic and infectious diseases | Immunizations and prophylaxis against Pneumocystis jirovecii, VZV, and encapsulated bacteria based on CDC guidelines. Consider immunoglobulin replacement based on levels and recurrent infections. Surveillance for infection (viral, bacterial, fungal, atypical). | Organism-specific antimicrobial agents. Empiric parenteral broadspectrum antibacterial coverage for fever. |
| Musculoskeletal | Surveillance for decreased ROM, bone densitometry, calcium levels and 25-OH vitamin D. Physical therapy, calcium, vitamin D, and bisphosphonates. Flexion-extension x-rays to look for instability. | Physical therapy, bisphosphonates for osteopenia, and osteoporosis. Spinal orthosis for instability and/or intractable pain. Walking program, resistance training, core strengthening. |

SSRI indicates selective serotonin reuptake inhibitors; CDC, Centers for Disease Control.

Carpenter PA, Kitko CL, Elad S. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: V. The 2014 Ancillary Therapy and Supportive Care Working Group Report. Biol Blood Marrow Transplant. 2015;21:1167–87.

<sup>\*</sup>In general, close serial monitoring of all organ systems is recommended to promote early detection and intervention directed toward reversing or preventing progression of chronic GVHD manifestations and treatment-associated toxicities. Ancillary and supportive care therapies are commonly employed in addition to systemic GVHD treatment, although in some cases their use may circumvent the need for systemic treatment or allow doses of systemic agents to be reduced.
Inamoto Y, Savani BN, Shaw BE, et al. Secondary solid cancer screening following hematopoietic cell transplantation. Bone Marrow Transplant. 2015. [Epub ahead of print].

Majhail NS, Rizzo JD, Lee SJ, et al. Recommended screening and preventive practices for long-term survivors after hematopoietic cell transplantation. Biol Blood Marrow Transplant. 2012;18:348–71.

Smith EM, Pang H, Cirrincione C, et al. Effect of duloxetine on pain, function, and quality of life among patients with chemotherapy-induced painful peripheral neuropathy: a randomized clinical trial. JAMA. 2013;309:1359–67.

IMBRUVICA® (ibrutinib)

Appendix M. Diagnosis of cGVHD - Signs and Symptoms of cGVHD

06 February 2019 FINAL

| ORGAN OR SITE | DIAGNOSTIC (Sufficient to establish the diagnosis of chronic GVHD) | DISTINCTIVE <sup>a</sup> (Seen in chronic GVHD, but insufficient alone to establish a diagnosis) | OTHER FEATURES OR<br>UNCLASSIFIED<br>ENTITIES <sup>b</sup> | COMMON° (Seen with both acute and chronic GVHD) |
|---|---|---|---|---|
| Skin | <ul> <li>Poikiloderma</li> <li>Lichen planus-like features</li> <li>Sclerotic features</li> <li>Morphea-like features</li> <li>Lichen sclerosus-like features</li> </ul> | Depigmentation Papulosquamous lesions | <ul> <li>Sweat impairment</li> <li>Ichthyosis</li> <li>Keratosis pilaris</li> <li>Hypopigmentation</li> <li>Hyperpigmentation</li> </ul> | <ul><li>Erythema</li><li>Maculopapular rash</li><li>Pruritus</li></ul> |
| Nails | | <ul> <li>Dystrophy <ul> <li>Longitudinal ridging,</li> <li>splitting or brittle features</li> </ul> </li> <li>Onycholysis</li> <li>Pterygium unguis</li> <li>Nail loss (usually symmetric, affects most nails)</li> </ul> | | |
| Scalp and body hair | | <ul> <li>New onset of scarring or nonscarring scalp alopecia (after recovery from chemoradiotherapy)</li> <li>Loss of body hair</li> <li>Scaling</li> </ul> | <ul> <li>Thinning scalp hair, typically patchy, coarse or dull (not explained by endocrine or other causes)</li> <li>Premature gray hair</li> </ul> | |
| Mouth | Lichen planus-like changes | <ul> <li>Xerostomia</li> <li>Mucoceles</li> <li>Mucosal atrophy</li> <li>Ulcers</li> <li>Pseudomembranes</li> </ul> | | <ul><li>Gingivitis</li><li>Mucositis</li><li>Erythema</li><li>Pain</li></ul> |
| Eyes | | <ul> <li>New onset dry, gritty, or painful eyes</li> <li>Cicatricial conjunctivitis</li> <li>Keratoconjunctivitis sicca</li> <li>Confluent areas of punctate keratopathy</li> </ul> | <ul> <li>Photophobia</li> <li>Periorbital <ul> <li>hyperpigmentation</li> </ul> </li> <li>Blepharitis (erythema of the eyelids with edema)</li> </ul> | |

| ORGAN OR SITE | DIAGNOSTIC (Sufficient to establish the diagnosis of chronic GVHD) | DISTINCTIVE <sup>a</sup> (Seen in chronic GVHD, but insufficient alone to establish a diagnosis) | OTHER FEATURES OR<br>UNCLASSIFIED<br>ENTITIES <sup>b</sup> | COMMON° (Seen with both acute and chronic GVHD) |
|---|---|---|---|---|
| Genitalia | <ul><li>Lichen planus-like features</li><li>Lichen sclerosus-like features</li></ul> | <ul><li>Erosions</li><li>Fissures</li></ul> | | |
| Females | <ul> <li>Vaginal scarring or clitoral/labial agglutination</li> <li>Phimosis or urethral/meatus</li> </ul> | • Ulcers | | |
| Muco | scarring or stenosis | | | |
| GI Tract | Esophageal web Strictures or stenosis in the upper to mid third of the esophagus | | Exocrine pancreatic insufficiency | <ul> <li>Anorexia</li> <li>Nausea</li> <li>Vomiting</li> <li>Diarrhea</li> <li>Weight loss</li> <li>Failure to thrive</li> <li>(infants</li> <li>and children</li> <li>Total bilimbin</li> </ul> |
| Liver | | | | I otal blirtubin, alkaline phosphatase >2 x upper limit of normal ALT >2 x upper limit of normal |
| Lung | <ul> <li>Bronchiolitis obliterans<br/>diagnosed with lung biopsy</li> <li>Bronchiolitis obliterans<br/>syndrome (BOS)<sup>d</sup></li> </ul> | Air trapping and bronchiectasis on chest CT | <ul> <li>Cryptogenic organizing pneumonia (COP)<sup>¢</sup></li> <li>Restrictive lung disease<sup>¢</sup></li> </ul> | |

FINAL

06 February 2019

| ORGAN OR SITE | DIAGNOSTIC (Sufficient to establish the diagnosis of chronic GVHD) | DISTINCTIVE <sup>a</sup> (Seen in chronic GVHD, but insufficient alone to establish a diagnosis) | OTHER FEATURES OR<br>UNCLASSIFIED<br>ENTITIES <sup>b</sup> | COMMON° (Seen with both acute and chronic GVHD) |
|---|---|---|---|---|
| Muscles, fascia,<br>joints | <ul> <li>Fasciitis</li> <li>Joint stiffness or contractures secondary to fasciitis or sclerosis</li> </ul> | Myositis or polymyositis <sup>f</sup> | <ul><li>Edema</li><li>Muscle cramps</li><li>Arthralgia or arthritis</li></ul> | |
| Hematopoietic and<br>Immune | | | <ul> <li>Thrombocytopenia</li> <li>Eosinophilia</li> <li>Lymphopenia</li> <li>Hypo- or hypergammaglobulinemia</li> <li>Autoantibodies (AIHA, ITP)</li> <li>Raynaud's phenomenon</li> </ul> | |
| Other | | | <ul> <li>Pericardial or pleural effusions</li> <li>Ascites</li> <li>Peripheral neuropathy</li> <li>Nephrotic syndrome</li> <li>Myasthenia gravis</li> <li>Cardiac conduction abnormality or cardiomyopathy</li> </ul> | |

Abbreviations: ALT indicates alanine aminotransferase; AIHA, autoimmune hemolytic anemia; ITP, idiopathic thrombocytopenic purpura.

Jagasia HM, Greinix HT, Arora M, et al. Biol Blood Marrow Transplant. 2015;21:389-401.

In all cases, infection, drug effect, malignancy, or other causes must be excluded.

Can be acknowledged as part of the chronic GVHD manifestations if diagnosis is confirmed.

Common refers to shared features by both acute and chronic GVHD.

BOS can be diagnostic for lung chronic GVHD only if distinctive sign or symptom present in another organ (see text).

Pulmonary entities under investigation or unclassified. Diagnosis of chronic GVHD requires biopsy.

# Appendix N. Staging of cGVHD

| | SCORE 0 | SCORE 1 | SCORE 2 | SCORE 3 |
|---|---|---|---|---|
| PERFORMANCE<br>SCORE:<br>KPS ECOG LPS | Asymptomatic and<br>fully active (ECOG<br>0; KPS or LPS<br>100%) | Symptomatic,<br>fully ambulatory,<br>restricted only in<br>physically<br>strenuous activity<br>(ECOG 1, KPS<br>or LPS 80-90%) | Symptomatic,<br>ambulatory, capal<br>of self-care, >50%<br>of waking hours of<br>bed (ECOG 2,<br>KPS or LPS 60-<br>70%) | >50% of waking |
| SKIN† SCORE % BSA GVHD features to be scored by BSA: Check all that apply: Maculopapular rash/eryth Lichen planus-like featur Sclerotic features | involved<br>nema<br>es | 1-18% BSA | 19-50% BSA | >50% BSA |
| Papulosquamous lesions<br>ichthyosis<br>Keratosis pilaris-like GV<br>SKIN FEATURES | | | | Check all that apply: |
| SCORE: | No sclerotic features | | Superficial<br>sclerotic features<br>"not hidebound"<br>(able to pinch) | Deep sclerotic features "Hidebound" (unable to pinch) Impaired mobility Ulceration |
| Other skin GVHD features Check all that apply: Hyperpigmentation Hypopigmentation Poikiloderma Severe or generalized pro Hair involvement Nail involvement Abnormality present but of | uritus | on-GVHD documented | cause (specify): | |
| MOUTH Lichen planus-like features present: Yes No Abnormality present but o | No symptoms | Mild symptoms with disease signs but not limiting oral intake significantly on-GVHD documented | disease signs with<br>partial limitation<br>of oral intake | Severe symptoms with<br>disease signs on<br>examination <b>with</b> major<br>limitation of oral intake |

| | SCORE 0 | SCORE 1 | SCORE 2 | SCORE 3 |
|---|---|---|---|---|
| EYES Keratoconjunctivitis sicca (KCS) confirmed by ophthalmologist: Yes No Not examined | No symptoms | Mild dry eye symptoms not affecting ADL (requirement of lubricant eye drops ≤ 3 x per day) | Moderate dry eye symptoms partially affecting ADL (requiring lubricant eye drops > 3 x per day or punctal plugs), WITHOUT new vision impairment due to KCS | Severe dry eye symptoms significantly affecting ADL (special eyeware to relieve pain) OR unable to work because of ocular symptoms OR loss of vision due to KCS |
| | i explained entirely b | y non-GVHD documented | i cause (specify) | |
| GI Tract Check all that apply: Esophageal web/ proximal stricture or ring Dysphagia Anorexia Nausea Vomiting Diarrhea Weight loss ≥5%* Failure to thrive Abnormality present bu | No symptoms t explained entirely b | Symptoms without significant weight loss* (<5%) | Symptoms associated with mild to moderate weight loss* (5-15%) OR moderate diarrhea without significant interference with daily living | Symptoms associated with significant weight loss*>15%, requires nutritional supplement fo most calorie needs <b>OR</b> esophageal dilation <b>OR</b> severe diarrhea with significant interference with daily living |
| | | | | The state of |
| Liver | Normal total<br>bilirubin and<br>ALT or AP<br>< 3 x ULN | Normal total<br>bilirubin with ALT<br>≥3 to 5 x ULN or<br>AP ≥ 3 x ULN | Elevated total<br>bilirubin but<br>≤3 mg/dL or<br>ALT > 5 ULN | Elevated total<br>bilirubin > 3 mg/dL |
| Abnormality present bu | t explained entirely b | y non-GVHD documented | d cause (specify): | |
| Lungs** | | | | |
| Symptom score: | No symptoms | Mild symptoms<br>(shortness of<br>breath after<br>climbing one flight<br>of steps) | Moderate<br>symptoms<br>(shortness of breath<br>after walking on<br>flat ground) | Severe symptoms (shortness of breath at rest; requiring $0_2$ ) |
| Lung score:<br>% FEV1 | FEV1≥80% | FEV1 60-79% | FEV1 40-59% | FEV1 ≤39% |
| Pulmonary function tests Not performed Abnormality present bu | t explained entirely b | y non-GVHD documented | l cause (specify): | |

| 5 | SCORE 0 | SCORE 1 | SCORE 2 | SCORE 3 |
|---|---|---|---|---|
| P-ROM score (see below) Shoulder (1-7): Elbow (1-7): Wrist/finger (1-7): Ankle (1-4): Abnormality present but | No symptoms | Mild tightness of arms or legs, normal or mild decreased range of motion (ROM) AND not affecting ADL | Tightness of arms or legs <b>OR</b> joint contractures, erythema thought due to fasciitis, moderate decrease ROM <b>AND</b> mild to moderate limitation of ADL ented cause (specify): | Contractures WITH significant decrease of ROM AND significant limitation of ADL (unable to tie shoes, button shirts, dress self etc.) |
| GENITAL TRACT (See Supplemental figure*) Not examined Currently sexually active Yes No | No signs | Mild signs <sup>‡</sup> and<br>females with or<br>without discomfort<br>on exam | Moderate signs <sup>‡</sup> and may have symptoms with discomfort on exam | Severe signs <sup>‡</sup> with<br>or without<br>symptoms |
| Abnormality present but explained entirely by non-GVHD documented cause (specify): Other indicators, clinical features or complications related to chronic GVHD (check all that apply and assign a | | | | |
| | | | ronic GVHD (check all the ble none – 0,mild -1, mod | |
| Ascites (serositis) | | henia Gravis | bie none – o,mila -1, moa | <u> </u> |
| Pericardial Effusion | | neral Neuropathy | Eosinop | bhilia > 500/μl |
| Pleural Effusion(s) | _ | nyositis | | s <100,000/µl |
| Nephrotic syndrome Weight loss>5%* without GI symptoms Others (specify): | | | | |
| Overall GVHD Severity<br>(Opinion of the evaluator) | □ No GV | THD Mild | ☐ Moderate | ☐ Severe |
| Photographic Range of Motion (P-ROM) | | | | |
| | Shoulder 1 Wer | 2 3 4 5 | 6 7(Normal) | |
| | Elbow | | 6 Tillowsh | |
| | Wrist/finger | | (rooma) | |
| | Ankle | Z 3 4(Normal) | | |

- † Skin scoring should use both percentage of BSA involved by disease signs and the cutaneous features scales. When a discrepancy exists between the percentage of total body surface (BSA) score and the skin feature score, OR if superficial sclerotic features are present (Score 2), but there is impaired mobility or ulceration (Score 3), the higher level should be used for the final skin scoring.
- \* Weight loss within 3 months.
- \*\*Lung scoring should be performed using both the symptoms and FEV1 scores whenever possible. FEV1 should be used in the final lung scoring where there is discrepancy between symptoms and FEV1 scores.

Abbreviations: ECOG (Eastern Cooperative Oncology Group), KPS (Karnofsky Performance Status), LPS (Lansky Performance Status); BSA (body surface area); ADL (activities of daily living); LFTs (liver function tests); AP (alkaline phosphatase); ALT (alanine aminotransferase); ULN (normal upper limit).

‡ To be completed by specialist or trained medical providers (see Supplemental Figure).

#### Source:

Jagasia HM, Greinix HT, Arora M, et al. Biol Blood Marrow Transplant. 2015;21:389–401.

# Appendix O. NIH Global Severity/Staging of cGVHD

#### Mild chronic GVHD

1 or 2 Organs involved with no more than score 1

plus

Lung score 0

### **Moderate chronic GVHD**

3 or More organs involved with no more than score 1

OR

At least 1 organ (not lung) with a score of 2

OR

Lung score 1

### **Severe chronic GVHD**

At least 1 organ with a score of 3

OR

Lung score of 2 or 3

### **Key points:**

- In skin: higher of the 2 scores to be used for calculating global severity.
- In lung: FEV1 is used instead of clinical score for calculating global severity.
- If the entire abnormality in an organ is noted to be unequivocally explained by a non-GVHD documented cause, that organ is not included for calculation of the global severity.
- If the abnormality in an organ is attributed to multifactorial causes (GVHD plus other causes) the scored organ will be used for calculation of the global severity regardless of the contributing causes (no downgrading of organ severity score).

### Reference:

Jagasia HM, Greinix HT, Arora M, et al. Biol Blood Marrow Transplant. 2015;21:389–401.

# Appendix P. Late Effects Surveillance for Adolescents

In addition to procedures listed in Appendix A and Appendix B, adolescents (≥12 to <22 years of age at the time of randomization) will be monitored for growth and development, immune reconstitution, and late effects up to 5 years post randomization.

| | Screening | Week 49±7 days | At month 24, 36,<br>48, 60 ±30 days |
|---|---|---|---|
| Additional measurements | | | |
| Height and Weight | X | X | X |
| Tanner Stage | X | X | X |
| Immune Reconstitution <sup>a</sup> Tests | | X | X |
| <b>History of Late Effects (chart review)</b> | X | X | Xb |

<sup>&</sup>lt;sup>a</sup> Immune reconstitution studies will include the following studies obtained as part of standard of care:

- o T and B cell enumeration
- Quantitative Immunoglobulins
- Post-vaccination titers
- b Are obtained annually. Post vaccination studies may not be performed annually

# **Medical Record Review for Transplant-Related Late Effects**

| | | yes | | |
|---|---|---|---|---|
| Symptom | No | Date of<br>Diagnosis | Was therapy<br>Given? | Was therapy still given at the time this assessment |
| Diabetes/hyperglycemia requiring chronic treatment | | | | |
| Hyperlipidemia requiring therapy | | | | |
| Hypothyroidism requiring hormone replacement | | | | |
| Gonadal dysfunction requiring hormone replacement (testosterone or estrogen/progesterone) | | | | |
| Growth hormone deficiency/short stature | | | | |
| Avascular necrosis | | | | |
| Osteoporosis | | | | |
| Osteoporotic fracture | | | | |
| Depression or anxiety requiring therapy | | | | |
| Post-traumatic stress disorder requiring therapy | | | | |
| Cataracts | | | | |
| Other impairment or disease | | | | |
| B-cell immune deficiency | | | | |
| vaccines received over the last year | | If vaccines admin | istered complete in | nmunization CRF |

# **Tanner Stage**

# **Boys – Development of external genitalia**

- Stage 1: Prepubertal
- Stage 2: Enlargement of scrotum and testes; scrotum skin reddens and changes in texture
- **Stage 3:** Enlargement of penis (length at first); further growth of testes
- **Stage 4:** Increased size of penis with growth in breadth and development of glans; testes and scrotum larger, scrotum skin darker
- Stage 5: Adult genitalia

## **Girls – Breast development**

- **Stage 1:** Prepubertal
- Stage 2: Breast bud stage with elevation of breast and papilla; enlargement of areola
- Stage 3: Further enlargement of breast and areola; no separation of their contour
- **Stage 4:** Areola and papilla form a secondary mound above level of breast
- Stage 5: Mature stage: projection of papilla only, related to recession of areola

### Boys and Girls – Pubic hair

- **Stage 1:** Prepubertal (can see velus hair similar to abdominal wall)
- **Stage 2:** Sparse growth of long, slightly pigmented hair, straight or curled, at base of penis or along labia
- Stage 3: Darker, coarser and more curled hair, spreading sparsely over junction of pubes
- **Stage 4:** Hair adult in type, but covering smaller area than in adult; no spread to medial surface of thighs
- **Stage 5:** Adult in type and quantity, with horizontal distribution ("feminine")

# Appendix Q. Corticosteroid-related toxicities and CTCAE preferred terms

| Corticosteroid symptom | CTCAE graded AE |
|---|---|
| Glucose intolerance related to steroid use | Glucose intolerance |
| Elevated lipids related to steroid use | Hypertriglyceridemia, Cholesterol high |
| Hypertension | Hypertension |
| Steroid myopathy | Generalized muscle weakness |
| Steroid skin toxicity (eg, striae, thinning of skin, etc.) | Skin atrophy |
| Neuropsychiatric symptoms including insomnia | Insomnia, Agitation, Psychosis, or other psychiatric symptoms |
| Oral/vaginal candidiasis or uncomplicated zoster infection | Mucosal infection (e.g. oral/vaginal candidiasis) |
| Any other infection | Infections |
| Diabetic nephropathy-related to steroid use | Proteinuria |
| Posterior reversible encephalopathy | Encephalopathy, Reversible posterior leukoencephalopathy syndrome |
| Abnormal bone density (>than - 2 Z score) | Osteoporosis (Osteopenia with a t-score -1 to -2.5) |
| Insufficiency (pathologic) bone fractures | Fracture |
| Adrenal insufficiency | Adrenal insufficiency |
| Gastrointestinal perforation | Gastric perforation, Esophageal perforation,<br>Duodenal perforation, Colonic perforation, Ileal<br>perforation |
| Peptic ulcer disease | Duodenal ulcer |
| Osteonecrosis of bones (avascular necrosis) | Periodontal disease, Avascular necrosis |
| Tendon rupture | Musculosceletal and connective disorders, other |
| Retinopathy (diabetic or central serous (choroidal) retinopathy) | Retinopathy |
| Intraocular pressure elevation | Glaucoma, papilledema or eye disorder, other |
| Posterior subcapsular cataract | Cataract |